# **Cover Page for Protocol**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT04017832 |
| Sponsor trial ID: | NN9924-4309 |
| Official title of study: | PIONEER 12 China multi-regional clinical trial: Efficacy and safety of oral semaglutide versus sitagliptin in subjects with type 2 diabetes mellitus treated with metformin |
| Document date*: | 28 January 2019 |

<sup>\*</sup>Document date refers to the date on which the document was most recently updated.

Note: The date in the header from Page 2 is the date of compilation of the documents and not of an update to content.

| Oral semaglutide |
|------------------------------------|
| Trial ID: NN9924 4309 (PIONEER 12) |
| Clinical Trial Report |
| Appendix 16.1.1 |

Date: Version: Status:

11 February 2022 | Novo Nordisk 1.0 Final

# 16.1.1 Protocol and protocol amendments

# List of contents

| Protocol | Link |
|---------------------|------|
| Appendix A | Link |
| Appendix B | Link |
| Appendix C | Link |
| Attachment I and II | Link |

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.

Protocol

Trial ID: NN9924-4309 UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38


Date: Version: Status: Page:

28 January 2019 3.0 Final 1 of 120

Novo Nordisk

# **Protocol**

Updated protocol including:

Protocol Final version 1.0, dated 31 January 2017

Protocol Amendment no. 1, Final version 1.0, dated 31 August 2018

Protocol Amendment no. 2. Final version 3.0, dated 15 January 2019

Trial ID: NN9924-4309

PIONEER 12 China multi-regional clinical trial: Efficacy and safety of oral semaglutide versus sitagliptin in subjects with type 2 diabetes mellitus treated with metformin

> Redacted protocol *Includes redaction of personal identifiable information only.*

> > Trial phase: 3a

### **Protocol originator**

Trial Operations, Semaglutide Diabetes & Diabetes Outcome

In the following, Novo Nordisk A/S and its affiliates will be stated as "Novo Nordisk".

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.

Protocol v 3 consol 1 of 145 Protocol Trial ID: NN9924-4309 UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38


Date: Version: Status: Page:

28 January 2019 | Novo Nordisk 3.0 Final 2 of 120

# **Table of contents**

| | | | | | Page |
|---|---|---|---|---|---|
| Ta | ble of c | ontents | | | 2 |
| Ta | ble of f | igures | ••••• | | 6 |
| | | _ | | | |
| 1 | Sumn | nary | ••••• | | 10 |
| 2 | Flow | chart | ••••• | | 13 |
| 3 | Back | ground inf | formation an | d rationale for the trial | 17 |
| | 3.1 | | ound informat | ion | 17 |
| | | 3.1.1 | Type 2 dia | nbetes mellitus | 17 |
| | | 3.1.2 | Glucagon- | ·like peptide-1 | 17 |
| | | 3.1.3 | Oral sema | glutide | 17 |
| | | 3.1.4 | Non-clinic | cal data | 18 |
| | | | 3.1.4.1 | Semaglutide | 18 |
| | | | 3.1.4.2 | SNAC | 19 |
| | | 3.1.5 | Clinical da | ata for oral semaglutide | 20 |
| | | | 3.1.5.1 | Pharmacokinetics | |
| | | | 3.1.5.2 | Efficacy | 21 |
| | | | 3.1.5.3 | Safety | |
| | | 3.1.6 | O 1 | | |
| | 3.2 | Rationa | le for the trial | | 22 |
| 4 | Objec | | | | |
| | 4.1 | Objectiv | | | |
| | | 4.1.1 | | bjective | |
| | | 4.1.2 | | objectives | |
| | 4.2 | Endpoir | | | |
| | | 4.2.1 | | ndpoint | |
| | | 4.2.2 | | endpoints | |
| | | | 4.2.2.1 | Confirmatory secondary endpoints | |
| | | | 4.2.2.2 | Supportive secondary endpoints | 23 |
| 5 | Trial | design | ••••• | | 25 |
| | 5.1 | Type of | `trial | | 25 |
| | 5.2 | Rationa | le for trial des | ign | 25 |
| | 5.3 | Treatme | ent of subjects | | 26 |
| | | 5.3.1 | Dosing ins | structions | 27 |
| | | 5.3.2 | | nd medication | |
| | 5.4 | | | ntinuation of trial product | |
| | 5.5 | Rationa | le for treatmen | nt | 28 |
| 6 | Trial | populatio | n | | 29 |
| | 6.1 | | | | |
| | 6.2 | | | | |
| | 6.3 | Exclusion | on criteria | | 29 |

| UTN | l ID: NN99<br>N: U1111-1 | 924-4309<br>1188-1256<br>2018-002589- | 38 | CONFIDENTI | <del>AL</del> | Date:<br>Version:<br>Status:<br>Page: | 28 January 2019<br>3.0<br>Final<br>3 of 120 | |
|---|---|---|---|---|---|---|---|---|
| | 6.4<br>6.5<br>6.6<br>6.7<br>6.8 | Criteria for<br>Withdrawa<br>Subject rep | r premature<br>al from tria<br>placement. | e discontinuation of | trial produc | t | | 31<br>32<br>32 |
| 7 | | | | • | | | | |
| 8 | Method | ds and asse | essments | | | | ••••• | 35 |
| | 8.1 | | | | | | | |
| | 011 | 8.1.1 | | | | | | |
| | | 8.1.2 | | | | | | |
| | | 8.1.3 | | | | | | |
| | | 8.1.4 | | | | | | |
| | | 8.1.5 | | | | | p (visits 8A and 9A) | |
| | | 8.1.6 | | | | | (VISIOS OTT UITA 571) | |
| | | 0.1.0 | 8.1.6.1 | | | | | |
| | | 8.1.7 | | | | | | |
| | 8.2 | | | | | | | |
| | 0.2 | 8.2.1 | | | | | | |
| | | 8.2.2 | | • | | | | |
| | | 8.2.3 | | | | | | |
| | | 8.2.4 | | | | | | |
| | | 8.2.5 | | | | | | |
| | | 8.2.6 | | | | | | |
| | 8.3 | | | | | | | |
| | 0.5 | 8.3.1 | I ahorator | v assessments for ef | ficacy | •••••• | | 42 |
| | | 8.3.2 | Self-meas | ured plasma glucose | (SMPG) | •••••• | | 42 |
| | | 0.5.2 | 8.3.2.1 | | | | ofile | |
| | | 8.3.3 | | | | | | |
| | | 8.3.4 | | $\mathcal{E}$ | | | | |
| | | 8.3.5 | | | | | | |
| | | 8.3.6 | | | | | | |
| | | 0.5.0 | 8.3.6.1 | | | | collection | |
| | | 8.3.7 | | | | | | |
| | | 8.3.8 | • | | | | | |
| | | 8.3.9 | | | | | | |
| | | 8.3.10 | | | | | | |
| | | 8.3.11 | | · / | | | | |
| | | 8.3.12 | | • | • | | | |
| | | 8.3.13 | | | | | | |
| | 8.4 | | • • • • | | | | | |
| | 8.5 | • | , | | | | | |
| | 0.5 | 8.5.1 | | | | | | |
| | 8.6 | | | • | | | | |
| | | Ü | • | | | | | |
| 9 | | | | | | | ••••• | |
| | 9.1 | | | | | | | |
| | 9.2 | _ | | | | | | |
| | 9.3 | Storage | | | | | | 54 |

| 9.4 Drug accountability and destruction | 55 |
|------------------------------------------------------------------------|----|
| 9.5 Auxiliary supplies | 56 |
| 10 Interactive voice/web response system | |
| 11 Randomisation procedure and breaking of blinded codes | |
| 11.1 Breaking of blinded codes | |
| 12 Adverse events, technical complaints and pregnancies | |
| 12.1 Definitions | 58 |
| 12.1.1 Adverse event | |
| 12.1.2 Serious adverse event | |
| 12.1.3 Non-serious adverse event | 60 |
| 12.1.4 Medication errors | 60 |
| 12.1.4.1 Misuse or abuse of trial product | |
| 12.1.5 Adverse events requiring additional data collection | 61 |
| 12.1.6 Technical complaints | |
| 12.2 Reporting of adverse events | |
| 12.3 Follow-up of adverse events | |
| 12.4 Technical complaints and technical complaint samples | |
| 12.4.1 Reporting of technical complaints | |
| 12.4.2 Collection, storage and shipment of technical complaint samples | |
| 12.5 Pregnancies in female subjects | |
| 12.6 Precautions and/or overdose | |
| 12.7 Committees related to safety | |
| 12.7.1 Novo Nordisk safety committee | |
| 12.7.2 Event adjudication committee | /0 |
| 13 Case report forms | |
| 13.1 Corrections to case report forms | |
| 13.2 Case report form flow | 76 |
| 14 Monitoring procedures | 77 |
| 15 Data management | |
| 16 Computerised systems | 80 |
| 17 Statistical considerations | |
| 17.1 Sample size calculation | |
| 17.2 Primary endpoint | |
| 17.2.1 Primary analysis for the primary estimand | |
| 17.2.2 Primary analysis for the secondary estimand | |
| 17.2.3 Sensitivity analyses | |
| 17.2.3.1 Other sensitivity analyses | |
| 17.2.4 Chinese subgroup analyses | |
| 17.3 Secondary endpoints | |
| 17.3.1 Confirmatory secondary endpoints | |
| 17.3.2 Supportive secondary endpoints | |
| <b>J</b> 1 | |
| 17.3.2.2 Safety endpoints | |
| 17.5 Patient-reported outcomes | |

| Tria<br>UTI | ocol<br>1 ID: NN99<br>N: U1111-1<br>raCT no.: 2 | | 9-38 | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 28 January 2019<br>3.0<br>Final<br>5 of 120 | Novo Nordisk |
|---|---|---|---|---|---|---|---|
| | | 17.5.1<br>17.5.2 | | ® (acute version) health si<br>er analyses | | | |
| 18 | Ethics. | ••••• | • | | ••••• | ••••• | 102 |
| | 18.1 | Benefit-r | | ent of the trial | | | |
| | | 18.1.1 | | l precautions | | | |
| | | | 18.1.1.1 | $\boldsymbol{\mathcal{E}}$ | | | |
| | | 18.1.2 | 18.1.1.2 | $\mathcal{U}$ 1 | | | |
| | | 18.1.2 | | benefit conclusion | | | |
| | 18.2 | | | | | | |
| | 18.3 | | | | | | |
| | 18.4 | Informat | ion to subjec | cts during trial | | | 107 |
| | 18.5 | Prematur | re termination | on of the trial and/or trial sit | te | | 107 |
| 19 | Protoco | ol compli | ance | | | | 108 |
| | 19.1 | _ | | | | | |
| | 19.2 | Prevention | on of missin | g data | | | 108 |
| 20 | Audits | and insp | ections | ••••• | | ••••• | 109 |
| 21 | Critica | l docume | nts | | | | 110 |
| 22 | Respon | sibilities | ••••• | | | ••••• | 111 |
| 23 | Report | s and pul | olications | | | | 112 |
| | 23.1 | | | esults | | | |
| | | 23.1.1 | | ip | | | |
| | | 23.1.2 | | ific publication(s) by invest | | | |
| | 23.2 | Investiga | itor access to | o data and review of results | | | 113 |
| 24 | Retenti | on of clir | nical trial do | ocumentation and human | biosamples | ••••• | 114 |
| | 24.1 | Retention | n of clinical | trial documentation | | | 114 |
| 25 | Institut | tional Re | view Boards | s/Independent Ethics Con | nmittees and regula | atory authorities | 115 |
| 26 | Indem | nity state | ment | | | ••••• | 116 |
| 27 | Refere | nces | ••••• | ••••• | •••••• | ••••• | 117 |
| ۸n | pendix A | ۸ ( | Calcitonin n | aonitorina | | | |
| - | pendix l | | | ents requiring additional of | lata collection | | |
| - | - | | | | | formation | |
| - | pendix ( | | | ve guidance and collection | | | |
| | achmen | | | f key staff and relevant d | | ppners | |
| Att | achmen | t II C | ountry list | of key staff and relevant | aepartments | | |

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


# **Table of figures**

EudraCT no.: 2018-002589-38

| | | Page |
|---|---|---|
| Figure 5–1 | Trial Design | 25 |
| Figure 12–1 | Reporting of adverse events | 65 |
| Figure 17–1 | Graphical illustration of the closed testing procedure | 85 |
| Figure 17–2 | ADA classification of hypoglycaemia | 98 |
| Table of | tables | |
| | | Page |
| Table 5–1 | Overview – treatment of subjects | 27 |
| Table 9–1 | Trial Products | 53 |
| Table 12–1 | Adverse events requiring completion of specific event forms and/or are subject to adjudication | |
| Table 12–2 | Adverse events for adjudication | 72 |
| Table 17–1 | Assumptions for sample size calculation | 84 |
| Table 17–2 | Calculated powers for individual hypotheses | 84 |
| Table 5–1 | Overview – treatment of subjects | 27 |
| Table 9–1 | Trial Products | 53 |
| Table 12–1 | Adverse events requiring completion of specific event forms and/or are subject to adjudication | |
| Table 12–2 | Adverse events for adjudication | 72 |
| Table 17–1 | Assumptions for sample size calculation | 84 |
| Table 17–2 | Calculated powers for individual hypotheses | 84 |
| Table 5–1 | Overview – treatment of subjects | 27 |
| Table 9–1 | Trial Products | 53 |
| Table 12–1 | Adverse events requiring completion of specific event forms and/or are subject to adjudication | |
| Table 12–2 | Adverse events for adjudication | 72 |
| Table 17–1 | Assumptions for sample size calculation | 84 |
| Table 17–2 | Calculated powers for individual hypotheses | 84 |
| Table 5–1 | Overview – treatment of subjects | 27 |
| Table 9–1 | Trial Products | 53 |
| Table 12–1 | Adverse events requiring completion of specific event forms and/or are subject to adjudication | |

| Protocol<br>Trial ID: NN9924-<br>UTN: U1111-1188 | 3-1256 | CONFIDENTIAL | Date:<br>Version:<br>Status: | 28 January 2019<br>3.0<br>Final | Novo Nordisk |
|---|---|---|---|---|---|
| EudraCT no.: 2018 | 3-002589-38 | | Page: | 7 of 120 | |
| Table 12–2 | Adverse events for | or adjudication | | | 72 |
| Table 17–1 | Assumptions for s | sample size calculation | | | 84 |
| Table 17–2 | Calculated power | s for individual hypotheses. | | | 84 |
| Table 5–1 | Overview – treatr | nent of subjects | | | 27 |
| Table 9–1 | Trial Products | | | | 53 |
| Table 12–1 | | quiring completion of speci | | | |
| Table 12–2 | Adverse events for | or adjudication | | | 72 |
| Table 17–1 | Assumptions for s | sample size calculation | | | 84 |
| Table 17–2 | Calculated power | s for individual hypotheses. | | | 84 |

Protocol v 3 consol | 7 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

# List of abbreviations

AACE American Association of Clinical Endocrinologists

ADA American Diabetes Association

AE adverse event

ALT alanine aminotransferase
ANCOVA analysis of covariance

AST aspartate aminotransferase

AUC area under the curve

BG blood glucose
BMI body mass index
CK creatine kinase

CKD-EPI Chronic Kidney Disease Epidemiology Collaboration

C<sub>max</sub> maximum concentration

CRF case report form
CTR clinical trial report
DPP-4 dipeptidyl peptidase-4

DUN dispensing unit number

EAC event adjudication committee

ECG electrocardiogram

eCRF electronic case report form

eGFR estimated glomerular filtration rate

EOT end-of-treatment
FAS full analysis set

FPG fasting plasma glucose
GCP Good Clinical Practice

GI gastrointestinal

GLP-1 glucagon-like peptide-1

GLP-1 RA glucagon-like peptide-1 receptor agonist

 $\begin{array}{ll} \mbox{HbA}_{1c} & \mbox{glycosylated haemoglobin} \\ \mbox{HDL} & \mbox{high-density lipoprotein} \end{array}$ 

IB Investigator's brochure

Protocol v 3 consol 8 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

ICH International Conference on Harmonisation of Technical

Requirements for Registration of Pharmaceuticals for Human Use

ICMJE International Committee of Medical Journal Editors

IEC independent ethics committee
IRB institutional review board

IWRS interactive web response system

LDL low-density lipoprotein

MAR missing at random

MI myocardial infarction

MMRM mixed model for repeated measurements

NYHA New York Heart Association

OAD oral antidiabetic drug

PG plasma glucose

PIONEER Peptide InnOvation for Early diabEtes tReatment

PRO patient-reported outcome
SAE serious adverse event
SAS safety analysis set
s.c. subcutaneous(ly)

SIF safety information form

SmPC summary of product characteristics

SMPG self-measured plasma glucose

SNAC sodium N-[8-(2-hydroxybenzoyl) amino]caprylate

SUSAR suspected unexpected serious adverse reaction

T2D type 2 diabetes mellitus

TE treatment effects

TEAE treatment-emergent adverse event

 $t_{max}$  time to reach maximum observed concentration

ULN upper limit of the normal UTN Universal Trial Number

VLDL very-low-density lipoprotein

Protocol v 3 consol 9 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


# 1 Summary

EudraCT no.: 2018-002589-38

# Objectives and endpoints:

### Primary objective

To compare the effect of three once-daily dose levels of oral semaglutide (3, 7 and 14 mg) versus sitagliptin 100 mg once-daily, both in combination with metformin, on glycaemic control in subjects with type 2 diabetes mellitus (T2D).

# Secondary objectives

To compare the effect of three once-daily dose levels of oral semaglutide (3, 7 and 14 mg) versus sitagliptin 100 mg once-daily, both in combination with metformin, on body weight in subjects with T2D.

To compare the safety and tolerability of three once-daily dose levels of oral semaglutide (3, 7 and 14 mg) versus situation in subjects with methors with methors, in subjects with T2D.

## **Primary endpoint**

Change from baseline to week 26 in HbA<sub>1c</sub>

# Key secondary endpoints

- Change from baseline to week 26 in body weight (kg)
- Change from baseline to week 26 in fasting plasma glucose
- If a subject after week 26 achieves (yes/no) HbA<sub>1c</sub> < 7.0 % (53 mmol/mol) (American Diabetes Association target)
- Number of treatment-emergent adverse events during exposure to trial product, assessed up to approximately 31 weeks
- Number of treatment-emergent severe or blood glucose confirmed symptomatic hypoglycaemic episodes during exposure to trial product, assessed up to approximately 31 weeks

# Trial design:

This is a 26-week, randomised, double-blinded, double-dummy, active-controlled, four-armed, parallel-group, multicentre, multinational trial comparing the efficacy and safety of three once-daily dose levels of oral semaglutide versus situagliptin once-daily in subjects with T2D inadequately controlled on metformin.

#### **Trial population:**

Number of subjects planned to be randomised: 1444

Protocol v 3 consol | 10 of 145

| Protocol | | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | EudraCT no.: 2018-002589-38 | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | Page: 12 of 1

#### Inclusion criteria:

- Informed consent obtained before any trial-related activities. Trial-related activities are any
  procedures that are carried out as part of the trial, including activities to determine suitability for
  the trial.
- Male or female, age above or equal to 18 years at the time of signing informed consent. <u>For Algeria only</u>: Male or female, age above or equal to 19 years at the time of signing informed consent.
  - <u>For Taiwan only</u>: Male or female, age above or equal to 20 years at the time of signing informed consent
- Diagnosed with type 2 diabetes mellitus  $\geq$  60 days prior to day of screening.
- HbA<sub>1c</sub> between 7.0-10.5% (53-91 mmol/mol) (both inclusive).
- Stable daily dose of metformin ( $\geq 1500$  mg or maximum tolerated dose as documented in the subject medical record)  $\geq 60$  days prior to day of screening

#### Key exclusion criteria:

- Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method (adequate contraceptive measure as required by local regulation or practice).
- Family or personal history of multiple endocrine neoplasia type 2 (MEN 2) or medullary thyroid carcinoma (MTC). Family is defined as a first degree relative.
- History or presence of pancreatitis (acute or chronic).
- History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).
- Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening and randomisation.
- Subjects presently classified as being in New York Heart Association (NYHA) Class IV.
- Planned coronary, carotid or peripheral artery revascularisation known on the day of screening.
- Renal impairment measured as estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m<sup>2</sup> as per Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI).
- Subjects with alanine aminotransferase (ALT) > 2.5 x upper limit of the normal (ULN).
- Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a pharmacologically pupil-dilated fundus examination performed by an ophthalmologist or another suitably qualified health care provider within the past 90 days prior to screening or in the period between screening and randomisation. Fundus examination without dilation is only allowed if the digital camera used for fundus photography has this feature.
- Presence or history of malignant neoplasms within the past 5 years prior to the day of screening. Basal and squamous cell skin cancer and any carcinoma in-situ is allowed.

Protocol v 3 consol | 11 of 145

# **Key assessments:**

# Efficacy:

- HbA<sub>1c</sub>
- Body weight
- Fasting plasma glucose

# Safety

- Adverse events
- Hypoglycaemic episodes

# **Trial product(s):**

Investigational medicinal products:

- Test product:
  - Semaglutide 3 mg, 7 mg and 14 mg tablets
- Reference therapy:
  - Semaglutide placebo tablet
  - Sitagliptin (Januvia®), 100 mg tablet
  - Sitagliptin (Januvia®) placebo tablet

Protocol v 3 consol | 12 of 145

 Protocol
 UTN: U1111-1188-1256
 Date:
 28 January 2019
 Status:
 Final
 Novo Nordisk

 Trial ID: NN9924-4309
 EudraCT no.: 2018-002589-38
 Version:
 3.0
 Page:
 Novo Nordisk

# 2 Flow chart

| Trial Periods | Protocol<br>section | Screening <sup>a</sup> | Randomisation <sup>e</sup> | | Treatment | | | End of<br>treatment | Follow-<br>up <sup>b</sup> | End of<br>treatment <sup>c</sup><br>premature<br>discontinuation | Follow-up <sup>c</sup><br>premature<br>discontinuation | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit (V), Phone contact (P) | | V1 | V2 | P3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 | V8A | V9A |
| Timing of visit (Weeks) | | -2 | 0 | 2 | 4 | 8 | 14 | 20 | 26 | 31 | Day of<br>discontinuation<br>of trial product | 5 weeks after<br>discontinuation<br>of trial product |
| Visit window (Days) | | -7 | | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | +3 | +3 | +3 |
| SUBJECT RELATED INFO/AS | SESSMENT | rs. | | | | | | | | | | |
| Informed consent | 18.2 | X | | | | | | | | | | |
| In/exclusion criteria | <u>6.2</u> , <u>6.3</u> | X | X | | | | | | | | | |
| Demography | <u>8.2.1</u> | X | | | | | | | | | | |
| Diabetes History | 8.2.2 | X | | | | | | | | | | |
| Concomitant illness and Medical history | 8.2.3 | х | | | | | | | | | | |
| Concomitant medication | 8.2.4 | X | X | X | X | X | X | X | X | X | x | X |
| History of gastrointestinal disease | 8.2.3 | х | | | | | | | | | | |
| History of gallbladder disease | 8.2.3 | Х | | | | | | | | | | |
| History of cardiovascular disease | 8.2.3 | Х | | | | | | | | | | |
| Childbearing potential | <u>8.2.5</u> | Х | | | | | | | | | | |
| Tobacco use | 8.2.6 | X | | | | | | | | | | |
| Randomisation | <u>8.1.3</u> | | X | | | | | | | | | |
| Rescue criteria | <u>6.4</u> | | | | | X | X | X | | | | |
| Criteria for premature discontinuation of trial product | <u>6.5, 8.1.5</u> | | | x | x | x | х | х | | | | |
| EFFICACY | | | | | | | | | | | | |
| HbA <sub>1c</sub> | 8.3.1 | X | X | | X | X | X | X | X | | x | |
| Fasting plasma glucose | 8.3.1 | | X | | X | X | X | | X | | x | |
| 7-point SMPG profile | <u>8.3.2</u> , | | X | | | | | | X | | X | |

 Protocol
 UTN: U1111-1188-1256
 Date:
 28 January 2019
 Status:
 Final
 Novo Nordisk

 Trial ID: NN9924-4309
 EudraCT no.: 2018-002589-38
 Version:
 3.0
 Page:
 Novo Nordisk

| Trial Periods | Protocol<br>section | Screening <sup>a</sup> | Randomisation <sup>e</sup> | | Treatment | | | | End of<br>treatment | Follow-<br>up <sup>b</sup> | End of<br>treatment <sup>c</sup><br>premature<br>discontinuation | Follow-up <sup>c</sup><br>premature<br>discontinuation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit (V), Phone contact (P) | | V1 | V2 | P3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 | V8A | V9A |
| Timing of visit (Weeks) | | -2 | 0 | 2 | 4 | 8 | 14 | 20 | 26 | 31 | Day of<br>discontinuation<br>of trial product | 5 weeks after<br>discontinuation<br>of trial product |
| Visit window (Days) | | -7 | | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | +3 | +3 | +3 |
| | 8.3.2.1 | | | | | | | | | | | |
| Height | <u>8.3.3</u> | | x | | | | | | | | | |
| Body weight | <u>8.3.3</u> | | x | | X | X | X | X | X | | x | |
| Waist circumference | <u>8.3.4</u> | | X | | | | X | | X | | X | |
| Lipids | <u>8.3.1</u> | | x | | | | X | | X | | x | |
| PRO questionnaire | <u>8.3.5</u> | | X | | | X | | | X | | X | |
| SAFETY | | | | | | | | | | | | |
| Adverse events <sup>h</sup> | <u>8.4.1</u> , <u>12</u> | X | X | X | X | X | X | X | X | X | X | X |
| Technical complaints | <u>12</u> | | X | X | X | X | X | X | X | | X | |
| Hypoglycaemic episodes | <u>8.4.9</u> | X | X | X | X | X | X | X | X | X | X | X |
| Eye examination <sup>d</sup> | <u>8.4.4</u> | X | | | | | | | X | | X | |
| Physical examination | <u>8.4.2</u> | X | | | | | | | X | | X | |
| Vital signs | <u>8.4.3</u> | | X | | X | X | X | X | X | X | X | X |
| Haematology | <u>8.4.6</u> | | X | | | X | X | | X | X | X | X |
| Calcitonin | <u>8.4.6</u> | | X | | | | X | | X | X | X | X |
| Biochemistry <sup>j</sup> | <u>8.4.6</u> | X | x | | | X | X | | X | X | x | x |
| Pregnancy test <sup>f</sup> | <u>8.4.7</u> | Х | x | | X | X | X | X | X | х | х | х |
| ECG | <u>8.4.5</u> | | x | | | | | | X | X | x | х |
| TRIAL MATERIAL | • | | • | | | | | | | | | |
| IWRS call | <u>10</u> | X | x | | X | X | х | X | X | | x | |
| Dispensing visit | <u>9</u> | | x | | х | X | X | X | | | | |
| Drug accountability | <u>9.4</u> | | x | | X | X | X | X | X | | х | |
| REMINDERS | | | | | | | | | | | | |

# VV-TMF-698732I1.0INN9924 -4309

 Protocol
 UTN: U1111-1188-1256
 Date:
 28 January 2019
 Status:
 Final
 Novo Nordisk

 Trial ID: NN9924-4309
 EudraCT no.: 2018-002589-38
 Version:
 3.0
 Page:
 Novo Nordisk

| Trial Periods | Protocol<br>section | Screening <sup>a</sup> | Randomisation <sup>e</sup> | | Treatment | | | | End of<br>treatment | Follow-<br>up <sup>b</sup> | End of<br>treatment <sup>c</sup><br>premature<br>discontinuation | Follow-up <sup>c</sup><br>premature<br>discontinuation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit (V), Phone contact (P) | | V1 | V2 | P3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 | V8A | V9A |
| Timing of visit (Weeks) | | -2 | 0 | 2 | 4 | 8 | 14 | 20 | 26 | 31 | Day of<br>discontinuation<br>of trial product | 5 weeks after<br>discontinuation<br>of trial product |
| Visit window (Days) | | -7 | | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | +3 | +3 | +3 |
| Handout and instruct in BG meter use | 8.3.2 | x | | | | | | | | | | |
| Handout ID card | 8.1.1 | X | | | | | | | | | | |
| Handout and instruct in diary | 8.6.1 | X | X | | X | X | X | X | X | X | X | x |
| Training in trial products and dosing instructions | 8.1.3 | | х | х | х | x | х | х | | | | |
| Attend visit fasting | <u>8.1.2</u> | | x | | X | X | X | | X | | x | |
| End of treatment | <u>8.1.4</u> | | | | | | | | X | | X | |
| End of trial <sup>g</sup> | <u>8.1.4</u> | | | | | | | | | X | | |

# VV-TMF-698732I1.0INN9924 -4309

 Protocol
 UTN: U1111-1188-1256
 Date:
 28 January 2019
 Status:
 Final
 Novo Nordisk

 Trial ID: NN9924-4309
 EudraCT no.: 2018-002589-38
 Version:
 3.0
 Page:
 Novo Nordisk

| Footer | Description |
|---|---|
| | The subject can be randomised as soon as all inclusion and exclusion criteria are confirmed. The screening assessments must not exceed 3 weeks prior to |
| a | V2. |
| | The follow-up visit (V9) should be scheduled 5 weeks after the last date on trial product (+3 days visit window). Subjects, who have discontinued trial |
| b | product prematurely, are not required to attend V9. |
| c | V8A and V9A are only applicable for subjects who have discontinued trial product prematurely. |
| | Fundus examination performed by an ophthalmologist or another suitably qualified health care provider (e.g. optometrist) within the past 90 days prior to screening or in the period between screening and randomisation.is acceptable if results are available for evaluation at V2, unless worsening of visual function since last examination. Fundus examination must be performed again: |
| | <ul> <li>at V8 or within 5 weeks thereafter (for subjects completing treatment)</li> <li>at V8A or within 5 weeks thereafter, and again within 5 weeks prior to V8 (for subjects who have prematurely discontinued trial product) unless overlapping with the V8A assessment.</li> </ul> |
| d | (The specific eye examination requirements are described in section 8.4.4) |
| e | At randomisation, the blood sampling must be done pre-dose. |
| f | For women of child-bearing potential: Urine pregnancy test should also be performed at any time during the trial if menstrual period is missed, and/or according to local regulations/law. |
| g | For subjects who have discontinued trial product prematurely, the end of trial is V8 (or V9A if it is scheduled after V8). |
| h | Adverse events reporting includes adverse events from the first trial related-activity after the subject has signed the informed consent at V1, Pre-existing conditions identified as a result of screening procedures should be reported as medical history. |
| i | Fasting blood sampling is defined as no food or liquid within the last 8 hours prior to blood sampling, however water is allowed up until 2 hours prior to blood sampling. |
| j | At V1, only ALT, creatinine and eGFR will be assessed as part of Biochemistry |

Protocol Date: 28 January 2019 Novo Nordisk
Trial ID: NN9924-4309 Version: 3.0

Status:

Page:

Final


UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38

3

# Background information and rationale for the trial

The trial will be conducted in compliance with this protocol, ICH GCP<sup>1</sup> and applicable regulatory requirements, and in accordance with the Declaration of Helsinki<sup>2</sup>.

In this document, the term investigator refers to the individual responsible for the overall conduct of the clinical trial at a trial site.

## 3.1 Background information

For an assessment of benefits and risks of the trial, see Section <u>18.1</u>

# 3.1.1 Type 2 diabetes mellitus

Type 2 diabetes mellitus (T2D) is a progressive metabolic disease primarily characterised by abnormal glucose metabolism. The pathogenesis is heterogeneous involving environmental, lifestyle and genetic factors leading to chronic hyperglycaemia caused by peripheral tissue insulin resistance, impaired insulin secretion due to abnormal beta-cell function and abnormal glucose metabolism in the liver<sup>3</sup>.

Optimal glycaemic control is the treatment goal in subjects with T2D in order to prevent long-term complications associated with chronic hyperglycaemia<sup>3</sup>. Despite the availability of several antidiabetic drugs, a significant proportion of subjects with T2D do not achieve the recommended targets for glycaemic control<sup>4,5</sup>.

### 3.1.2 Glucagon-like peptide-1

Glucagon-like peptide-1 (GLP-1) is an incretin hormone with a glucose-dependent stimulatory effect on insulin and inhibitory effect on glucagon secretion from the pancreatic islets<sup>6,7</sup>. Subjects with T2D have a decreased incretin effect<sup>8,9</sup>. However, the insulinotropic action of GLP-1 and thus, the ability to lower blood glucose (BG) levels, is preserved when GLP-1 is administered at supraphysiological levels<sup>10</sup>. In addition, supraphysiological levels of GLP-1 induce reduction in body weight<sup>11</sup>. GLP-1 is a physiological regulator of appetite and food intake and GLP-1 receptors are present in several areas of the brain involved in appetite regulation<sup>12,13</sup>. Physiologically, GLP-1 also has a pronounced inhibitory effect on gastric emptying; however this effect seems to diminish upon chronic exposure<sup>11,13</sup>. These mechanisms of action make GLP-1 receptor agonists (GLP-1 RA) an attractive pharmacological treatment for T2D<sup>14,15</sup>.

#### 3.1.3 Oral semaglutide

Semaglutide is a long-acting GLP-1 RA structurally similar to liraglutide (Victoza<sup>®</sup>), a once-daily GLP-1 RA developed by Novo Nordisk and approved worldwide for the treatment of T2D. Compared to human native GLP-1, which has a short half-life, the semaglutide molecule has three minor but important modifications ensuring protraction of its action: amino acid substitutions at position 8 (alanine to alpha-aminoisobutyric acid, a synthetic amino acid) and position 34 (lysine to

Protocol v 3 consol | 17 of 145

EudraCT no.: 2018-002589-38

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


arginine) and acylation of the peptide backbone with a spacer and C-18 fatty di-acid chain to lysine in position 26<sup>16</sup>. The fatty di-acid side chain and the spacer mediate strong binding to albumin, thereby reducing renal clearance. The amino acid substitution at position 8 makes semaglutide less susceptible to degradation by dipeptidyl peptidase-4 (DPP-4). The change in position 34 from a lysine to an arginine is included to have only one lysine in the sequence whereto a spacer can be attached.

Semaglutide is in development for oral once-daily treatment of T2D. As the bioavailability of GLP-1 RAs is low when administered orally, semaglutide has been co-formulated with the absorption-enhancing excipient sodium N-[8-(2-hydroxybenzoyl) amino]caprylate (SNAC) to increase the bioavailability of semaglutide. The absorption-enhancing properties of SNAC co-formulation are based on the Eligen<sup>®</sup> Carrier concept developed by Emisphere Technologies Inc.

SNAC facilitates the absorption of semaglutide in a strictly time and size dependent manner, primarily via the transcellular route. The available data for semaglutide co-formulated with SNAC support that the absorption takes place in the stomach in a localised, buffered environment in close proximity to the tablet erosion. The absorption process is hampered if dosed with food, liquid or in the presence of significant stomach content.

The absorption enhancement requires co-formulation between semaglutide and SNAC. Throughout this document "oral semaglutide" will refer to the drug product, that is, semaglutide co-formulated with 300 mg SNAC.

#### 3.1.4 Non-clinical data

#### 3.1.4.1 Semaglutide

The non-clinical programme for semaglutide was designed according to the ICH M3 guideline to support the clinical development<sup>17</sup>. The standard non-clinical data package required to support phase 3 clinical trials has been completed. In addition, 2-year carcinogenicity studies and a pre- and postnatal development toxicity study have been completed. Semaglutide was generally well tolerated in animals (mice, rats and cynomolgus monkeys). Two potential safety issues have been identified and these are detailed below.

#### **Thyroid C-cell tumours in rodents**

Treatment-related non-genotoxic proliferative changes in the thyroid C-cells of mice and rats were observed in 2-year carcinogenicity studies with semaglutide; thyroid hyperplasia was preceded by an increase in serum calcitonin. C-cell changes have not been observed in long-term studies in non-human primate. The observed pattern of effects in mice and rats and lack of these effects in the non-human primate and in man suggest that the mechanism by which semaglutide acts on the thyroid C-cells in rodents is the same as has been demonstrated for other GLP-1 RAs, including liraglutide. According to this mechanism, C-cell hyperplasia is mediated by the GLP-1 receptor and is not

Protocol v 3 consol | 18 of 145

EudraCT no.: 2018-002589-38

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


associated with RET (re-arranged during transfection) gene activation and rodents appear to be particularly sensitive, whereas humans are not. The relevance for human subjects is currently unknown, but considered to be low<sup>18</sup>.

#### Embryo-foetal development toxicity

Semaglutide caused embryo-foetal development toxicity in the rat through a GLP-1 receptor mediated effect on the inverted yolk sac placenta leading to impaired nutrient supply to the developing embryo. Primates do not have an inverted yolk sac placenta which makes this mechanism unlikely to be of relevance to humans and cynomolgus monkeys. In the developmental toxicity studies in cynomolgus monkey, a marked maternal body weight loss associated with the pharmacological effect of semaglutide coincided with increased early foetal loss; however, there was no indication of a teratogenic potential of semaglutide in this species.

A review of the results from the non-clinical studies can be found in the investigator's brochure (IB) for oral semaglutide (NN9924), or any update of this document.

#### 3.1.4.2 SNAC

SNAC was developed as an absorption-enhancing excipient for the oral route of administration. The non-clinical programme to support clinical phase 3 development and marketing authorisation application submission has been conducted including a 26-week carcinogenicity study in transgenic rasH2 mice and a 2-year carcinogenicity study in Sprague-Dawley rats.

The most common observations related to oral dosing of SNAC were, depending on species, salivation, emesis and other clinical signs such as hypoactivity, lethargy, somnolence and ataxia. When SNAC was administered at high doses (200 mg/kg/day or more, depending on species) mortality has been observed in all toxicology species. The mortality is considered to be due to inhibition of cellular respiration, mainly via an inhibition of complex 1 in the electron transport chain. The mortality was found to be related to high doses of SNAC and high initial plasma concentrations of SNAC in animals. Similar plasma concentrations of SNAC have not been observed in clinical trials with oral semaglutide and are not achievable following administration of oral semaglutide tablets containing 300 mg SNAC per tablet.

The carcinogenicity studies demonstrated that SNAC was not carcinogenic to the transgenic rasH2 mouse or the Sprague-Dawley rat. The doses tested covered total exposures of SNAC in plasma (in terms of area under the curve (AUC)) of 2-fold in the mouse and up to 44-fold in the rat when compared to the mean total exposure of SNAC in humans following a clinical dose of 300 mg SNAC/day.

A review of the SNAC results from the non-clinical studies can be found in the IB for oral semaglutide (NN9924), or any updates hereof.

Protocol v 3 consol | 19 of 145

28 January 2019 | Novo Nordisk Protocol Date: Trial ID: NN9924-4309 Version: 3.0

Final

UTN: U1111-1188-1256 Status: EudraCT no.: 2018-002589-38 

#### 3.1.5 Clinical data for oral semaglutide

A comprehensive clinical pharmacology programme including 12 trials has been completed, as well as a 26-week phase 2 dose-finding trial involving more than 600 subjects with T2D.

For details on the individual trials, please see the IB for oral semaglutide (NN9924)<sup>19</sup> or any updates hereof.

#### 3.1.5.1 **Pharmacokinetics**

In the multiple-dose trial (NN9924-3991), oral semaglutide has demonstrated a long mean terminal half-life ( $t_{1/2}$ ) ranging from 153 to 161 hours (~1 week) and a median time to reach maximum observed concentration  $(t_{max})$  ranging from 1 to 2 hours in healthy subjects.

In multiple-dose pharmacokinetics trials, the exposure to oral semaglutide increased with increasing dose. Overall, the pharmacokinetic properties of semaglutide appeared similar in healthy subjects and in subjects with T2D.

Exposure to semaglutide exhibits a substantially greater dose-to-dose variation following oral administration compared to s.c. administration. However, when administered orally once-daily the pharmacokinetic properties of semaglutide, i.e. low clearance and long half-life, will limit the variation in exposure at steady state.

Data obtained following investigation of different dosing conditions for oral semaglutide have demonstrated that subjects should take the oral semaglutide tablet in the morning in a fasting state and at least 30 minutes before the first meal of the day.

Drug-drug interaction investigations have explored the effect of oral semaglutide on the exposure to lisinopril, warfarin, metformin and digoxin as well as the effect of omeprazole on oral semaglutide and SNAC. It was demonstrated that oral semaglutide did not change the exposure to lisinopril, warfarin or digoxin, but increased the exposure to metformin when taken simultaneously. The increase in exposure to metformin may be related to delayed gastric emptying caused by semaglutide as observed for other GLP-1 RAs. Based on the wide therapeutic index of metformin, the increased exposure to metformin was however not considered clinically relevant. Further, it was demonstrated that the exposure to semaglutide appeared to be slightly higher when administered with omeprazole in comparison to semaglutide alone, but the effect was not statistically significant or considered clinically relevant.

In subjects with mild to end-stage renal impairment, the exposure to semaglutide appeared similar in subjects with normal and impaired renal function, whereas the exposure to SNAC was greater in subjects with impaired renal function than in subjects with normal renal function. The C<sub>max</sub> of SNAC appeared similar in subjects with normal and impaired renal function. The renal clearance of all SNAC metabolites was decreased in subjects with renal impairment.

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

In subjects with mild to severe hepatic impairment, the exposure to semaglutide appeared to be unaffected by the degree of hepatic impairment, whereas the exposure to SNAC (in terms of both AUC and  $C_{max}$ ) was increased for subjects with hepatic impairment as compared to subjects with normal hepatic function.

All tablets of oral semaglutide contain 300 mg of SNAC regardless of the semaglutide dose. SNAC is rapidly absorbed with a median  $t_{max}$  ranging from 0.35–0.5 hours in healthy subjects and from 0.52–1.43 hours in subjects with T2D. It is extensively metabolised and no accumulation of SNAC has been observed in clinical trials.

### **3.1.5.2 Efficacy**

The efficacy of oral semaglutide in adult subjects with T2D was investigated in a 26-week phase 2 dose-finding trial (NN9924-3790). In this trial, placebo or one of the following doses of oral semaglutide were administered once-daily: 2.5, 5, 10, 20 and 40 mg.

Results from the trial showed that oral semaglutide effectively lowered glycosylated haemoglobin (HbA $_{1c}$ ) and body weight. Placebo-adjusted reductions in HbA $_{1c}$  were dose-dependent and statistically significant for all oral semaglutide treatment arms at week 26 (range: -0.40% to -1.59%). Placebo-adjusted reductions in body weight were dose-dependent and statistically significant for oral semaglutide treatment doses of 10 mg and above at week 26 (range: -3.61 kg to -6.98 kg).

#### 3.1.5.3 Safety

In the clinical trials completed so far, no unexpected safety findings have been identified for oral semaglutide administered up to 40 mg once-daily. Consistent with other GLP-1 RAs, commonly reported adverse events (AEs) included nausea and vomiting, most of them were mild to moderate in severity. In line with findings for other GLP-1 RAs, an increase in heart rate and serum levels of lipase and amylase has also been observed in subjects exposed to oral semaglutide.

In addition to the 13 completed clinical trials with oral semaglutide, SNAC has been investigated in the programme of orally administrated heparin in combination with SNAC (heparin/SNAC). The heparin/SNAC programme (Emisphere Technologies, Inc.) included 29 phase 1 trials (SNAC doses ranged from 0.172-10.5 g). In three of these trials, SNAC alone was investigated (to a maximum dose of 10.5 g). The trials covered formulation development, food effect, hepatic and renal impairment, age-effect and drug-drug interaction. The programme also included a total of three phase 2 and 3 trials in which the effects of orally delivered heparin solution (with >1.5 g SNAC three times a day) was investigated. The overall safety profile of oral semaglutide and heparin/SNAC indicates that SNAC is safe and well-tolerated.

For further details, please see the IB for oral semaglutide (NN9924)<sup>19</sup>, or any updates hereof.

Protocol v 3 consol 21 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


EudraCT no.: 2018-002589-38

# 3.1.6 Sitagliptin

The selected active comparator in this trial is sitagliptin, an oral antidiabetic drug (OAD) of the DPP-4 inhibitor class suitable for once-daily oral administration. Sitagliptin was developed by Merck & Co and has been marketed since 2006 under the trade name Januvia<sup>®</sup>. The net effects of inhibition of DPP-4 are increased insulin secretion and reduced release of glucagon<sup>20</sup>.

Further information can be obtained in the locally approved Januvia<sup>®</sup> label added (Chinese prescribing information<sup>21</sup> and EU Summary of Product Characteristics (SmPC)<sup>22</sup>)

#### 3.2 Rationale for the trial

Many patients with T2D are not in glycaemic control with the currently marketed OADs. Nevertheless, treatment with more efficacious injectable therapies such as GLP1-RAs and insulin are rarely added during the early stages of the disease. Oral semaglutide is the first GLP-1 RA in development in a tablet formulation and it has the potential of becoming a new attractive treatment option early in the treatment cascade due to its effects on both hyperglycaemia and body weight.

The purpose of the present trial is to compare three dose levels of oral semaglutide with sitagliptin, an established OAD within the drug class of DPP4-inhibitors, in terms of glycaemic control, weight loss and other efficacy and safety parameters in subjects with T2D inadequately controlled on metformin.

This trial resembles trial NN9924-4222 (PIONEER 3) in the PIONEER programme (i.e. the global clinical phase 3a development programme for oral semaglutide). The rationale for the trial is to confirm the results of PIONEER 3 in a trial mainly including subjects from China. The design has been adjusted to fulfil the requirements to support registrations of oral semaglutide in China.

Protocol v 3 consol 22 of 145

Protocol Date: 28 January 2019 Novo Nordisk

UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38 Version:3.0Status:FinalPage:23 of 120

# 4 Objectives and endpoints

### 4.1 Objectives

# 4.1.1 Primary objective

To compare the effect of three once-daily dose levels of oral semaglutide (3, 7 and 14 mg) versus sitagliptin 100 mg once-daily, both in combination with metformin, on glycaemic control in subjects with T2D.

## 4.1.2 Secondary objectives

To compare the effect of three once-daily dose levels of oral semaglutide (3, 7 and 14 mg) versus sitagliptin 100 mg once-daily, both in combination with metformin, on body weight in subjects with T2D.

To compare the safety and tolerability of three once-daily dose levels of oral semaglutide (3, 7 and 14 mg) versus situation in subjects with methods in combination with methods in subjects with T2D.

## 4.2 Endpoints

### 4.2.1 Primary endpoint

Change from baseline to week 26 in HbA<sub>1c</sub>

### 4.2.2 Secondary endpoints

# 4.2.2.1 Confirmatory secondary endpoints

Change from baseline to week 26 in body weight (kg)

### 4.2.2.2 Supportive secondary endpoints

# Supportive secondary efficacy endpoints

- Change from baseline to week 26 in:
  - Fasting plasma glucose (FPG)
  - 7 point self-measured plasma glucose (SMPG) profile
    - Mean 7-point profile
    - Mean postprandial increment (over all meals)
  - Body weight (%)
  - Body mass index (BMI)
  - Waist circumference

Protocol v 3 consol 23 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

- Fasting lipid profile (total cholesterol, low-density lipoprotein (LDL) cholesterol, very-low-density lipoprotein (VLDL) cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides, free fatty acids)
- Patient-reported outcome
  - Short Form-36 version 2 (SF-36v2<sup>TM</sup>) (acute version) health survey
- If a subject after week 26 achieves (yes/no):
  - HbA<sub>1c</sub> < 7.0 % (53 mmol/mol) (American Diabetes Association (ADA) target)
  - $HbA_{1c} \le 6.5 \%$  (48 mmol/mol) (American Association of Clinical Endocrinologists (AACE) target)
  - $HbA_{1c}$  reduction  $\geq 1$  %-point (10.9 mmol/mol)
  - Body weight loss  $\geq 3 \%$
  - Body weight loss  $\geq 5 \%$
  - Body weight loss  $\geq 10 \%$
  - ${\rm HbA_{1c}}$  < 7.0 % (53 mmol/mol) without hypoglycaemia (treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes) and no body weight gain
  - HbA<sub>1c</sub> reduction  $\geq$  1 %-point (10.9 mmol/mol) and body weight loss  $\geq$  3 %
- Time to event:
  - Time to rescue medication

#### Supportive secondary safety endpoints

- Number of treatment-emergent adverse events (TEAEs) during exposure to trial product, assessed up to approximately 31 weeks
- Number of treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes during exposure to trial product, assessed up to approximately 31 weeks
- Treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes during exposure to trial product, assessed up to approximately 31 weeks (yes/no)
- Change from baseline to week 26 in:
  - Haematology
  - Biochemistry
  - Calcitonin
  - Pulse rate
  - Systolic blood pressure
  - Diastolic blood pressure
  - Electrocardiogram (ECG) category
  - Physical examination category
  - Eye examination category

Protocol v 3 consol | 24 of 145

28 January 2019 Novo Nordisk Protocol Date: Trial ID: NN9924-4309 Version: 30 CONFIDENTIAL UTN: U1111-1188-1256 Status: Final Page:


#### 5 Trial design

EudraCT no.: 2018-002589-38

#### 5 Type of trial

This is a 26-week, randomised, double-blinded, double-dummy, active-controlled, four-armed, parallel-group, multicentre, multinational trial comparing the efficacy and safety of three once-daily dose levels of oral semaglutide versus sitagliptin once-daily in subjects with T2D inadequately controlled on metformin.

Subjects will be randomised in a 1:1:1:1 ratio to receive one of the following treatments:

- oral semaglutide 3 mg and sitagliptin placebo
- oral semaglutide 7 mg and sitagliptin placebo
- oral semaglutide 14 mg and sitagliptin placebo
- sitagliptin 100 mg and oral semaglutide placebo

The randomisation will be stratified according to whether the subject is from the China region (including Taiwan and Hong Kong) or not.

Total trial duration for the individual subject will be up to 33 weeks. The trial includes a 2-week screening period, followed by a 26-week randomised treatment period and a follow-up period of 5 weeks. The trial design is illustrated in Figure 5-1.



Figure 5 Trial Design

### Rationale for trial design

The trial has been designed as a parallel-group, four-armed trial to ensure a direct comparison between three dose levels of oral semaglutide and the active comparator sitagliptin. Subjects will be randomised between the four treatment arms and the trial will be double-blinded to minimise bias. Since oral semaglutide and situation are not visually identical a double-dummy design will be applied to maintain the blinding of the trial. Accordingly, subjects randomised to oral semaglutide will also receive sitagliptin placebo and subjects randomised to sitagliptin will also receive oral semaglutide placebo.

Protocol v 3 consol 25 of 145 
 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


Randomisation will be stratified to ensure an even distribution of the four treatment arms within

each stratum.

EudraCT no.: 2018-002589-38

The treatment duration of 26 weeks is considered adequate to evaluate the effect of oral semaglutide versus sitagliptin and furthermore, for the assessment of safety and tolerability. The 5-week follow-up period is included to allow for wash-out of semaglutide.

# 5.3 Treatment of subjects

Treatment of subjects is summarised in Table 5–1.

# Oral semaglutide treatment arm

Oral semaglutide is a long-acting GLP-1 RA to be administered orally once daily. All subjects randomised to oral semaglutide will initiate treatment with 3 mg once daily. Subjects randomised to a treatment dose of 7 and 14 mg will follow a fixed 4-week dose escalation regimen. The maintenance dose of 7 mg once daily will be reached after 4 weeks on 3 mg once daily. The maintenance dose of 14 mg once daily will be reached after 4 weeks on 3 mg, followed by 4 weeks on 7 mg once daily (Table 5–1). All dose levels, including the dose-escalation, will be blinded (see Section 9.1). To mitigate the risk of gastrointestinal (GI) AEs, it is important to follow the fixed 4-week dose-escalation intervals. The dose of oral semaglutide must not be changed during the trial once the maintenance dose has been reached. In addition, all subjects randomised to oral semaglutide will receive sitagliptin placebo once daily.

# Sitagliptin treatment arm

The selected active comparator in this trial is sitagliptin, an OAD of the DPP4-inhibitor class suitable for once-daily administration. Subjects randomised to sitagliptin will receive 100 mg once daily throughout the trial. In addition, all subjects randomised to sitagliptin will receive oral semaglutide placebo once daily.

Protocol v 3 consol | 26 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

Table 5–1 Overview – treatment of subjects

| Trial periods | | Screening | Treatment<br>period 1 | Treatment period 2 | Treatment period 3 | Follow-up |
|---|---|---|---|---|---|---|
| First visit in each period | V1 | V2 | V4 | V5 | V9 | |
| Duration of each period | 2 weeks | 4 weeks | 4 weeks | 18 weeks | 5 weeks | |
| Treatment arm | N* | | | | | |
| oral semaglutide 3 mg | 361 | Screening | 3 mg oral<br>semaglutide +<br>sitagliptin<br>placebo | 3 mg oral<br>semaglutide +<br>sitagliptin<br>placebo | 3 mg oral<br>semaglutide +<br>sitagliptin<br>placebo | Follow-up |
| oral semaglutide 7 mg | 361 | Screening | 3 mg oral<br>semaglutide +<br>sitagliptin<br>placebo | 7 mg oral<br>semaglutide +<br>sitagliptin<br>placebo | 7 mg oral<br>semaglutide +<br>sitagliptin<br>placebo | Follow-up |
| oral semaglutide 14 mg | 361 | Screening | 3 mg oral<br>semaglutide +<br>sitagliptin<br>placebo | 7 mg oral<br>semaglutide +<br>sitagliptin<br>placebo | 14 mg oral<br>semaglutide +<br>sitagliptin<br>placebo | Follow-up |
| sitagliptin 100 mg | 361 | Screening | 100 mg<br>sitagliptin +<br>oral<br>semaglutide<br>placebo | 100 mg<br>sitagliptin +<br>oral<br>semaglutide<br>placebo | 100 mg<br>sitagliptin +<br>oral<br>semaglutide<br>placebo | Follow-up |

<sup>\*</sup>N: Number of subjects planned to be randomised

In addition to the treatment subjects must continue their pre-trial dose of metformin throughout the trial (see Section 5.3.2)

#### 5.3.1 Dosing instructions

Absorption of oral semaglutide is significantly affected by food and fluid in the stomach, hence dosing should be once daily in the morning in a fasting state and at least 30 minutes before the first meal of the day. Due to the double-dummy design, subject will take one semaglutide/semaglutide placebo tablet first in the morning with up to half a glass of water(approximately 120ml/4 fluid oz).

Then after 30 minutes subject will take the sitagliptin/sitagliptin placebo tablet together with other oral medication. This is to be done once-daily, in the morning. Both tablets must be swallowed whole by the subject and must not be broken or chewed.

#### 5.3.2 Background medication

After signing the informed consent, subjects must continue their antidiabetic pre-trial background medication (metformin) throughout the entire trial. The background medication must be maintained at the same dose level as given at trial entrance and at the same frequency during the entire treatment period unless rescue medication is needed (see Section <u>6.4</u>) or a safety concern related to the background medication arises.

Protocol v 3 consol 27 of 145

| Protocol | | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | EudraCT no.: 2018-002589-38 | | CONFIDENTIAL | Page: 28 January 2019 | Novo Nordisk | Version: 3.0 | Status: Final | | CONFIDENTIAL | | CONFIDENTIAL | Page: 28 January 2019 | Novo Nordisk | Version: 3.0 | Status: Final | | CONFIDENTIAL | Page: 28 January 2019 | Novo Nordisk | Version: 3.0 | Status: Final | | CONFIDENTIAL | Page: 28 January 2019 | Novo Nordisk | Version: 3.0 | Status: Final | | CONFIDENTIAL | Page: 28 January 2019 | Novo Nordisk | Version: 3.0 | Status: Final | | CONFIDENTIAL | Page: 28 January 2019 | Novo Nordisk | Version: 3.0 | Status: Final | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | C

In addition, the background medication (metformin):

- is considered to be non-investigational medicinal product
- will not be provided by Novo Nordisk A/S unless required by local law and should be purchased or otherwise delivered to subjects in accordance with local health plans
- should be used in accordance with standard of care or local label in the individual country

# 5.4 Treatment after discontinuation of trial product

When discontinuing trial products, either at the scheduled end-of-treatment (EOT) visit (see Section 8.1.4) or if trial product is discontinued prematurely (see Section 8.1.5), the subject should be switched to a suitable marketed product at the discretion of the investigator (for Brazil only: or it will be made available according to local regulations). After discontinuation of trial product, GLP-1 RAs are not allowed before completion of the follow-up visit 5 weeks after the last date on trial product. Throughout the protocol, last date on trial product is defined as date of the subject's last dosage of trial product.

As this trial is a phase 3a trial, oral semaglutide will not be available for prescription until after marketing authorisation.

#### 5.5 Rationale for treatment

For oral semaglutide, the three dose levels (3, 7 and 14 mg), treatment initiation with the lowest dose and the 4-week dose escalation steps have been chosen based on data from the phase 2 dose-finding trial (NN9924-3790). This regimen is expected to have the optimal benefit-risk for treatment of T2D.

Sitagliptin has been chosen as the active comparator because it is an established OAD of the DPP4-inhibitor drug class.

There will be strict glycaemic rescue criteria in place to ensure acceptable glycaemic control during the trial for all treatment arms.

Protocol v 3 consol | 28 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

# 6 Trial population

# 6.1 Number of subjects

Number of subjects planned to be screened: 2063

Number of subjects planned to be randomised: 1444

For China only: 1084 subjects from the China region (including Hong Kong and Taiwan) are planned to be randomised with an approximate equal distribution across the 4 treatment arms

Number of subjects expected to complete the trial on or off trial product: 1300

# 6.2 Inclusion criteria

For an eligible subject, all inclusion criteria must be answered "yes".

- 1. Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
- 2. Male or female, age above or equal to 18 years at the time of signing informed consent.

<u>For Algeria only</u>: Male or female, age above or equal to 19 years at the time of signing informed consent.

<u>For Taiwan only</u>: Male or female, age above or equal to 20 years at the time of signing informed consent.

- 3. Diagnosed with type 2 diabetes mellitus  $\geq$  60 days prior to day of screening.
- 4. HbA<sub>1c</sub> between 7.0-10.5% (53-91 mmol/mol) (both inclusive).
- 5. Stable daily dose of metformin ( $\geq 1500$  mg or maximum tolerated dose as documented in the subject medical record)  $\geq 60$  days prior to day of screening.

The criteria will be assessed at the investigator's discretion unless otherwise stated

#### 6.3 Exclusion criteria

For an eligible subject, all exclusion criteria must be answered "no".

- 1. Known or suspected hypersensitivity to trial products or related products.
- 2. Previous participation in this trial. Participation is defined as signed informed consent.

Protocol v 3 consol | 29 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

- 3. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method. For more information on requirements, see Appendix C
- 4. Receipt of any investigational medicinal product within 90 days before screening.
- 5. Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
- 6. Family or personal history of multiple endocrine neoplasia type 2 (MEN 2) or medullary thyroid carcinoma (MTC). Family is defined as a first degree relative.
- 7. History or presence of pancreatitis (acute or chronic).
- 8. History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).
- 9. Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening and randomisation.
- 10. Subjects presently classified as being in New York Heart Association (NYHA) Class IV.
- 11. Planned coronary, carotid or peripheral artery revascularisation known on the day of screening.
- 12. Renal impairment measured as estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m<sup>2</sup> as per Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI).
- 13. Subjects with alanine aminotransferase (ALT)  $\geq$  2.5 x upper limit of the normal (ULN).
- 14. Treatment with once-weekly Glucagon-like peptide 1 (GLP-1) receptor agonist or thiazolidinedione within the past 90 days prior to the day of screening.
- 15. Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 60 days prior to the day of screening. However, short-term insulin treatment for a maximum of 14 days prior to the day of screening is allowed.
- 16. Use of non-herbal Chinese medicine or other non-herbal local medicine with unknown or unspecified content. Herbal traditional Chinese medicine or other local herbal medicines may, at the Investigator's discretion, be continued throughout the trial
- 17. Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between

Protocol v 3 consol | 30 of 145

| Protocol | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | EudraCT no.: 2018-002589-38 | Status: Final |

screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

18. Presence or history of malignant neoplasms within the past 5 years prior to the day of screening. Basal and squamous cell skin cancer and any carcinoma in-situ is allowed.

The criteria will be assessed at the investigator's discretion unless otherwise stated.

#### 6.4 Rescue criteria

Subjects with persistent and unacceptable hyperglycaemia should be offered treatment intensification. To allow time for dose escalation and to observe the expected effect of trial treatment on glycaemic parameters, rescue criteria will be applied from week 8 (visit 5) and onwards. If any of the FPG values (including fasting SMPG) exceed the limits outlined below and no intercurrent cause of the hyperglycaemia can be identified, a confirmatory FPG (at central laboratory) should be obtained by calling the subject for a re-test. If the confirmatory FPG also exceeds the value described below, the subject should be offered rescue medication (i.e. intensification of existing antidiabetic background medication and/or initiation of new antidiabetic medication):

- 14.4 mmol/L (260 mg/dL) from week 8 to end of week 13
- 13.3 mmol/L (240 mg/dL) from week 14 to EOT

It is important for trial integrity that only subjects actually needing treatment intensification (as defined above) are started on rescue medication. Subjects started on rescue medication should continue to follow the protocol-specified visit schedule. Rescue medication should be prescribed at investigators's discretion as add-on to randomised treatment and according to ADA/European Association for the Study of Diabetes guidelines<sup>23, 24</sup> (excluding GLP-1 RAs, DPP-4 inhibitors and amylin analogues) and the local label of sitagliptin.

Rescue medication and any changes hereto should be captured on the concomitant medication form in the electronic case report from (eCRF) (see Section 8.2.4).

# 6.5 Criteria for premature discontinuation of trial product

All efforts should be made to keep the subject on trial product. However, the subject may be prematurely discontinued from trial product at the discretion of the investigator due to a safety concern. For additional guidance regarding acute pancreatitis, hepatic events and hypersensitivity see Appendix B.

The subject must be prematurely discontinued from trial product if the following applies:

1. Safety concern related to trial product or unacceptable intolerability

Protocol v 3 consol | 31 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

- 2. Included in the trial in violation of the inclusion and/or exclusion criteria
- 3. Pregnancy
- 4. Intention of becoming pregnant
- 5. Simultaneous participation in another clinical trial of an approved or non-approved investigational medicinal product.
- 6. Calcitonin  $\geq 100 \text{ ng/L}$

If a criterion for premature discontinuation of trial product is met, trial product should not be reinitiated but subjects should continue with the scheduled site contacts.

See Section <u>8.1.5</u> for procedures to be performed for subjects discontinuing trial product prematurely.

#### 6.6 Withdrawal from trial

The subject may withdraw consent at will at any time. The subject's request to withdraw from the trial must always be respected. A subject who does not complete the trial is also considered withdrawn from the trial. Hence a subject is considered withdrawn if the following applies:

- Subject is lost to follow up (only to be used if there is no contact with the subject by the time of the subject's last scheduled visit (see Section 8.1.4 8.1.6.1))
- Subject withdraws consent
- Death

See Section <u>8.1.6</u> for procedures to be performed for subjects withdrawing consent.

#### 6.7 Subject replacement

Subjects who withdraw from trial or discontinue trial product prematurely will not be replaced.

### 6.8 Rationale for trial population

The trial population will include subjects with T2D, treated with stable doses of metformin for at least 60 days prior to screening, since changes in background OAD medication shortly before trial participation may potentially impact data interpretation. The HbA<sub>1c</sub> limits of 7.0-10.5% (53-91 mmol/mol) have been chosen to include subjects needing intensification of their antidiabetic treatment. The upper limit will ensure that subjects with severely dysregulated T2D are not enrolled in the trial.

Subjects with abnormal liver parameters (ALT >2.5 x ULN) will be excluded to avoid potential confounding of liver safety assessments.

Protocol v 3 consol | 32 of 145

| Protocol | | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | EudraCT no.: 2018-002589-38 | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | Page: 34 o

Subjects with moderate, severe or end-stage renal impairment will be excluded in this trial, due to restrictions in the labels of sitagliptin and metformin. The safety and efficacy of oral semaglutide in subjects with moderate renal impairment are addressed in a global phase 3a clinical trial (trial NN9924-4234).

In addition, subjects with recent cardiovascular disease (myocardial infarction (MI), stroke, hospitalisation for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening and randomisation) will be excluded to avoid potential confounding of cardiovascular safety assessments. The cardiovascular safety of oral semaglutide is investigated in a global phase 3a cardiovascular outcomes trial (trial NN9924-4221).

Overall, the eligibility criteria will allow for enrolment of a relatively broad trial population, resembling the target population in common practice.

Protocol v 3 consol 33 of 145

Protocol Date: 28 January 2019 Novo Nordisk

UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38 
 Version:
 3.0

 Status:
 Final

 Page:

# 7 Milestones

Planned duration of recruitment period (first subject first visit – last subject first visit) is 18 months.

End of trial is defined as last subject last visit.

#### **Recruitment:**

The screening and randomisation rate will be followed closely via the interactive web response system (IWRS) in order to estimate when to stop screening. All investigators will be notified immediately when the recruitment period ends, after which no further subjects may be screened and the IWRS will be closed for further screening. All subjects screened during the recruitment period and found eligible for randomisation can be randomised within the timelines specified in the flow chart (see Section 2).

#### **Trial registration:**

Information of the trial will be disclosed at clinicaltrials.gov, chinadrugtrials.org.cn and novonordisk-trials.com. According to the Novo Nordisk Code of Conduct for Clinical Trial Disclosure<sup>25</sup>, it will also be disclosed according to other applicable requirements such as those of the International Committee of Medical Journal Editors (ICMJE)<sup>26</sup>, the Food and Drug Administration Amendment Act (FDAAA)<sup>27</sup>, European Commission Requirements<sup>28,29</sup> and other relevant recommendations or regulations including requirements by China Food and Drug administration (CFDA). If a subject requests to be included in the trial via the Novo Nordisk e-mail contact at these web sites, Novo Nordisk may disclose the investigator's contact details to the subject. As a result of increasing requirements for transparency, some countries require public disclosure of investigator names and their affiliations.

Primary Completion Date is the last assessment of the primary endpoint, and is for this protocol last subject first visit + 28 weeks corresponding to Visit 8. If the last subject is withdrawn/dropout early the Primary Completion Date is the date when the last subject would have completed Visit 8. The Primary Completion Date determines the deadline for results disclosure at Clinicaltrials.gov according to FDAAA.

Protocol v 3 consol 34 of 145
Protocol Trial ID: NN9924-4309 Date: 28 January 2019 Novo Nordisk
Version: 3.0

Final


# 8 Methods and assessments

#### 8.1 Visit procedures

The following sections describe the assessments and procedures. These are also included in the flow chart (see Section  $\underline{2}$ ). Informed consent must be obtained before any trial related activity (see Section  $\underline{18.2}$ ).

All subjects must be provided with a copy of their own signed and dated informed consent form.

Refer to flowchart (see Section 2) for number and timing of visits and specific assessments to be performed.

Each subject will attend 8 site visits and 1 phone contact. It is the responsibility of the investigator to ensure that all site visits occur according to the flow chart.

Planned visits can be conducted and re-scheduled within the allowed visit window. If a visit is missed and it is not possible to re-schedule, every effort should be made to ensure information is collected at a telephone contact (within the visit window) and entered into the eCRF. Subjects will be invited for the next scheduled visit according to the visit schedule.

The investigator must keep a log of staff and a delegation of task(s) list at site. Investigator must sign the log of staff and the delegation of task(s) at site prior to the delegation of tasks.

The investigator must keep a subject screening log, a subject identification code list and a subject enrolment log. Only subjects who have signed the informed consent form should be included on the logs. The subject screening log and subject enrolment log may be combined in one log.

## 8.1.1 Screening, visit 1

At screening, subjects will be provided with a card stating that they are participating in a trial and giving contact address(es) and telephone number(s) of relevant trial site staff. Subjects should be instructed to return the card to the investigator at the last trial visit or to destroy the card after the last visit.

A screening session must be made in the IWRS. Each subject will be assigned a unique 6-digit subject number which will remain the same throughout the trial.

In- or exclusion criteria must not be ticked "Yes" or "No" in the eCRF before source data is available. In case source data is not available "Result pending" must be chosen. This is particularly relevant for lab samples and eye examination results. Once all data relating to visit 1 have been obtained, these must be reviewed, dated and signed by the investigator and/or documented in medical records to assess that the subject is eligible to continue in the trial.

Protocol v 3 consol | 35 of 145

Protocol Trial ID: NN9924-4309 Date: 28 January 2019 Version: 3.0 Novo Nordisk

UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38 CONFIDENTIAL

Date: 28 January 2019
Status: Final


## **Screening failures**

For screening failures the screening failure form in the eCRF must be completed with the reason for not continuing in the trial. Serious adverse events (SAEs) from screening failures must be transcribed by the investigator into the eCRF. Follow-up on SAEs must be carried out according to Section 12.

A screening failure session must be made in the IWRS. The casebook must be signed.

#### Re-screening

Re-screening is NOT allowed if the subject has failed one of the inclusion or exclusion criteria, this includes re-sampling if the subject has failed one of the inclusion or exclusion criteria related to laboratory parameters. However, in case laboratory samples are lost (e.g. haemolysed or displaced), re-sampling is allowed.

#### 8.1.2 Fasting visits

The subjects must attend several visits in a fasting state (see Section  $\underline{2}$ ).

Fasting for blood sampling is defined as no food or liquid within the last 8 hours prior to blood sampling, however water is allowed up until 2 hours prior to blood sampling.

Trial products must be taken after blood sampling (see Section <u>5.3.1</u> for dosing instructions). Other oral medication can be taken 30 minutes after trial products. Injectable medications can be administered after blood sampling.

In case a subject attends a fasting visit in a non-fasting state, all non-fasting measurements should be performed. The subject should return to the site in a fasting state to have the fasting blood samples done within the visit window for the relevant visit and at visit 2 before randomisation to trial product.

#### **Fasting samples:**

- FPG
- fasting lipid profile (total cholesterol, LDL cholesterol, VLDL cholesterol, HDL cholesterol, triglycerides, free fatty acids)

# 8.1.3 Randomisation and trial product administration

Eligible subjects will be randomised into one of four treatment arms. The randomisation session must be performed in the IWRS which will allocate the dispensing unit number (DUN) of trial product to be dispensed to the subject. A drug accountability session confirming dispensing of allocated trial products should also be performed when dispensing trial products.

Protocol v 3 consol | 36 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


All visit 2 assessments, including ECG, must be performed before administration of first dose of trial product. Additionally, all in- and exclusion criteria should be checked at visit 2 prior to randomisation.

Trial products (see Section 9) will be dispensed to the subject by the site, hospital pharmacy or equivalent at each site visit during the trial from randomisation to last visit before the EOT visit (see Section 2). The investigator must document that subjects are trained in the dosing instructions, according to Section 2 and 5.3.1.

Date of first administration of trial product will be captured in the eCRF.

# 8.1.4 End-of-treatment (visit 8) and Follow-up (visit 9)

Subjects, who stay on trial product throughout the trial, must attend the EOT visit (visit 8) 26 weeks after randomisation and the Follow-up visit (visit 9) 5 weeks after the last date on trial product. Visit 9 has a +3 days visit window. A completion call must be performed in the IWRS after completion of visit 8 (see Section 10).

At visit 8 the subject should be reminded about the importance of attending the follow-up visit (visit 9). Should the subject, nonetheless, miss to attend visit 9, the site should make efforts to obtain contact with the subject within the visit window.

Treatment period completion is defined as when randomised subject has received the required treatment, and attended the EOT visit (visit 8).

A trial completer is defined as a subject who attends, or is in contact with the site, at the subject's last scheduled visit. For subjects who complete treatment, the last scheduled visit is visit 9. (For subjects who discontinue trial product, see Section 8.1.5)

#### 8.1.5 Premature discontinuation of trial product and follow-up (visits 8A and 9A)

Subjects, who discontinue trial product prematurely, should attend visit 8A scheduled to take place on the day of discontinuation of trial product (+ 3 days visit window). Visit 9A should be scheduled 5 weeks (+3 days visit window) after the last date on trial product.

The primary reason for premature discontinuation of trial product must be specified in the eCRF, and final drug accountability must be performed. A treatment discontinuation session must be made in the IWRS.

If premature discontinuation of trial product is decided during a scheduled visit, the visit will be converted into a visit 8A and trial procedures must be performed accordingly.

Subjects should perform the 7-point SMPG profile and other visit 8A assessments before initiating new antidiabetic treatment.

Protocol v 3 consol | 37 of 145

| Protocol | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | Status: Final |

Page:


Subjects should continue with the originally scheduled site contacts after visit 9A and up to and including visit 8 (week 26). If necessary, in order to retain the subject in the trial, site visits can be replaced by phone contacts after visit 9A. However, if a subject is unable or unwilling to attend subsequent visit(s), the investigator should at least aim to have the subject attend the EOT visit (visit 8) (week 26) as this visit should be performed for all subjects, if at all possible (except subjects who withdraw consent (see Section 8.1.6)). It should be documented in the medical records if subject refuses to attend a visit from visit 8A and onwards.

A subject who prematurely discontinued trial product is still considered a trial completer if the subject attends or is in contact with the site, at the subject's last scheduled visit. For subjects who prematurely discontinue trial product, the last scheduled visit is visit 8 (26 weeks after the randomisation visit) (or visit 9A if it is scheduled after visit 8). The site should in due time prepare for establishing contact with the subject within the visit window of the scheduled visit 8, if the subject has agreed to attend this visit.

In summary, subjects should stay in the trial irrespective of lack of adherence to randomised treatment, lack of adherence to visit schedule, missing assessments or trial product discontinuation for any reason. Only subjects who decline any further contact with the site in relation to the trial should be considered as having withdrawn consent (for withdrawal procedures, see Section 8.1.6).

#### 8.1.6 Withdrawal

If a subject withdraws consent, the investigator must aim to undertake procedures similar to those for visit 8A as soon as possible and visit 9A should be scheduled 5 weeks (+3 days visit window) after the last date on trial product, if the subject agrees to it.

The end-of-trial form must be completed, and final drug accountability must be performed even if the subject is not able to come to the trial site. A treatment discontinuation session must be made in the IWRS. The casebook must be signed.

Although a subject is not obliged to give his/her reason(s) for withdrawing consent, the investigator must make a reasonable effort to ascertain the reason(s), while fully respecting the subject's rights. Where the reasons are obtained, the primary reason for withdrawing consent must be specified in the end-of-trial form in the eCRF.

#### 8.1.6.1 Lost to follow-up

In case contact to the subject is lost during the trial, the site should immediately undertake efforts to re-establish contact. If the subject cannot be reached (by clinic visit or phone contact) and the subject has consented to it, the site should consult the contacts provided by the subject (e.g. close relatives), relevant physicians, medical records and locator agencies (if allowed according to local law) in an attempt to regain contact with the subject or to obtain relevant safety information from other sources. Efforts to regain contact should continue until the end of the subject's last scheduled

Protocol v 3 consol | 38 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


visit: visit 9 for subjects who have completed treatment, whereas for subjects who have discontinued trial product prematurely the last visit 8 (or visit 9A if it is scheduled after visit 8). Only if contact with the subject is not regained by the end of the visit window of the last scheduled visit can the subject be considered lost to follow up (see Section 6.6).

#### 8.1.7 Investigator assessments

Review of diaries, patient-reported outcomes (PROs), laboratory reports, ECGs and eye examinations must be documented either on the documents or in the subject's medical record. The documents must be retained at the site as source documentation.

If clarification of entries or discrepancies in the diary or PRO is needed, the subject must be questioned and a conclusion made in the subject's medical record. Care must be taken not to bias the subject.

For ECGs, physical examinations and eye examinations, the evaluations must follow the categories:

- Normal
- Abnormal
  - Was the result clinically significant? (yes/no)

The evaluation should be based on investigator's judgement.

For laboratory report values outside the reference range, the investigator must specify whether the value is clinically significant or not clinically significant. All laboratory printouts must be signed and dated by the investigator prior to the following visit. The signed laboratory report is retained at the site as source documentation.

In case of abnormal clinically significant findings found as a result of screening procedures conducted at visit 1 or trial procedures revealing baseline conditions at visit 2, the investigator must state a comment in the subject's medical record and record this in the concomitant illness/medical history form in the eCRF.

The investigator or his/her delegate must collect and review the PROs and diaries for completeness and to ensure that AEs are reported.

# 8.2 Subject related information/assessments

### 8.2.1 Demography

Demography will be recorded in the eCRF at screening and consists of:

- Date of birth (according to local regulation)
- Sex
- Ethnicity (according to local regulation)
- Race (according to local regulation)

Protocol v 3 consol | 39 of 145

| Protocol | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | Status: Final |

Page:


EudraCT no.: 2018-002589-38

# 8.2.2 Diabetes history and diabetes complications

Diabetes history and diabetes complications will be recorded on a disease specific form in the eCRF at screening and consists of:

- Date of diagnosis of T2D
- Information regarding diabetes complications including date of onset
  - Diabetic retinopathy
  - Diabetic neuropathy
  - Diabetic nephropathy

Please note that macroangiopathy (including peripheral arterial disease) should be reported on the disease specific form **History of cardiovascular disease** (see Section 8.2.3).

#### 8.2.3 Concomitant illness and medical history

A **concomitant illness** is any illness that is present at the start of the trial (visit 1) or found as a result of a screening procedure or other trial procedures performed before exposure to trial product.

**Medical history** is a medical event that the subject has experienced in the past. Only relevant medical history as judged by the investigator should be reported.

The information collected for concomitant illness and medical history should include diagnosis, date of onset and date of resolution or continuation, as applicable.

The following must be recorded in the eCRF on the disease specific forms only, i.e. not on the medical history/concomitant illness form:

- **History of cardiovascular disease** (e.g. ischaemic heart disease, MI, heart failure incl. NYHA class, hypertension, stroke, peripheral arterial disease)
- History of gallbladder disease (e.g. gallstone, cholecystitis, cholecystectomy)
- **History of gastrointestinal disease** (e.g. gastroesophageal reflux disease, ulcer disease, chronic gastritis)

Any change to a concomitant illness should be recorded during the trial. A clinically significant worsening of a concomitant illness must be reported as an AE(see Section 12.2).

It must be possible to verify the subject's medical history in source documents such as subject's medical record. If a subject is not from the investigators own practice; the investigator must make reasonable effort to obtain a copy of subject's medical record from relevant party e.g. primary physician. The investigator must document any attempt to obtain external medical information by noting the date(s) when information was requested and who has been contacted.

Protocol v 3 consol | 40 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


#### 8.2.4 Concomitant medication

EudraCT no.: 2018-002589-38

A **concomitant medication** is any medication, other than the trial products, which is taken during the trial, including the screening, treatment and follow-up periods.

Details of any concomitant medication must be recorded at the first visit. Changes in concomitant medication must be recorded at each visit as they occur.

The information collected for each concomitant medication includes

- trade name or generic name
- indication
- start date and stop date or continuation
- only applicable for antidiabetic medication: total daily dose

If a change is due to an AE, then this must be reported according to Section 12. If the change influences the subject's eligibility to continue in the trial, the monitor must be informed.

### 8.2.5 Childbearing potential

It must be recorded in the eCRF whether female subjects are of childbearing potential.

Pregnancy testing must be performed on female subjects of childbearing potential as described in Section <u>8.4.7</u>. Female subjects of childbearing potential must be instructed to use highly effective contraceptive methods throughout the trial and until 5 weeks after EOT. For more information on requirements see Appendix C.

Female of non-childbearing potential is defined as:

- Female who has undergone a hysterectomy, bilateral oophorectomy or bilateral tubal ligation
- Postmenopausal defined as no menses for 12 months without an alternative medical cause
- Other medical reasons preventing childbearing potential

#### 8.2.6 Tobacco use

Details of tobacco use must be recorded at visit 1. Smoking is defined as smoking at least one cigarette or equivalent daily.

#### Smoking status:

- Never smoked
- Previous smoker, smoking stop date
- Current smoker

Protocol v 3 consol | 41 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38

## 8.3 Efficacy assessments

## 8.3.1 Laboratory assessments for efficacy

For overall laboratory process see Section 8.5.

Blood samples will be drawn according to flow chart (see Section 2) and will be analysed at the central laboratory to determine levels of the following efficacy laboratory parameters (for fasting see Section 8.1.2):

#### Glucose metabolism:

- HbA<sub>1c</sub>
- FPG

#### Fasting lipid profile:

- Total cholesterol
- LDL cholesterol
- VLDL cholesterol
- HDL cholesterol
- Triglycerides
- Free fatty acids

#### Fasting plasma glucose

FPG is measured at the central laboratory in order to evaluate glycaemic control. The subject must attend these visits fasting (see Section 8.1.2).

A central laboratory FPG result  $\leq$  3.9 mmol/L (70 mg/dL) in relation to planned fasting visits should not be reported as a hypoglycaemic episode but as a clinical laboratory adverse event (CLAE) at the discretion of the investigator (see Section 12.1.1).

#### 8.3.2 Self-measured plasma glucose (SMPG)

At visit 1 subjects will be provided with a BG meter including auxiliaries as well as instructions for use. The subjects will be instructed in how to use the device and the instructions will be repeated as necessary during the trial. In case a hypoglycaemic episode is suspected, the provided BG meter should be used for SMPG measurement.

The BG meters use test strips calibrated to plasma values. Therefore, all measurements performed with capillary blood are automatically calibrated to plasma equivalent glucose values, which will be shown on the display.

Only the BG meter provided by Novo Nordisk should be used for the measurements required in the protocol.

Protocol v 3 consol | 42 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

Subjects should be instructed in how to record the results of the SMPG values in the diaries. The record of each SMPG value should include date, time and value. All data from the diary must be transcribed into the eCRF during or following the contact. If obtained via phone and a discrepancy is later detected, between the diary and the SMPG data obtained at the phone contact, the values in the eCRF must be corrected.

Occasional review by the investigator of the values stored in the memory of the BG meter and correct reporting of these in the diary is advised in order to ensure adequacy of the data reported in the trial database.

#### 8.3.2.1 7-point self-measured plasma glucose profile

The subject will be instructed to perform a 7-point SMPG profile twice during the trial period (see Section 2) using the BG meter provided for the trial. The 7-point SMPG profile should be performed on a day where the subject does not anticipate unusual strenuous exercise. The 7-point profile should preferably be taken within a week prior to the visit.

The record of each SMPG measurement should include the following seven time points:

- before breakfast
- 90 minutes after start of breakfast
- before lunch
- 90 minutes after start of lunch
- before dinner
- 90 minutes after start of dinner
- at bedtime

#### 8.3.3 Body weight and height

**Body weight** must be measured and recorded in the eCRF in kilogram or pound (kg or lb), with one decimal (with an empty bladder, without shoes and only wearing light clothing). The body weight should be assessed on the same calibrated weighing scale equipment throughout the trial, if possible.

**Height** is measured without shoes in centimetres or inches and recorded in the eCRF to nearest ½ cm or ¼ inch.

#### **8.3.4** Waist circumference

The **waist circumference** is defined as the minimal abdominal circumference located midway between the lower rib margin and the iliac crest.

The measurement of waist circumference must be performed and recorded in the eCRF. Waist circumference is measured in the horizontal plane and rounded up or down to the nearest ½ cm or ¼

Protocol v 3 consol 43 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


inches using a non-stretchable measuring tape. The same measuring tape should be used throughout the trial.

The circumference should be measured when the subject is in a standing position, with an empty bladder and wearing light clothing. The subject should be standing, feet together with arms down their side and waist accessible. The tape should touch the skin but not compress soft tissue and twists in the tape should be avoided. The subject should be asked to breathe normally and the measurement should be taken when the subject is breathing out gently.

# 8.3.5 Patient-reported outcome questionnaire

Following PROs will be assessed:

• SF-36v2 (acute version) health survey<sup>30, 31, 32, 33, 34</sup>

The questionnaire must be completed by the subject as specified in the flow chart (see Section 2), preferably before any other trial-related activities for that visit. It takes approximately fifteen minutes to complete the questionnaire. Subjects should be given the opportunity to complete the questionnaire by themselves without interruption. The completed questionnaire must be reviewed for potential AEs and missing data while the subject is still at the site. All results from the PRO questionnaires must be transferred into the eCRF.

The questionnaire SF-36v2<sup>TM</sup> is commonly used PRO instrument, also in the T2D area.

All the questionnaires will be translated to local languages, and also be linguistically validated before being handed out to the subjects participating in the trial.

#### SF-36 acute version

SF-36v2<sup>TM</sup> acute version measures the individual overall health related quality of life on 8 domains; Physical functioning, Role physical, Bodily pain, General health, Vitality, Social functioning, Role emotional and Mental health. The acute version's questions are based on a recall period of one week. SF-36v2<sup>TM</sup> contains 36 itemsSafety assessments

#### 8.3.6 Adverse events

AEs must be reported at each visit in accordance with the procedures outlined in Section <u>12</u> and Appendix B.

# 8.3.6.1 Adverse events requiring additional data collection

For the following AEs additional data collection is required and specific event forms must be completed in the eCRF in addition to the AE form:

- Acute coronary syndrome (MI or unstable angina pectoris requiring hospitalisation)
- Acute gallstone disease
- Cerebrovascular event (stroke or transient ischaemic attack)

Protocol v 3 consol | 44 of 145

- Heart failure
- Hypersensitivity reaction
- Neoplasm (excluding thyroid neoplasm)
- Pancreatitis
- Renal Event
- Thyroid disease (including thyroid neoplasm)
- Medication error
- Lactic acidosis
- Creatine kinase (CK) > 10x ULN
- Hepatic event defined as:
  - ALT or AST > 5x ULN and total bilirubin  $\le 2x$  ULN
  - ALT or AST > 3x ULN and total bilirubin > 2x ULN\*
  - Hepatic event leading to trial product discontinuation.
- Diabetic retinopathy and related complications

See Section 12.1.4.1 and Appendix B for details about the additional information to report.

Note that additional assessments may be required according to Appendix B in case of:

- suspicion of acute pancreatitis
- suspicion of hypersensitivity reaction
- increased levels of creatine kinase
- increased levels of aminotransferase

In case any of these events fulfil the criteria for a SAE, please report accordingly (see Section 12).

#### 8.3.7 Physical examination

A physical examination will be performed by the investigator according to local procedure (see Section 2 and 8.1.7). A physical examination must include:

- General appearance
- Head, ears, eyes, nose, throat, neck
- Thyroid gland\*
- Respiratory system
- Cardiovascular system
- GI system including mouth
- Musculoskeletal system
- Central and peripheral nervous system
- Skin

Protocol v 3 consol | 45 of 145

<sup>\*</sup>Please note that in case of a hepatic event defined as ALT or AST >3 x ULN and total bilirubin >2 x ULN, where no alternative aetiology exists (Hy's law), this must be reported as an SAE using the important medical event criterion if no other seriousness criteria are applicable.

| Protocol | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | CONFIDENTIAL | Status: Final |

Page:


#### • Lymph node palpation

EudraCT no.: 2018-002589-38

\*Please note that the diagnostic evaluation of thyroid nodules should be in accordance with the American Thyroid Association Management Guidelines or any updates hereof <sup>35</sup> adapted to local treatment guidelines if applicable.

#### 8.3.8 Vital signs

#### Systolic and diastolic blood pressure

Systolic and diastolic blood pressure should be measured in a sitting position after the subject has been resting for at least 5 minutes and by using the standard clinical practice at the site. The data must be recorded in the eCRF. The actual value of the blood pressure measurement should be recorded in the eCRF (without rounding). The same equipment should be used throughout the trial.

#### Pulse rate

Pulse rate (beats per minute) must be recorded in the eCRF at site visits after the subject has been resting for 5 minutes in a sitting position.

# 8.3.9 Eye examination

Subjects with uncontrolled and potentially unstable diabetic retinopathy or maculopathy are not eligible as this indicates retinopathy that has recently progressed to a level that requires intervention or is approaching intervention, but has yet to be brought under control.

Results of an eye examination performed by an ophthalmologist or another suitably qualified health care provider (e.g. optometrist) must be available and evaluated by the investigator before randomisation to assess eligibility. The eye examination should be performed as a fundus photography (e.g. 2-field 60 degree or better, colour or red-free) or by slit-lamp biomicroscopy examination (e.g. using a pre-corneal or corneal contact lens examination) and performed with pharmacologically dilated pupils. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

If the subject had such an eye examination performed within 90 days prior to screening, the investigator may base his/her evaluation upon the results of that examination. The examination must be repeated before randomisation if the subject has experienced worsening of visual function since the last examination. If the applicable eye examination was performed before the subject signed the informed consent form, it must be documented that the reason for performing the examination was not related to this trial.

After randomisation an eye examination performed according to above must be performed as per the flowchart in section 2. The investigator should indicate the outcome of each eye examination.

Relevant findings prior to randomisation must be recorded as concomitant illness/medical history. While relevant findings occurring after randomisation should be reported as an AE.

Protocol v 3 consol | 46 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


#### 8.3.10 Electrocardiogram (12-lead)

12-lead ECG will be performed as per flowchart (see Section 2) and the assessment must be reviewed as described in Section 8.1.7 by the investigator. The baseline ECG at visit 2 must be performed before administration of first dose of trial product.

If the ECG evaluation of a baseline ECG is suggestive of a prior MI, the investigator should consider if an update of the History of cardiovascular disease form is required.

Additional ECG recordings can be performed at the investigator's site at investigator's discretion at other visits than the planned ECG visits. The reason for additional ECG assessments should be documented and an AE should be reported if applicable.

All findings suggestive of a new MI should be reported as an AE or SAE for adjudication at the investigator's discretion and according to section 12.

#### 8.3.11 Laboratory assessments for safety

For overall laboratory process see Section 8.5.

Blood samples will be drawn according to flow chart (see Section  $\underline{2}$ ) and will be analysed at the central laboratory to determine levels of the following safety laboratory parameters:

#### Haematology:

- Haemoglobin
- Haematocrit
- Leucocytes
- Thrombocytes
- Differential count (eosinophils, neutrophils, basophils, lymphocytes and monocytes)

#### Biochemistry:

- ALT
- Albumin
- Alkaline phosphatase
- Amylase
- AST
- Bilirubin, total
- Calcium, total
- Creatinine
- eGFR per CKD-EPI<sup>36</sup>
- CK
- Lipase

Protocol v 3 consol | 47 of 145

- Potassium
- Sodium
- Urea

At visit 1, only ALT, creatinine and eGFR will be measured as part of biochemistry.

#### Hormones:

Calcitonin

In case any calcitonin value at any time during the trial is  $\geq 10$  ng/L, the algorithm in Appendix A must be followed.

#### 8.3.12 Pregnancy testing

Females of childbearing potential will have a urine dip-stick pregnancy test performed at site as specified in Section  $\underline{2}$  or as required by local law. For definition of female of non-childbearing potential and contraceptive methods see Section  $\underline{8.2.5}$ 

In case a menstrual period is missed or if pregnancy is suspected between the scheduled visits, a urine pregnancy test should be performed. Investigator should instruct the subject to contact the site in case the pregnancy test is positive. At visit 2, females of childbearing potential will be provided with a urine dip-stick pregnancy test.

#### 8.3.13 Hypoglycaemic episodes

Plasma glucose (PG) should always be measured and recorded when a hypoglycaemic episode is suspected.

#### All PG values:

- $\leq 3.9 \text{ mmol/L} (70 \text{ mg/dL}) \text{ or}$
- > 3.9 mmol/L (70 mg/dL) occurring in conjunction with hypoglycaemic symptoms

should be reported in the diary according to the instructions below throughout the trial from visit 1 to end of trial by the subject. In case a subject is not able to fill in the diary, (e.g. in case of hospitalisation), then investigator should report the hypoglycaemic episode in the eCRF.

Upon onset of a hypoglycaemic episode the subject is recommended to measure PG every 15 minutes until the SMPG value is >3.9 mmol/L (70 mg/dL) and/or symptoms have been resolved in accordance with current guidelines<sup>37</sup>.

A SMPG value ≤ 3.9 mmol/L (70 mg/dL) or hypoglycaemic symptoms must trigger a hypoglycaemic episode form to be completed by the subject. Repeated SMPG measurements and/or symptoms will per default be considered as one hypoglycaemic episode until a succeeding SMPG

Protocol v 3 consol | 48 of 145

| Protocol | Date: | 28 January 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT no.: 2018-002589-38 | Page: | 49 of 120 | |

value is > 3.9 mmol/L (70 mg/dL) and/or symptoms have been resolved. One hypoglycaemic episode form is to cover these measurements and/or symptoms.

In case of several low SMPG values within the hypoglycaemic episode, the lowest value is the one that will be reported as the SMPG value for the hypoglycaemic episode but the start time of the episode will remain as the time for the first SMPG value and/or symptom.

The record should include the following information:

- Start date and time of the hypoglycaemic episode
- Stop date and time of the hypoglycaemic episode (stop time is the first time the PG value is >3.9 mmol/L (70 mg/dL) and/or symptoms have been resolved). If a stop date and time is not reported, a hypoglycaemic episode will cover a period of 60 minutes.
- The PG level before treating the episode (if available) and any follow up measurements.
- The lowest value measured during the hypoglycaemic episode will be reported as the PG value for the episode, the remaining values will be kept as source data in the diary.
- Whether the episode was symptomatic (Yes/No)
- A hypoglycaemic episode starting without symptoms should be updated to symptomatic if the subject experiences symptoms later during the episode.
- Whether the subject was able to treat him/herself.

  If the severity of a hypoglycaemic episode aggravates, only one hypoglycaemic episode should be reported, reflecting the most severe degree of hypoglycaemia.
- Date and time of last trial product administration and for selected antidiabetic medications administered prior to the episode, date and time as well as dose must also be collected
- Date and time of last main meal (not including snacks) prior to the episode
- Whether the episode occurred in relation to physical activity
- Change in any concomitant illness
- Any sign of fever and/or other acute disease
- Whether the subject was asleep when the episode occurred
  - If yes, whether the symptoms of the episode woke up the subject

The answer to the question: "Was the subject able to treat him/herself?" must be answered "No" for an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. PG concentrations may not be available during an event, but neurological recovery following the return of PG to normal is considered sufficient evidence that the event was induced by a low PG concentration<sup>37</sup>.

Oral carbohydrates must not be given if the subject is unconscious.

Protocol v 3 consol 49 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

If the question "Was the subject able to treat him/herself?" is answered "No", the following information should be recorded by the subject:

- Who assisted in the treatment of the hypoglycaemic episode (i.e. medical person or non-medical person)?
- Where the treatment was administered (in clinic/emergency room/hospital or other. If the subject was treated in clinic/emergency room/hospital, whether they were transported in an ambulance or not)
- Type of treatment provided by another person (i.e. oral carbohydrates, glucagon, IV glucose or other)
- Were symptoms alleviated after administration of treatment?
- Factors contributing to the episode (i.e. physical activity, missed meal, diet change, medication error (i.e., mix-up between products, incorrect use of device), overdose and other factors not listed or unknown)
- Did the subject experience seizure?
- Was the subject unconscious/comatose?
- Did the subject experience any of the following symptoms<sup>38</sup>(layman term used in the diary is specified in brackets if different from the protocol term)?
  - Autonomic: sweating, trembling, hunger or palpitations (rapid or irregular heart beat)
  - Neuroglycopenic: confusion, drowsiness, speech difficulty, visual disturbances, odd behaviour, impaired balance or incoordination (reduced ability to coordinate movement)
  - General malaise: headache or malaise (feeling discomfort/unease)
- Other symptoms

The investigator must review the diary for low SMPG values not reported as hypoglycaemic episodes (see Section 2 for relevant visits). The subject must be questioned whether any of the low values were severe, i.e. whether the subject was able to self-treat or not. If the subject was not able to self-treat, it has to be reported as a severe hypoglycaemic episode on a hypoglycaemic episode form.

Low SMPG values for non-severe hypoglycaemic episodes not having a hypoglycaemic episode form completed within 7 days since the SMPG measurement should be reported on a hypoglycaemic episode form with as much information as possible. Novo Nordisk will not query for additional data except for the start date, SMPG value and whether the subject was able to self-treat due to decreased validity of such data<sup>39, 40</sup>.

The subject must be re-trained in how to report hypoglycaemic episodes if the investigator identifies low SMPG values not reported as hypoglycaemic episodes.

If the hypoglycaemic episode fulfils the criteria for an SAE then an AE form and a safety information form must also be filled in (see Section 12).

Protocol v 3 consol | 50 of 145

| Protocol | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | CONFIDENTIAL | Status: Final |

Page:


# 8.4 Laboratory assessments

The laboratory analyses will mainly be performed by a central laboratory. For some of the analyses related to suspicion of acute pancreatitis and hypersensitivity, see Appendix B.

The handling, transportation and storage of biological samples are described in the laboratory manual (for central and special laboratory details see Attachment I).

Samples will be coded in order to keep subject identity anonymous.

Laboratory samples not drawn on the day of the actual visit should preferably be drawn on another day within the visit window stated in the flow chart (see Section 2). Please note that a laboratory sample pertaining to a specific visit must always be reported to that visit.

For some of the samples drawn during the trial, subjects will be asked to attend the site visits fasting (fasting for blood sampling is defined in Section 8.1.2).

The central laboratory will provide laboratory results to the investigator on an ongoing basis.

The laboratory provides results to the trial sites in the units preferred by the trial sites while the results that are transferred to the trial database will always be in SI units.

Laboratory samples will be destroyed at the latest at the completion of the CTR, or according to local regulations.

#### 8.5 Other assessments

#### 8.5.1 Subject diary

The diaries should be handed out at the visits described in the flow chart (see Section  $\underline{2}$ ). The recordings must be reviewed as described in Section  $\underline{8.1.7}$  and transcribed to the eCRF at the following visit.

Entries in the diaries are only to be made by the subject, unless otherwise specified.

The investigator should instruct the subject in recording the following data in the diary:

- date of first trial product administration
- hypoglycaemic episodes
- changes in concomitant medication
- AEs
- SMPG 7-point profile (prior to selected site visits (see Section <u>8.3.2.1</u>))

Protocol v 3 consol | 51 of 145

Protocol Trial ID: NN9924-4309

Date: 28 January 2019 Novo Nordisk

# 8.6 Subject compliance

Throughout the trial, the investigator will remind the subjects to follow the trial procedures and requirements to ensure subject compliance.

**Treatment compliance:** Will be assessed by monitoring of drug accountability and by discussing treatment compliance and dosing conditions with the subject. The subject will be asked to return all used, partly used and unused trial product including empty packaging material during the trial as instructed by the investigator. The investigator must assess the amount of trial products returned compared to what was dispensed at the previous visit and, in case of discrepancies, question the subject. If a subject is found to be non-compliant, the investigator will remind the subject of the importance of following the instructions given including taking the trial products as prescribed and should document this discussion in the subject's medical record.

Compliance is defined as taking between 80%-120% of the dose as prescribed between visits. If the subject has been off treatment for more than 10 consecutive days, then Novo Nordisk should be contacted for guidance regarding continuation of trial medication..

Protocol v 3 consol | 52 of 145

Protocol
Trial ID: NN9924-4309


Date: 28 January 2019 Novo Nordisk

# 9 Trial supplies

Trial supplies comprise trial products and auxiliary supplies. Additional details regarding trial supplies can be found in the trial materials manual.

Trial products must not be dispensed to any person not included in the trial.

# 9.1 Trial products

The following trial products are considered as Investigational medicinal products (IMPs) and will be provided by Novo Nordisk A/S, Denmark:

Table 9-1 Trial Products

| Trial product | Strength | Dosage form | Route of administration | Container/<br>delivery device |
|---|---|---|---|---|
| Semaglutide 3 mg tablet (IMP, test product) | 3 mg | | | |
| Semaglutide 7 mg tablet (IMP, test product) | 7 mg | Tablet | Oral | Dosepack |
| Semaglutide 14 mg tablet (IMP, test product) | 14 mg | | | - |
| Semaglutide placebo tablet (IMP, reference therapy) | NA | | | |
| Sitagliptin (Januvia®) tablet<br>(IMP, reference therapy) | 100 mg | Tablet | Oral | Dosepack |
| Sitagliptin placebo tablet (IMP, reference therapy) | NA | | | |

One dosepack of semaglutide/placebo contains 7 tablets.

One dosepack of sitagliptin/placebo contains 14 tablets

Metformin and rescue medication are considered non-investigational medicinal products and will not be supplied by Novo Nordisk. However, during the 26-week treatment period and the 5-week follow-up period, the subjects' de-facto cost (actual patient cost, not covered by the Health Authorities/any insurance) of metformin will be reimbursed if required by local legislation or institutional review board (IRB)/independent ethics committee (IEC).

The active drug and the corresponding placebo are identical with regard to visual appearance. Furthermore, all oral semaglutide tablets are visually identical to each other, irrespective of dose

Protocol v 3 consol | 53 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


levels. Semaglutide and both placebo products are manufactured and supplied by Novo Nordisk, Denmark. Sitagliptin 100 mg is packed for use in clinical trials and supplied by Novo Nordisk, Denmark.

# 9.2 Labelling

EudraCT no.: 2018-002589-38

The trial products will be labelled in accordance with Annex 13<sup>41</sup>, local regulations and trial requirements.

Each trial site will be supplied with sufficient trial products for the trial on an on-going basis controlled by the IWRS. Trial product will be distributed to the trial sites according to enrolment and randomisation.

# 9.3 Storage

Storage conditions of the trial products are outlined in Trial Materials Manual (TMM).

The investigator must ensure that trial product is kept under proper storage conditions and record and evaluate the temperature. The investigator must inform Novo Nordisk **immediately** if any trial product has been stored outside specified conditions (e.g. outside temperature range). Additional details regarding handling of temperature deviations can be found in the trial materials manual.

Trial product that has been stored improperly must not be dispensed to any subject before it has been evaluated and approved for further use by Novo Nordisk. The investigator must take appropriate action to ensure correct storage.

# 9.4 Drug accountability and destruction

Drug accountability of all trial products received at site is the responsibility of the investigator.

Subjects must be instructed to return all used, partly used and unused trial products including empty packaging material as instructed by the investigator.

Returned trial product (used/partly used and/or unused), expired or damaged trial product can be stored outside controlled temperature areas, separated from non-allocated trial product.

Non-allocated trial products including expired or damaged products must be accounted as unused at the latest at closure of the trial site.

Drug accountability is performed by using the IWRS. Drug accountability must be done on tablet level.

Destruction of trial products can be performed on an on-going basis and will be done according to local procedures after accountability is finalised and reconciled by the monitor. Destruction of products must be documented in the IWRS.

Protocol v 3 consol | 54 of 145

# 9.5 Auxiliary supplies

The following will be provided by Novo Nordisk in accordance with the trial materials manual:

• BG meter and BG meter auxiliaries

Protocol v 3 consol | 55 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

# 10 Interactive voice/web response system

A trial-specific IWRS will be set up which can be accessed at any time via the internet or telephone. Access to the IWRS must be restricted to and controlled by authorised persons.

#### IWRS is used for:

- Medication arrival
- Screening
- Screening failure
- Randomisation
- Dispensing
- Dispensing verification (when barcode scanner is used)
- Treatment discontinuation
- Completion
- Code break
- Drug accountability
- Data change

IWRS user manuals will be provided to each trial site.

Protocol v 3 consol | 56 of 145

Protocol Trial ID: NN9924-4309

Date: 28 January 2019 Novo Nordisk

# 11 Randomisation procedure and breaking of blinded codes

The trial is a double-blinded trial. A randomisation session will be carried out for all subjects using the IWRS.

At the randomisation visit (visit 2), subjects meeting all eligibility criteria will be randomised to one of four parallel treatment arms as described in Section 5.1.

Randomisation will be stratified according to whether a subject is from the China region (including Taiwan and Hong Kong) or not.

- Region:
  - China
  - Non-China

# 11.1 Breaking of blinded codes

The IWRS will notify Novo Nordisk (monitor and the Global Safety department) immediately after the code is broken.

The code for a particular subject may be broken in a medical emergency if knowing the actual treatment would influence the treatment of the subject. Whenever a code is broken the person breaking the code must print the Code Break Confirmation Notification generated by the IWRS, record the reason, and sign and date the document.

When the code is broken, the treatment allocation will be accessible to the investigator and the Novo Nordisk Global Safety department. If IWRS is not accessible at the time of code break the IWRS helpdesk should be contacted. Contact details are listed in Attachment I. If the code has been broken by investigator, the subject must discontinue treatment with trial product but be asked to continue in the trial (see Section 8.1.5). A treatment discontinuation session must be completed in IWRS.

Protocol v 3 consol | 57 of 145

Protocol Trial ID: NN9924-4309 Date: 28 January 2019 Novo Nordisk Version: 3.0

# 12 Adverse events, technical complaints and pregnancies

#### 12.1 Definitions

#### 12.1.1 Adverse event

An AE is any untoward medical occurrence in a subject administered a medicinal product, and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product.

#### An AE includes:

- A clinically significant worsening of a concomitant illness.
- A clinical laboratory adverse event (CLAE): a clinical laboratory abnormality which is clinically significant, i.e. an abnormality that suggests a disease and/or organ toxicity and is of a severity that requires active management. Active management includes active treatment or further investigations, for example change of medicine dose or more frequent follow-up due to the abnormality.

#### The following should **not** be reported as AEs:

- Pre-existing conditions, including those found as a result of screening or other trial procedures performed before exposure to trial product (pre-existing conditions should be reported as medical history or concomitant illness).
- Pre-planned procedures unless the condition for which the procedure was planned has worsened from the first trial related activity after the subject has signed the informed consent.
- Non-serious hypoglycaemia is an AE, but is reported on a hypoglycaemic episode form instead of on an AE form (see Section <u>8.4.9</u>).

The following three definitions are used when assessing an AE:

#### Severity

- **Mild** no or transient symptoms, no interference with the subject's daily activities.
- Moderate marked symptoms, moderate interference with the subject's daily activities.
- Severe considerable interference with the subject's daily activities; unacceptable.

### Causality

Relationship between an AE and the relevant trial product(s):

- Probable Good reason and sufficient documentation to assume a causal relationship.
- Possible A causal relationship is conceivable and cannot be dismissed.
- **Unlikely** The event is most likely related to aetiology other than the trial product.

Protocol v 3 consol | 58 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

#### • Final outcome

- Recovered/resolved The subject has fully recovered, or by medical or surgical treatment
  the condition has returned to the level observed at the first trial-related activity after the
  subject signed the informed consent.
- Recovering/resolving The condition is improving and the subject is expected to recover from the event. This term is only applicable if the subject has completed the trial or has died from another AE.
- Recovered/resolved with sequelae The subject has recovered from the condition, but with lasting effect due to a disease, injury, treatment or procedure. If a sequela meets an SAE criterion, the AE must be reported as an SAE.
- Not recovered/not resolved The condition of the subject has not improved and the symptoms are unchanged, or the outcome is not known.
- Fatal This term is only applicable if the subject died from a condition related to the reported AE. Outcomes of other reported AEs in a subject before he/she died should be assessed as "recovered/resolved", "recovering/resolving", "recovered/resolved with sequelae" or "not recovered/not resolved". An AE with fatal outcome must be reported as an SAE.
- Unknown This term is only applicable if the subject is lost to follow-up.

#### 12.1.2 Serious adverse event

A SAE is an AE that fulfils at least one of the following criteria:

- Death.
- A life-threatening<sup>a</sup> experience.
- In-patient hospitalisation or prolongation of existing hospitalisation.
- A persistent or significant disability or incapacity<sup>c</sup>.
- A congenital anomaly or birth defect.
- Important medical events that may not result in death, be life threatening<sup>a</sup> or require hospitalisation<sup>b</sup> may be considered an SAE when based on appropriate medical judgement they may jeopardise the subject and may require medical or surgical intervention to prevent one of the outcomes listed in the definition of SAE<sup>d</sup>.
- <sup>a.</sup> The term "life threatening" in the definition of SAE refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event which hypothetically might have caused death if it was more severe.
- b. The term "hospitalisation" is used when a subject:
  - Is admitted to a hospital or in-patient, irrespective of the duration of physical stay, or
  - Stays at the hospital for treatment or observation for more than 24 hours

Medical judgement must always be exercised, and when in doubt, the hospital contact should be regarded as a hospitalisation. Hospitalisations for administrative, trial related and social purposes do

Protocol v 3 consol 59 of 145

| Protocol | 1 | Date: | 28 January 2019 | Novo Nordisk |
|---|---|---|---|---|
| EudraCT no.: 2018-002589-38 | | Page: | 60 of 120 | |

not constitute AEs and should therefore not be reported as AEs or SAEs. Hospital admissions for surgical procedures, planned before trial inclusion, are not considered AEs or SAEs.

The following AEs must always be reported as an SAE using the important medical event criterion if no other seriousness criteria are applicable:

- suspicion of transmission of infectious agents via the trial product
- risk of liver injury defined as ALT or AST >3 x ULN and total bilirubin >2 x ULN, where no alternative aetiology exists (Hy's law)

Additional assessments should be made for events meeting the criterion of Hy's law as stated above (see Appendix B).

#### 12.1.3 Non-serious adverse event

A non-serious AE is any AE which does not fulfil the definition of an SAE.

#### 12.1.4 Medication errors

A medication error<sup>42</sup> is an unintended failure in the trial drug treatment process that leads to, or has the potential to lead to, harm to the subject, such as:

- Administration of wrong drug
   Note: Use of wrong DUN is not considered a medication error unless it results in administration of wrong drug
- Wrong route of administration.

Accidental administration of a lower or higher dose than intended. The administered dose must deviate from the intended dose to an extent where clinical consequences for the trial subject were likely to happen as judged by the investigator, although they did not necessarily occurMedication errors must be reported on an AE form and a specific event form (see Section 12.1.4.1 and Appendix B).

Protocol v 3 consol | 60 of 145

<sup>&</sup>lt;sup>c.</sup> A substantial disruption of a subject's ability to conduct normal life functions (e.g. following the event or clinical investigation the subject has significant, persistent or permanent change, impairment, damage or disruption in his/her body function or structure, physical activity and/or quality of life).

<sup>&</sup>lt;sup>d.</sup> For example intensive treatment in an emergency room or at home of allergic bronchospasm, blood dyscrasia or convulsions that do not result in hospitalisation, or development of drug dependency or drug abuse.

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

# 12.1.4.1 Misuse or abuse of trial product

Abuse and misuse of trial product must be reported as an adverse event.

Misuse is defined as:

Situations where the medicinal product is intentionally and inappropriately used not in accordance with the protocol

Abuse is defined as:

Persistent or sporadic, intentional excessive use, which is accompanied by harmful physical or psychological effects (e.g. overdose with the intention to cause harm).

Suspected primary reason for the abuse/misuse must be collected.

# 12.1.5 Adverse events requiring additional data collection

AEs requiring additional data collection are AEs where the additional data will benefit the evaluation of the product safety. A number of AEs that always require additional data collection have been pre-specified. See Appendix B for details about these events and the additional information to report.

Some events in this trial will be adjudicated by an independent external committee as described in Section 12.7.2.

<u>Table 12–1</u> lists AEs that require completion of specific event forms in the eCRFs and/or are subject to event adjudication.

Table 12-1 Adverse events requiring completion of specific event forms and/or are subject to event adjudication

| Event | Specific event form | Event<br>adjudication |
|---|---|---|
| Acute coronary syndrome (MI or unstable angina pectoris requiring hospitalisation) | Yes | Yes |
| Acute gallstone disease | Yes | No |
| Cerebrovascular event (stroke or transient ischaemic attack) | Yes | Yes |
| Heart failure | Yes | Yes (only if requiring hospitalisation) |
| Hypersensitivity reaction | Yes | No |

Protocol v 3 consol 61 of 145

| Protocol | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | EudraCT no.: 2018-002589-38 | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | Page: 62 of

| Neoplasm (excluding thyroid neoplasm) | Yes | Yes (only if malignant) |
|---|---|---|
| Thyroid disease (including thyroid neoplasm) | Yes | Yes, (only if<br>malignant thyroid<br>neoplasm or C-cell<br>hyperplasia) |
| Pancreatitis | Yes | Yes (only if acute pancreatitis) |
| Renal Event | Yes | Yes (only if acute kidney injury) |
| Death | No | Yes |
| Medication error | Yes | No |
| Abuse and misuse of trial product | Yes | No |
| Lactic acidosis | Yes | Yes |
| CK > 10x ULN | Yes | No |
| <ul> <li>Hepatic event defined as:</li> <li>ALT or AST &gt; 5x ULN and total bilirubin ≤ 2x ULN</li> <li>ALT or AST &gt; 3x ULN and total bilirubin &gt; 2x ULN*</li> <li>Hepatic event leading to trial product discontinuation.</li> </ul> | Yes | No |
| Diabetic retinopathy and related complications | Yes | No |

<sup>\*</sup> Please note that in case of a hepatic event defined as ALT or AST > 3 x ULN and total bilirubin > 2 x ULN, where no alternative aetiology exists (Hy's law), this must be reported as an SAE using the important medical event criterion if no other seriousness criteria are applicable.

For details about specific event forms, see Section 8.4.1.1, and Appendix B.

# 12.1.6 Technical complaints

A technical complaint is any written, electronic, or oral communication that alleges product (medicine or device) defects. The technical complaint may be associated with an AE, but does not concern the AE itself.

Examples of technical complaints:

- The physical or chemical appearance of trial products (e.g. discoloration, particles or contamination)
- All packaging material including labelling

Only technical complaints related to AEs will be reported in the CTR.

Protocol v 3 consol 62 of 145

Protocol Date: 28 January 2019 Novo Nordisk Version: 3.0

Final


#### 12.2 Reporting of adverse events

All events meeting the definition of an AE must be collected and reported. This includes events occurring from the first trial-related activity after the subject has signed the informed consent until the end of the post-treatment follow-up period (visit 9) for subjects on trial product OR until the end of trial (visit 8 or visit 9A, whichever comes last) for the subjects who have discontinued trial product prematurely. Events for withdrawn subjects will be collected and reported until last trial related contact with the subject. The events must be recorded in the applicable eCRF forms in a timely manner (see timelines below and

Figure 12–1 Figure 12–1).

During each contact with the trial site staff, the subject must be asked about AEs and technical complaints, for example by asking: "Have you experienced any problems since the last contact?"

All AEs, either observed by the investigator or subject, must be reported by the investigator and evaluated.

All AEs must be recorded by the investigator in the eCRF AE form. The investigator should report the diagnosis, if available. If no diagnosis is available, the investigator should record each sign and symptom as individual AEs using separate AE forms in the eCRF.

For SAEs, a safety information form (SIF) must be completed in addition to the AE form. A SIF is a form to collect supplementary clinical information. If several symptoms or diagnoses occur as part of the same clinical picture, one safety information form can be used to describe all the SAEs.

AEs requiring additional data collection must be reported using both the AE form and the specific event form. A specific event form is a form tailored to collect specific information related to the individual event. See Appendix B for details about the events and the additional information to report.

In case any of these events fulfil the criteria for seriousness in Section 12.1, then the event should be reported as serious.

Some events will undergo event adjudication by the Event Adjudication Committee (EAC), please refer to Section 12.7.2. For AEs qualifying for event adjudication, the adjudication form will also have to be completed in the eCRF. The adjudication form is a checklist of clinical data to be collected and uploaded by site to the adjudication database.

For an overview of AEs requiring additional data collection and AEs that will undergo event adjudication, please see <u>Table 12–1</u>.

Protocol v 3 consol 63 of 145

Protocol
Trial ID: NN9924-4309
UTN: U1111-1188-1256
EudraCT no.: 2018-002589-38

Date: 28 January 2019 Novo Nordisk
Status: Final


For all non-serious AEs, the applicable forms should be signed when the event is resolved or at the end of the trial at the latest.

#### **Timelines for initial reporting of AEs:**

The investigator must complete the following forms in the eCRF within the specified timelines:

• **SAEs:** The AE form **within 24 hours** and the SIF **within 5 calendar** days of the investigator's first knowledge of the SAE.

Both forms must be signed within 7 calendar days from the date the information was entered in the eCRF.

- For SAEs requiring reporting on a specific event form: In addition to the above the specific event form within 14 calendar days from the investigator's first knowledge of the AE.
- Events for Adjudication: The adjudication form should be completed within 14 calendar days of the investigator's first knowledge of the AE (see Section 12.7.2). The investigator should preferably provide the medical documentation within 4 weeks of event identification according to instructions in the event adjudication site manual.

If the eCRF is unavailable, the concerned AE information must be reported on a paper AE form and sent to Novo Nordisk by fax, e-mail or courier within the same timelines as stated above. When the eCRF becomes available again, the investigator must enter the information on the form into the eCRF.

Contact details (fax, telephone, e-mail and address) are provided in the investigator trial master file.

Protocol v 3 consol 64 of 145





Timelines are for the completion of forms from the time of investigator's awareness

AE: Adverse event SAE: Serious adverse event SIF: Safety information form

Figure 12-1 Reporting of adverse events

#### Novo Nordisk assessment of AE expectedness:

Novo Nordisk assessment of expectedness is performed according to the following reference documents:

- IB for oral Semaglutide (NN9924)<sup>43</sup>; current version and any updates thereto.
- Januvia<sup>®</sup> (sitagliptin): EU SmPC<sup>22</sup>, current version and any updates thereto.

# Reporting of trial product-related SUSARs by Novo Nordisk:

Novo Nordisk will notify the investigator of trial product-related suspected unexpected serious adverse reactions (SUSARs) in accordance with local requirements and ICH GCP44. In addition, the investigator will be informed of any trial-related SAEs that may warrant a change in any trial procedure.

In accordance with regulatory requirements, Novo Nordisk will inform the regulatory authorities, including European Medicines Agency (EMA), of trial product-related SUSARs. In addition, Novo Nordisk will inform the IRBs/IECs of trial product-related SUSARs in accordance with local requirement and ICH GCP<sup>44</sup>, unless locally this is an obligation of the investigator.

Protocol v 3 consol 65 of 145

| Protocol | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | Status: Final |

Page:


# Novo Nordisk products used as concomitant medication or non-investigational medicinal product:

If an AE is considered to have a causal relationship with a Novo Nordisk marketed product used as non-investigational medicinal product or concomitant medication in the trial, it is important that the suspected relationship is reported to Novo Nordisk, e.g. in the alternative aetiology section on the safety information form. Novo Nordisk may need to report this AE to relevant regulatory authorities.

## 12.3 Follow-up of adverse events

The investigator must record follow-up information by updating the medical records and the forms in the eCRF.

Follow-up information must be reported to Novo Nordisk according to the following:

• SAEs: All SAEs must be followed until the outcome of the event is "recovered/resolved", "recovered/resolved with sequelae" or "fatal", and until all queries have been resolved. Cases of chronic conditions, cancer or AEs ongoing at time of death (where death is due to another AE) may be closed with the outcome "recovering/resolving" or "not recovered/not resolved". Cases can be closed with the outcome of "recovering/resolving" when the subject has completed the follow-up period and is expected by the investigator to recover.

The SAE follow-up information should only include new (e.g. corrections or additional) information and must be reported **within 24 hours** of the investigator's first knowledge of the information. This is also the case for previously non-serious AEs which subsequently become SAEs.

- Non-serious AEs: Non-serious AEs must be followed until the outcome of the event is "recovering/resolving", "recovered/resolved" or "recovered/resolved with sequelae" or until the end of the follow-up period stated in the protocol, whichever comes first, and until all queries related to these AEs have been resolved. Cases of chronic conditions, cancer or AEs ongoing at time of death (where death is due to another AE) may be closed with the outcome "recovering/resolving" or "not recovered/not resolved". Cases can be closed with the outcome of "recovering/resolving" when the subject has completed the follow-up period and is expected by the investigator to recover.
- Events for adjudication: If new information becomes available for events in scope for adjudication, this must be uploaded to the adjudication database in order for the EAC to evaluate if re-adjudication is needed.

The investigator must ensure that the recording of the worst case severity and seriousness of an event is kept throughout the trial. A worsening of an unresolved AE must be reported as follow up with re-assessment of severity and/or seriousness of the event.

Protocol v 3 consol | 66 of 145

Protocol
Trial ID: NN9924-4309
UTN: U1111-1188-1256
EudraCT no.: 2018-002589-38

Date: 28 January 2019 Version: 3.0
Status: Final


Queries or follow-up requests from Novo Nordisk or event adjudication vendor must be responded to **within 14 calendar days** from the date of receipt of the request, unless otherwise specified in the follow-up request.

**SAEs after end of trial:** If the investigator becomes aware of an SAE with a suspected causal relationship to the investigational medicinal product occurring to a subject after the subject has ended the trial, the investigator should report this SAE within the same timelines as for SAEs during the trial.

# 12.4 Technical complaints and technical complaint samples

# 12.4.1 Reporting of technical complaints

All technical complaints on any of the following products:

- semaglutide 3 mg/7 mg/14 mg or placebo tablets, dose-pack
- sitagliptin 100 mg or placebo tablets, dose-pack

which occur from the time of first usage of the product until the time of the last usage of the product, must be collected and reported to Customer Complaint Center, Novo Nordisk.

Contact details (fax, e-mail and address) are provided in Attachment I to the protocol.

The investigator must assess whether the technical complaint is related to any AEs or SAEs.

Technical complaints must be reported on a separate technical complaint form:

- One technical complaint form must be completed for each affected DUN
- If DUN is not available, a technical complaint form for each code or batch number must be completed

The investigator must complete the technical complaint form in the eCRF within the following timelines of the trial site obtaining knowledge of the technical complaint:

- Technical complaint assessed as related to an SAE within 24 hours
- All other technical complaints within 5 calendar days

If the eCRF is unavailable or when reporting a technical complaint that is not subject related, the information must be provided on a paper form by fax, e-mail or courier to Customer Complaint Center, Novo Nordisk, within the same timelines as stated above. When the eCRF becomes available again, the investigator must enter the information on the technical complaint form in the eCRF.

Protocol v 3 consol | 67 of 145

Protocol Date: 28 January 2019 Novo Nordisk

#### 12.4.2 Collection, storage and shipment of technical complaint samples

The investigator must collect the technical complaint sample and all associated parts that were packed in the same and DUN and and notify the monitor within 5 calendar days of obtaining the sample at trial site. The monitor must coordinate the shipment to Customer Complaint Center, Novo Nordisk (the address is provided in Attachment I) and ensure that the sample is sent as soon as possible. A copy of the technical complaint form must be included in the shipment of the sample. If several samples are shipped in one shipment, the sample and the corresponding technical complaint form should be kept together.

The investigator must ensure that the technical complaint sample contains the code or batch number and, if available, the DUN. All parts of the DUN should be returned.

If the technical complaint sample is unobtainable, the investigator must specify on the technical complaint form why it is unobtainable.

Storage of the technical complaint sample must be done in accordance with the conditions prescribed for the product.

# 12.5 Pregnancies in female subjects

Female subjects must be instructed to notify the investigator immediately if they become pregnant during the trial. The investigator must report any pregnancy in subjects who have received trial product(s).

The investigator must follow the pregnancy until the pregnancy outcome and the newborn infant is one month of age.

The investigator must report information about the pregnancy, pregnancy outcome, and health of the newborn infant(s), as well as AEs in connection with the pregnancy, and AEs in the foetus and newborn infant.

The following must be collected and reported by the investigator to Novo Nordisk - electronically (e.g. in PDF format), or by fax or courier:

#### 1. Reporting of pregnancy information

Information about the pregnancy and pregnancy outcome/health of the newborn infant(s) has to be reported on Maternal Form 1A and 1B, respectively.

When the pregnancy outcome is abnormal (i.e. congenital anomalies, foetal death including spontaneous abortion and/or any anomalies of the foetus observed at gross examination or during autopsy), and/or when a congenital anomaly is diagnosed within the first month, further information has to be reported for the female subject on Maternal Form 2. In addition,

Protocol v 3 consol | 68 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


information from the male partner has to be reported on the Paternal Form, after an informed consent has been obtained from the male partner.

Initial reporting and follow-up information must be reported within 14 calendar days of the investigator's first knowledge of initial or follow-up information.

# 2. Reporting of AE information

The investigator has to report AEs in connection with the pregnancy as well as in the foetus and newborn infant(s). The SAEs that must be reported include abnormal outcome, such as foetal death (including spontaneous abortion), and congenital anomalies (including those observed at gross examination or during autopsy of the foetus), as well as other pregnancy complications fulfilling the criteria of an SAE.

# Forms and timelines for reporting AEs:

Non-serious AEs:

• AE form<sup>a</sup> within 14 calendar days of the investigator's first knowledge of the initial or follow-up information to the non-serious AE.

#### SAEs:

- AE form within 24 hours of the investigator's first knowledge of the SAE.
- SIF within 5 calendar days of the investigator's first knowledge of the SAE.
- **SAE follow-up information** to the AE form and/or safety information form **within 24 hours** of the investigator's first knowledge of the follow-up information.
  - <sup>a</sup> It must be clearly stated in the AE diagnosis field on the AE form if the event occurred in the subject, foetus or newborn infant. If the AE occurred in the foetus or newborn infant, the AE can only be reported on paper AE and safety information form.

Any queries or follow-up requests from Novo Nordisk to non-serious AEs, SAEs and pregnancy forms must be responded to by the investigator **within 14 calendar days** from the date of receipt of the request, unless otherwise specified in the follow-up request.

#### 12.6 Precautions and/or overdose

There are no specific antidotes to semaglutide. Treatment of an overdose should be symptomatic.

There is a potential risk of hypoglycaemia during dosing with semaglutide. The typical signs and symptoms of a non-severe hypoglycaemia include: hunger, slight headache, nausea, lightheadedness, palpitations and sweating. Symptoms of non-severe hypoglycaemia should be treated by ingestion of carbohydrates.

Severe hypoglycaemia resulting in loss of consciousness should be treated according to best available medical practise.

Protocol v 3 consol | 69 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


One case of accidental overdose of oral semaglutide was reported in the NN9924-3692 trial. The subject accidentally took the trial product twice the same day and was thus treated with 20 mg of oral semaglutide. The subject did not report any symptoms and treatment was continued without any change.

One case of accidental overdose has been reported in subjects treated with s.c. semaglutide once weekly. The subject inadvertently injected 4 mg of semaglutide instead of 0.4 mg, which corresponds to a 2.5-fold higher dose than the maximum dose included in that trial. After 4–5 hours the subject felt nauseated, vomited and had a headache. The subject was instructed to drink sufficient amounts of fluids. Symptoms had improved within one day of dosing and the subject wished to continue in the trial. No symptoms of hypoglycaemia or any other symptoms or signs were noted.

For further details please see the current edition of the IB for oral semaglutide (NN9924)<sup>43</sup>, and any updates hereof.

#### 12.7 Committees related to safety

#### 12.7.1 Novo Nordisk safety committee

Novo Nordisk will constitute an internal oral semaglutide safety committee to perform ongoing safety surveillance. The oral semaglutide safety committee may recommend unblinding of any data for further analysis, and in this case an independent ad hoc group will be established in order to maintain the blinding of the trial personnel.

#### 12.7.2 Event adjudication committee

An independent external EAC is established to perform validation of selected AEs according to predefined diagnostic criteria. The validation is based on review of pre-defined clinical data related to the specific AE. Pre-defined clinical data consist of copies of source documents collected and delivered by the investigational sites.

The EAC is composed of permanent members covering required medical specialities. EAC members must disclose any potential conflicts of interest and must be independent of Novo Nordisk.

The events are reviewed by the EAC in a blinded manner. The EAC will have no authorisations to impact on trial conduct, trial protocol or amendments.

The EAC works in accordance with written guidelines included in the EAC Charter describing in details the composition, tasks, responsibilities and work processes of the committee.

Protocol v 3 consol | 70 of 145
Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

The events outlined in <u>Table 12–2</u> have been selected for adjudication in order to obtain an external independent validation of the diagnosis. In addition, cardiovascular events are being adjudicated according to U.S. Food and Drug Administration (FDA) requirements<sup>45</sup>.

The EAC will review copies in English (translated if necessary) of medical documentation received in the adjudication packages (e.g. x-ray, ECGs, ultrasound images, discharge summaries, pathology reports and death certificates). The investigator must provide medical documentation as soon as possible, when they receive the request from Novo Nordisk or the event adjudication vendor.

The AEs for adjudication are listed in <u>Table 12–2</u>:

Protocol v 3 consol 71 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

## Table 12-2 Adverse events for adjudication

| Events | Description | Adjudication outcome |
|---|---|---|
| Death* | All-cause death | Cardiovascular death (including undetermined cause of death) Non-Cardiovascular death |
| Acute Coronary Syndrome | <ul> <li>Acute Coronary Syndrome conditions include:</li> <li>ST-elevation acute myocardial infarction (STEMI)</li> <li>Non-ST elevation acute myocardial infarction (NSTEMI)</li> <li>Silent MI</li> <li>Unstable angina pectoris (UAP) requiring hospitalisation</li> </ul> | <ul> <li>Acute myocardial<br/>infarction (STEMI or<br/>NSTEMI), silent MI</li> <li>Unstable angina pectoris<br/>requiring hospitalisation</li> </ul> |
| Cerebrovascular event | <ul> <li>Stroke<sup>46</sup> is defined as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord or retinal vascular injury as a result of haemorrhage or infarction</li> <li>Transient Ischaemic Attack (TIA) is defined as a transient episode (&lt; 24 hours) of focal neurological dysfunction caused by brain, spinal cord, or retinal ischaemia, without acute infarction</li> </ul> | Ischaemic stroke Haemorrhagic stroke Undetermined stroke TIA |
| Heart failure requiring hospitalisation | Hospitalisation with a primary diagnosis of heart failure (new episode or worsening of existing heart failure) | Heart failure requiring<br>hospitalisation |
| Acute pancreatitis | The diagnosis of acute pancreatitis requires two of the following three features: • Abdominal pain consistent with acute pancreatitis (acute onset of a persistent, severe, epigastric pain often radiating to the back) • Serum lipase activity (and/or amylase activity) at least three times greater than the ULN • Characteristic findings of acute pancreatitis on imaging | Acute pancreatitis • Mild • Moderately severe • Severe |
| Malignant neoplasm | Malignant neoplasms are defined as neoplasms in which abnormal cells divide without control and can invade nearby tissues and/or spread to other parts of the body through the blood and lymph systems Thyroid neoplasms are excluded from this event category | Malignant neoplasm |

Protocol v 3 consol | 72 of 145

| Protocol Trial ID: NN9924-4309 UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38 | Date:<br>Version:<br>Status:<br>Page: | 28 January 2019<br>3.0<br>Final<br>73 of 120 | Novo Nordisk |
|---|---|---|---|
|---|---|---|---|

| Thyroid disease, if malignant<br>thyroid neoplasm or C-cell<br>hyperplasia | <ul> <li>Malignant thyroid neoplasms are defined as</li> <li>thyroid neoplasms in which abnormal cells divide without control and can invade nearby tissues and/or spread to other parts of the body through the blood and lymph systems</li> <li>C-cell hyperplasia is defined as</li> <li>hyperplasia of the parafollicular C-cells of the thyroid gland</li> </ul> | <ul> <li>Malignant thyroid neoplasm</li> <li>C-cell hyperplasia</li> </ul> |
|---|---|---|
| Acute kidney injury | <ul> <li>Acute kidney injury<sup>47</sup> is defined as any of the following (not graded):</li> <li>Increase in serum creatinine by ≥ 0.3 mg/dL (≥ 26.5 μmol/L) within 48 hours, or</li> <li>Increase in serum creatinine to ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days, or</li> <li>Urine volume &lt; 0.5 mL/kg/h for 6 hours</li> </ul> | Acute kidney injury |
| Lactic acidosis | Lactic acidosis is characterised by increased<br>blood lactate level in association with metabolic<br>acidosis | Lactic acidosis |

<sup>\*</sup>Death is not a separate event, but an outcome

There are different processes for capturing events for adjudication:

- Direct reporting by investigator:
  - All AEs need to be assessed by the investigator if any AE category is applicable. If the selected AE category is in scope for adjudication, the relevant adjudication form for the specific event will be populated for site to complete
  - AEs with fatal outcome
- Screening:
  - All AEs will be screened by Novo Nordisk for potential missed events for adjudication and if needed, the investigator will be asked to provide additional information EAC identified events:
  - The EAC can decide to have an event adjudicated even if not initially reported as an event for adjudication by the investigator.

Event adjudication will be performed for AEs in randomised subjects including AEs with an onset date during the screening period. Event adjudication will not be performed for AEs in screening failures.

AEs for adjudication must be reported according to Section 12.2. In addition the specific adjudication form should be completed within 14 calendar days of the investigator's first knowledge of the AE, and all relevant predefined documents provided within 4 weeks according to instructions in the event adjudication site manual.

Protocol v 3 consol | 73 of 145

The assessment made by the EAC will be included in the CTR as well as the assessments made by the investigator. However, the adjudication made by the EAC, given its independent analysis of each event, will be attributed with greater importance of the two.

Protocol v 3 consol | 74 of 145

Protocol Trial ID: NN9924-4309

Date: 28 January 2019 Novo Nordisk

# 13 Case report forms

Novo Nordisk will provide a system for the eCRF. This system and support services to the system will be provided by an external supplier.

Ensure that all relevant questions are answered, and that no empty data field exists. If a test or an assessment has not been done and will not be available, or if the question is irrelevant (e.g. is not applicable), indicate this according to the data entry instructions.

The following will be provided as paper case report forms (CRFs):

Pregnancy forms

The following will be provided as paper CRFs to be used when access to the eCRF is revoked or if the eCRF is unavailable:

- AE forms
- Safety information forms
- Technical complaint forms (also to be used to report complaints that are not subject related (e.g. discovered at trial site before allocation)

On the paper CRF forms print legibly, using a ballpoint pen. Ensure that all questions are answered, and that no empty data blocks exist. Ensure that no information is recorded outside the data blocks. If a test/assessment has not been done and will not be available, indicate this by writing "ND" (not done) in the appropriate answer field in the CRF. If the question is irrelevant (e.g. is not applicable) indicate this by writing "NA" (not applicable) in the appropriate answer field. Further guidance can be obtained from the instructions in the CRF.

The investigator must ensure that all information is consistent with the source documentation. By electronically signing the casebook in the eCRF, the investigator confirms that the information in the eCRF and related forms is complete and correct.

#### 13.1 Corrections to case report forms

Corrections to the eCRF data may be made by the investigator or the investigator's delegated staff. An audit trail will be maintained in the eCRF application containing as a minimum: the old and the new data, identification of the person entering the data, date and time of the entry and reason for the correction.

If corrections are made by the investigator's delegated staff after the date the investigator has signed the casebook, the casebook must be signed and dated again by the investigator.

Protocol v 3 consol | 75 of 145

| Protocol | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | CONFIDENTIAL | Status: Final |

Page:


## 13.2 Case report form flow

EudraCT no.: 2018-002589-38

The investigator must ensure that data is recorded in the eCRF as soon as possible, preferably within 5 days after the visit. Once data has been entered, it will be available to Novo Nordisk for data verification and validation purposes.

At the end of the trial, the investigator must ensure that all remaining data have been entered into the eCRF no later than 3 days after last subject last visit at the site in order to ensure the planned lock of the database.

Site specific eCRF data (in an electronic readable format) will be provided to the trial site before access to the eCRF is revoked. This data must be retained at the trial site. When the final CTR is available, the data will be archived by Novo Nordisk A/S.

Protocol v 3 consol | 76 of 145

Protocol Trial ID: NN9924-4309 Date: 28 January 2019 Novo Nordisk

Final


# 14 Monitoring procedures

Monitoring will be conducted using a risk based approach including risk assessment, monitoring plans, centralised monitoring and visits to trial sites.

During the course of the trial, the monitor will visit the trial site to ensure that the protocol is adhered to, that all issues have been recorded, to perform source data verification and to monitor drug accountability. The first monitoring visit will be performed as soon as possible after first subject first visit at the trial site and no later than 4 weeks after. The monitoring visit intervals will depend on the outcome of the centralised monitoring of the eCRFs (remote assessment of data by Novo Nordisk), the trial site's recruitment rate and the compliance of the trial site to the protocol and Good Clinical Practice (GCP), but will not exceed 12 weeks until last subject last visit at the trial site (for sites with active subjects (defined as subjects in screening, treatment or follow-up)).

The monitor must be given direct access to all source documents (original documents, data and records). Direct access includes permission to examine, analyse, verify and reproduce any record(s) and report(s) that are important to the evaluation of the trial. If the electronic medical record does not have a visible audit trail, the investigator must provide the monitor with signed and dated printouts. In addition the relevant trial site staff should be available for discussions at monitoring visits and between monitoring visits (e.g. by telephone).

All data must be verifiable in source documentation other than the eCRF.

For all data recorded the source document must be defined in a source document agreement at each trial site. There must only be one source defined at any time for any data element.

Source data generated by the trial site can be corrected by another person than the person entering the source data if accepted by local regulations; any correction must be explained, signed and dated by the person making the correction.

The original of the completed diaries and/or PROs must not be removed from the trial site, unless they form part of the eCRF and a copy is kept at the site.

The monitor will ensure that the eCRFs are completed and that paper CRFs are collected.

The following data will be source data verified for screening failures:

- Date for obtaining informed consent.
- Screening failure date and reason
- Date of visit
- Demography (date of birth, sex and race (according to local regulation))
- Eligibility criteria
- SAEs

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

Monitors will review the subject's medical records and other source data (e.g. the diaries and PROs) to ensure consistency and/or identify omissions compared to the eCRF. If discrepancies are found, the investigator must be questioned about these.

A follow-up letter (paper or electronic) will be sent to the investigator following each monitoring visit. This should address any action to be taken.

Protocol v 3 consol | 78 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

# 15 Data management

Data management is the responsibility of Novo Nordisk. Data management may be delegated under an agreement of transfer of responsibilities to a Contract Research Organisation (CRO).

Appropriate measures, including encryption of data files containing person identifiable data, will be used to ensure confidentiality of subject data, when they are transmitted over open networks.

Data from central laboratories will be transferred electronically. In cases where data is transferred via non-secure electronic networks, data will be encrypted during transfer.

The subject and any biological material obtained from the subject will be identified by subject number and trial ID. Appropriate measures such as encryption or leaving out certain identifiers will be enforced to protect the identity of subjects in all presentations and publications as required by local, regional and national requirements.

Protocol v 3 consol | 79 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

# 16 Computerised systems

Novo Nordisk will capture and process clinical data using computerised systems that are described in Novo Nordisk Standard Operating Procedures and IT architecture documentation. The use and control of these systems are documented.

Investigators working on the trial may use their own electronic systems to capture source data.

Protocol v 3 consol | 80 of 145

Protocol Trial ID: NN9924-4309 Date: 28 January 2019 Novo Nordisk

Final


## 17 Statistical considerations

If necessary, a statistical analysis plan (SAP) may be written in addition to the protocol, including a more technical and detailed elaboration of the statistical analyses. The SAP will be finalised before database lock.

The blinding of the randomised treatments will be maintained until the database has been released for statistical analysis. No interim analyses or other analyses of unblinded data will be performed before the database is locked.

Data from all sites will be analysed and reported together.

China including Taiwan and Hong Kong will be considered as a separate region unless otherwise specified. The information regarding region (China/non-China) will be included based on country details from the IWRS.

The latest available measurement, at or prior to the randomisation visit, will be used as the baseline measurement. If no measurement(s) have been obtained, at or prior to randomisation, the baseline value will be left missing.

Laboratory values below the lower limit of quantification (LLoQ) will be set to ½LLoQ. Number of values below LLoQ by treatment and visit will be summarised if deemed relevant.

Results from a statistical analysis will as a minimum be presented by the estimated treatment contrasts for the below three comparisons with associated two-sided 95% confidence intervals and p-values corresponding to two-sided tests of no difference:

- oral semaglutide 14 mg vs. sitagliptin 100 mg
- oral semaglutide 7 mg vs. sitagliptin 100 mg
- oral semaglutide 3 mg vs. sitagliptin 100 mg

If no statistical analysis is specified, data will be presented using relevant summary statistics.

## Primary and secondary estimands

Two estimands addressing different aspects of the trial objective will be defined; a primary 'Hypothetical' estimand and a secondary 'Treatment-policy estimand:

- Primary estimand 'Hypothetical'
  - Treatment difference at week 26 for all randomised subjects if all subjects adhered to treatment and did not initiate rescue medication

The hypothetical estimand assesses the glycaemic benefit a future subject is expected to achieve if initiating and continuing treatment with oral semaglutide as compared to sitagliptin. It is considered

Protocol v 3 consol | 81 of 145

EudraCT no.: 2018-002589-38

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


a clinically relevant estimand as it provides information to treating clinicians about the expected glycaemic efficacy of oral semaglutide compared to sitagliptin for purposes of treating individual subjects. Generalisation of this estimand depends among other things on the extent to which the adherence to trial product administration in this trial reflects the behaviour of the target population. Accordingly, only data collected prior to discontinuation of trial product or initiation of rescue medication will be used to draw inference. This will avoid confounding from rescue medication.

- Secondary estimand 'Treatment-policy'
  - Treatment difference at week 26 for all randomised subjects regardless of adherence to randomised treatment and initiation of rescue medication.

The treatment policy estimand assesses the expected glycaemic benefit in a future population that results from subjects initiating treatment with oral semaglutide including potential rescue medication(s) as compared to initiating treatment with sitagliptin including potential rescue medication(s). Generalisation of this estimand depends among other things on the extent to which the use of rescue medication in this trial reflects clinical practice and the adherence to trial product administration in this trial reflects the behaviour of the target population. Accordingly, data collected regardless of discontinuation of trial product or initiation of rescue medication(s) will be used to draw inference.

The confirmation of the confirmatory hypotheses will be based on the primary analysis results for the primary estimand (hypothetical). However, to address a different aspect of the trial objective and to be able to compare the trial results with the global trial (PIONEER 3), the secondary estimand (treatment-policy) has been included as well.

#### Missing data considerations at week 26

When estimating the primary estimand, data collected after discontinuation of trial product or initiation of rescue medication(s) will be set to missing. Across treatment arms the main reasons for missing data are expected to be early treatment discontinuation due to GI AEs and initiation of rescue medication. The proportion of missing data is expected to be 20% based on the sitagliptin phase 3 trials<sup>48</sup>, the oral semaglutide phase 2 trial (NN9924-3790) that indicated that a low starting dose with gradual dose escalation diminishes GI AEs compared with more aggressive dosing regimens. Initiation of rescue medication is expected to be more frequent in the sitagliptin arm and in the oral semaglutide 3 mg arm than for the two highest dose levels of oral semaglutide. A higher proportion of subjects are expected to discontinue treatment due to AEs in the oral semaglutide 14 mg arm compared to the other treatment arms. So, overall, the frequency of missing data is expected to be similar across treatment arms.

When estimating the secondary estimand, the proportion of missing data, i.e., data that do not exist even though subjects are intended to stay in the trial regardless of treatment status and initiation of rescue medication(s) is expected to be maximum 10% based on the oral semaglutide phase 2 trial

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

(NN9924-3790). Thus, missing data will mainly be due to withdrawal from trial or lost to follow-up.

Descriptive summaries and graphical representation of extent, reason(s) for and pattern of missing data will be presented by treatment arm.

#### 17.1 Sample size calculation

The primary endpoint is change from baseline to week 26 in HbA<sub>1c</sub>. For HbA<sub>1c</sub>, both non-inferiority and superiority versus sitagliptin are planned to be tested at each dose level. The confirmatory secondary endpoint is change from baseline to week 26 in body weight (kg). For body weight, superiority versus sitagliptin is planned to be tested at each dose level. The sample size calculation is made for the primary estimand and ensures power of at least 85% for testing the below three out of the nine pre-specified confirmatory hypotheses shown in Figure 17–1. The closed testing procedure described in Bretz et al 2011<sup>49</sup> is used to control the overall type I error at a nominal two-sided 5% level. The three hypotheses are:

- HbA<sub>1c</sub> superiority of semaglutide 14 mg vs. sitagliptin 100 mg
- HbA<sub>1c</sub> superiority of semaglutide 7 mg vs. sitagliptin 100 mg
- HbA<sub>1c</sub> non-inferiority of semaglutide 3 mg vs. sitagliptin 100 mg (margin of 0.3%-point)

The statistical testing strategy is based on the following two principles:

- Within a dose level, glycaemic effect must be established in terms of HbA<sub>1c</sub> non-inferiority before testing for added benefits in terms of superiority for HbA<sub>1c</sub> and/or superiority of body weight.
- Glycaemic effect in terms of HbA<sub>1c</sub> non-inferiority must be established on all higher dose levels before continuing testing hypotheses on lower dose levels.

The sample size is calculated using the calcPower function in the R package, gMCP<sup>50</sup> using 10000 simulations. All of the nine pre-specified confirmatory tests are assumed to be independent. Since positive correlations among the tests are expected, the assumption of independence is viewed as conservative.

The sample size assumptions for treatment effects (TE), adjusted TE and the common standard deviations (SD) used across dose levels are given in <u>Table 17–1</u>. These are based on the oral semaglutide phase 2 results (NN9924-3790), sitagliptin phase 3a trial results<sup>48</sup> and supported by results from the s.c. semaglutide phase 2 trial (NN9535-1821).

An adjustment in TE will be implemented for the 20% of subjects who are expected to have missing data. The TE used in the sample size calculation will be adjusted according to a 50% smaller effect in these subjects. The adjusted treatment effect is defined as  $0.8 \times TE + 0.2 \times TE \times 0.50$ .

Protocol v 3 consol | 83 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

Table 17-1 Assumptions for sample size calculation

| Oral semaglutide vs. sitagliptin | HbA1c (%-point) | | | Body weight (kg) | | |
|---|---|---|---|---|---|---|
| Treatment dose | 14 mg | 7 mg | 3 mg | 14 mg | 7 mg | 3 mg |
| Treatment effect (TE) | -0.5 | -0.3 | -0.1 | -3.0 | -2.0 | -1.0 |
| Adjusted TE, | -0.45 | -0.27 | -0.09 | -2.7 | -1.8 | -0.9 |
| Standard deviation | 1.1 | 1.1 | 1.1 | 4.0 | 4.0 | 4.0 |

With the above assumptions, allocating 361 subjects to each of the oral semaglutide treatment arms and sitagliptin 100 mg provides 85% power to jointly confirm HbA<sub>1c</sub> superiority of oral semaglutide 14 mg vs. sitagliptin 100 mg, HbA<sub>1c</sub> superiority of semaglutide 7 mg vs. sitagliptin 100 mg and HbA<sub>1c</sub> non-inferiority of semaglutide 3 mg vs. sitagliptin 100 mg for the primary estimand. Calculated powers for selected individual hypotheses are presented in Table 17–2. In total  $4\times361=1444$  subjects are planned to be randomised. The planned number of subjects from China region (including Hong Kong and Taiwan) is about  $\frac{3}{4}$  of the total sample size equal to 1084.

Table 17-2 Calculated powers for individual hypotheses

| Statistical test | HbA₁c sup | eriority | | Body weight superiority | | rity | HbA <sub>1c</sub> non-inferiority<br>(margin = 0.3%) |
|---|---|---|---|---|---|---|---|
| Treatment dose | 14 mg | 7 mg | 3 mg | 14 mg | 7 mg | 3 mg | 3 mg |
| Power (%) | > 99 | 85 | 16 | > 99 | > 99 | 84 | > 99 |

For the secondary estimand the TE in the 10% of subjects who are expected to discontinue trial product or initiate rescue medication and for the 10% of subjects who are expected to have missing data is expected to be less compared to the primary estimand. In addition, when testing for non-inferiority, the non-inferiority margin of 0.3% for HbA $_{1c}$  is added to the imputed values for the 10% of the subjects with missing data. Assuming a 75% adjustment , the same TE and standard deviations as presented in Table 17–1, the power to jointly meet HbA $_{1c}$  superiority of oral semaglutide 14 mg vs. sitagliptin 100 mg, HbA $_{1c}$  superiority of semaglutide 7 mg vs. sitagliptin 100 mg and HbA $_{1c}$  non-inferiority of semaglutide 3 mg vs. sitagliptin 100 mg is 80% for the secondary estimand.

Protocol v 3 consol 84 of 145



Figure 17-1 Graphical illustration of the closed testing procedure

The overall significance level of  $\alpha$ =0.05 (two-sided) is initially allocated to the HbA<sub>1c</sub> non-inferiority test of semaglutide 14 mg vs. sitagliptin 100 mg. The local significance level ( $\alpha$ -local) will be reallocated if a hypothesis is confirmed according to the weight given by the directed edges between nodes (hypotheses). The sample size is based on the hypotheses in the dark boxes.

Protocol v 3 consol 85 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


#### Definition of analysis sets

EudraCT no.: 2018-002589-38

The following analysis sets will be defined:

Full analysis set (FAS): Includes all randomised subjects. Subjects in the FAS will contribute to the evaluation "as randomised".

**Safety analysis set (SAS):** Includes all subjects exposed to at least one dose of trial product. Subjects in the SAS will contribute to the evaluation based on the trial product received for the majority of the period where they were on treatment. This will be referred to as contributing to the evaluation "as treated".

Per protocol (PP) analysis set: Includes all subjects in the FAS who fulfil the following criteria:

- have not violated any inclusion criteria
- have not fulfilled any exclusion criteria
- have a baseline HbA<sub>1c</sub> measurement
- is exposed to trial product and have at least one valid HbA<sub>1c</sub> measurement while on treatment without rescue medication at or after week 14

Subjects in the PP analysis set will, as in the SAS, contribute to the analysis "as treated".

## Data selections and observation periods

Unless subjects withdraw their informed consent, data collection will continue for the full duration of the trial. The full duration of the trial is defined as up to and including:

- the follow-up visit (visit 9) for subjects on trial product
- the latest occurring visit of the EOT visit (visit 8) or the follow-up premature discontinuation visit (visit 9A), for subjects who have discontinued trial product prematurely

Subjects and data to be used in an analysis will be selected in a two-step manner:

- Firstly, subjects will be selected based on the specified analysis set
- Secondly, data points on the selected subjects from first step will be selected based on the specified observation period

## Definition of the observation periods:

**In-trial:** This observation period represents the time period where subjects are considered to be in the trial, regardless of discontinuation of trial product or initiation of rescue medication. The in-trial observation period starts at randomisation (as registered in the IWRS) and ends at the date of:

- the last direct subject-site contact, which is scheduled to take place 5 weeks after planned last dose of trial product at the follow-up visit
- withdrawal for subjects who withdraw their informed consent
- the last subject-investigator contact as defined by the investigator for subjects who are lost to follow-up

Protocol v 3 consol | 86 of 145

EudraCT no.: 2018-002589-38

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


- death for subjects who dies before any of the above

**On-treatment:** This observation period represents the time period where subjects are considered treated with the trial product. The observation period is a subset of the in-trial observation period. It starts at the date of first dose of trial product. Two slightly different end dates will be needed to cover all assessments appropriately. For adjudicated events, ECGs, eye examination category, and AEs including hypoglycaemic episodes, the observation period ends at the first date of:

- the follow-up visit (visit 9)
- the follow-up prematurely discontinuation visit (visit 9A)
- the last date on trial product + 38 days
- the end-date for the in-trial observation period

The follow-up visit is scheduled to take place 5 weeks after the last date on trial product corresponding to approximately five half-lives of oral semaglutide. The visit window for the follow-up visit is + 3 days.

For efficacy and other safety assessments (laboratory assessments, physical examination and vital signs) the observation period ends at the last date on trial product + 3 days. This will be used in order to ensure specificity to reversible effects of treatment.

**On-treatment without rescue medication:** This observation period is a subset of the ontreatment observation period, where subjects are considered treated with trial product, but have not initiated any rescue medications. Specifically it starts at date of first dose of trial product and the observation period ends at the first date of:

- the last dose of trial product +3 days
- initiation of rescue medication

The on-treatment without rescue medication observation period will be the primary observation period when estimating the primary estimand (hypothetical). The in-trial observation period will be the primary observation period when estimating the secondary estimand (treatment-policy Safety will be evaluated based on the in-trial and the on-treatment observation periods.

Data points collected outside an observation period will be treated as missing in the analysis. Baseline data will always be included in an observation period. For adjudicated events, the onset date will be the EAC adjudicated onset date.

Before data are locked for statistical analysis and the randomisation code is broken, a review of all data will take place. Any decision to exclude either a subject or single observations from the statistical analysis is the joint responsibility of the members of the Novo Nordisk study group. Exclusion of data from analyses should be used restrictively, and normally no data should be excluded from the FAS. The subjects or observations to be excluded, and the reasons for their

Protocol v 3 consol | 87 of 145

| Protocol | Date: | 28 January 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT no.: 2018-002589-38 | Page: | 88 of 120 | |

exclusion must be documented and signed by those responsible before database lock. The subjects and observations excluded from analysis sets, and the reason for this, will be described in the CTR.

#### **Confirmatory hypotheses**

For the primary  $HbA_{1c}$  endpoint and the secondary confirmatory body weight endpoint, the following three confirmatory one-sided hypotheses are planned to be tested at each dose level of oral semaglutide versus sitagliptin. Let the mean treatment difference at week 26 be defined as  $\mu$  = (oral semaglutide minus sitagliptin):

- HbA<sub>1c</sub>, non-inferiority, using a non-inferiority margin of 0.3%-point
  - $H_0$ :  $\mu \ge 0.3\%$ -point against Ha:  $\mu < 0.3$ -point%
- HbA1c superiority
  - $H_0$ :  $\mu \ge 0.0\%$ -point against Ha:  $\mu < 0.0\%$ -point
- Body weight superiority
  - $H_0$ :  $\mu \ge 0.0$  kg against Ha:  $\mu < 0.0$  kg

Operationally the hypotheses will be evaluated by two-sided tests at the 5% significance level.

#### Multiplicity and criteria for confirming hypotheses

The type I error for testing the nine confirmatory hypotheses related to the HbA<sub>1c</sub> and body weight endpoints will be preserved in the strong sense at 5% (two-sided) using the weighted Bonferroni-based closed testing procedure described in Bretz et al 2011 and outlined in Figure 17–1.

The first hypothesis to be tested is non-inferiority of  $HbA_{1c}$  at the highest dose level. It will be tested at the overall significance level (5%) while allocating 0% local significance level to the remaining of the hypotheses. For this hypothesis, and in general, if a hypothesis is confirmed, then the significance level will be reallocated according to the weight and the direction of the edges going from the confirmed hypothesis to the next hypotheses as specified in Figure 17–1. Each of the following hypotheses will be tested at their updated local significance level ( $\alpha$ -local). This process will be repeated until no further hypotheses can be confirmed.

Non-inferiority and/or superiority will be considered confirmed if the mean treatment difference is supporting the corresponding alternative hypothesis and the two-sided p-value from the primary analysis of the primary estimand is strictly below its local two-sided significance level as defined by the closed testing procedure in Figure 17–1. This is equivalent to using a one-sided p-value (nominal  $\alpha$ = 0.025) and a one-sided 2.5% overall significance level in the closed testing procedure.

Protocol v 3 consol | 88 of 145

Protocol Trial ID: NN9924-4309 Date: 28 January 2019 Version: 3.0 Novo Nordisk

UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38 Version: 3.0 Status: Final 

## 17.2 Primary endpoint

The primary endpoint is change from baseline to week 26 in HbA<sub>1c</sub>.

#### 17.2.1 Primary analysis for the primary estimand

The primary estimand will be estimated based on the FAS using post-baseline measurements up to and including week 26 from the on-treatment without rescue medication observation period. The primary analysis for the primary estimand will be a Mixed Model for Repeated Measurements (MMRM). A restricted maximum likelihood (REML) will be used. The model will include all post-baseline  $HbA_{1c}$  measurements collected at scheduled visits up to and including week 26 as dependent variables. The independent effects included in the model will be treatment and region as categorical fixed effects and baseline  $HbA_{1c}$  as a covariate, all nested within visit. An unstructured covariance matrix for  $HbA_{1c}$  measurements within the same subject will be employed, assuming measurements from different subjects are independent. For subjects who do not have post-baseline assessments for planned visits available in the on-treatment without rescue medication period, the baseline value will be carried forward to the first planned visit to ensure that all randomised subjects will contribute to the statistical analysis.

The MMRM is a well-established method that accounts for the uncertainty pertaining to missing data. This analysis assumes that the missing data mechanism is missing at random (MAR). Under this assumption, the statistical behaviour of the missing data (given the observed responses and model fixed effects and covariates) is assumed to be same as for the observed data.

## 17.2.2 Primary analysis for the secondary estimand

The secondary estimand will be estimated based on the FAS using week-26 measurements from the in-trial observation period. The primary statistical analysis will be a pattern mixture model using multiple imputation to handle missing data assuming that the missing data mechanism is MAR within the groups used for imputation. Imputation of missing data at week 26 will be done within 8 groups of subjects defined by randomised treatment arm, and whether subjects at week 26; (i) have discontinued treatment or initiated rescue medication or (ii) are still on treatment and have not initiated rescue medication. It is hereby assumed that the likely values of what the missing data would have been if available are best described by information from subjects who at week 26 are similar in terms of randomised treatment arm and treatment adherence/rescue status.

Missing values for each group will be imputed as follows:

- An analysis of covariance (ANCOVA) with region as categorical fixed effects and baseline
   HbA<sub>1c</sub> measurement as a covariate will be fitted to observed values of the change from baseline
   in HbA<sub>1c</sub> at week 26.
- The estimated parameters for location and dispersion will be used to impute 1000 values for each subject with missing week-26 data based on region as categorical and baseline HbA<sub>1c</sub>. Thus, 1000 complete data sets will be generated including observed and imputed values.

Protocol Date: 28 January 2019 Novo Nordisk

Status:

Page:

Final


UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38

For each of the 1000 (now complete) imputed data sets, the change in  $HbA_{1c}$  from baseline to week 26 will be analysed using an ANCOVA with treatment and region as categorical fixed effects and baseline  $HbA_{1c}$  as covariate. The results obtained from analysing the data sets will be combined using Rubin's rule<sup>51</sup> to draw inference.

#### Analysis used for non-inferiority versus sitagliptin at week 26:

Analysis used for superiority versus sitagliptin at week 26:

Prior to analysing the data using the same model and approach as used for superiority (see above), a value of 0.3% (the non-inferiority margin) will be added to imputed values at week 26 for the oral semaglutide treatment arms only<sup>52</sup>. For evaluating non-inferiority versus sitagliptin unadjusted two sided p-values for testing no difference from the non-inferiority margin will be presented.

## 17.2.3 Sensitivity analyses

To investigate the sensitivity of the primary analysis results, a complementary and separate analysis will be performed for the primary and secondary estimand. In line with European Medicines Agency (EMA) recommendations<sup>53</sup> and with a report from the US National Research Council<sup>54</sup>, these analyses will primarily evaluate the sensitivity of the results due to the impact of missing data. Since conservatism, i.e. avoiding bias in favour of oral semaglutide, depends on the context, separate sensitivity analyses will be made for non-inferiority and superiority testing.

The evaluation of the robustness of the primary analysis results will be based on a pattern mixture model approach using multiple imputation. The pattern mixture model sensitivity analyses aim to stress-test the primary  $HbA_{1c}$  results by changing the assumptions for the missing data in the oral semaglutide treatment arms, while maintaining the MAR data assumption for the sitagliptin Additionally a sensitivity analysis for the primary analysis will be described that is not based on the pattern mixture model approach (see Section 17.2.3.1).

#### Sensitivity analyses for the primary estimand

The estimation of the primary estimand will be repeated using a tipping-point multiple imputation analysis based on FAS using the on-treatment without rescue medication observation period:

In this sensitivity analysis, missing data will first be imputed using a sequential multiple imputation approach assuming MAR. The imputation will be done as described below:

- Intermittent missing values in the on-treatment without rescue medication observation period will be imputed using a Markov Chain Monte Carlo (MCMC) method, in order to obtain a monotone missing data pattern. This imputation is done for each treatment group separately and a 1000 copies of the data set will be generated.
- A sequential regression approach for imputing monotone missing values at planned visits will be implemented starting with the first visit after baseline and sequentially continuing to the planned end of treatment visit. For each treatment group an analysis of covariance model will

Protocol Trial ID: NN9924-4309

Date: 28 January 2019 Novo Nordisk

be used to impute missing values at each planned visit. The model will include region as categorical effect and baseline and post-baseline values prior to the visit in question as covariates.

Secondly, for all oral semaglutide treatment arms a penalty will be added to the imputed values at week 26. The approach is to gradually increase this penalty until all confirmed HbA<sub>1c</sub> conclusions from the primary analysis are reversed. For each hypothesis tested the specific value of the penalty that reverses the conclusion will be used to evaluate the robustness of the primary analysis results.

#### Sensitivity analyses for the secondary estimand

The estimation of the secondary estimand will be repeated using a tipping-point multiple imputation analysis based on FAS using the in-trial observation period. For all oral semaglutide treatment arms a penalty will be added to the imputed values at week 26 from the primary analysis for the secondary estimand. The approach is to gradually increase this penalty until all confirmed HbA<sub>1c</sub> conclusions from the primary analysis are reversed. For each hypothesis tested the specific value of the penalty that reverses the conclusion will be used to evaluate the robustness of the primary analysis results.

## 17.2.3.1 Other sensitivity analyses

• Per-protocol analysis: This sensitivity will be based on the per-protocol analysis set. Data from the on-treatment without rescue medication observation period will be analysed using the primary MMRM analysis approach for the primary estimand. This sensitivity analysis will be used to evaluate the robustness of the HbA<sub>1c</sub> non-inferiority conclusions.

#### 17.2.4 Chinese subgroup analyses

Subgroup analyses for the primary endpoint and the confirmatory secondary endpoint will be performed by region with the aim to assess the TE in China region. They will be performed in a combined model using all data similar to the main analysis of the respective parameter but with an interaction between treatment and region. In addition, the safety in China region will be assessed.

## 17.3 Secondary endpoints

#### 17.3.1 Confirmatory secondary endpoints

Change from baseline to week 26 in body weight (kg) will be a confirmatory secondary endpoint.

The primary and secondary estimands will be estimated using the same approaches as described for the primary  $HbA_{1c}$  endpoint. Body weight will only be tested for superiority. Baseline body weight will be used as a covariate instead of baseline  $HbA_{1c}$  in both the MMRM and the multiple imputation analysis models.

Protocol v 3 consol 91 of 145

Protocol
Trial ID: NN9924-4309
UTN: U1111-1188-1256
EudraCT no.: 2018-002589-38

Date: 28 January 2019 Novo Nordisk
Status: Final


Superiority will be considered confirmed if the mean treatment difference is supporting the corresponding hypothesis and the two-sided p-value from the analysis of the primary estimand is strictly below its local two-sided significance level resulting from the closed testing procedure in Figure 17–1. Sensitivity analyses similar to the ones pre-specified for testing superiority for the primary HbA<sub>1c</sub> endpoint will be made to evaluate the robustness of the body weight results.

## 17.3.2 Supportive secondary endpoints

## 17.3.2.1 Efficacy endpoints

The below supportive secondary efficacy endpoints will be evaluated for:

- the primary estimand based on FAS using the on-treatment without rescue medication observation period. For endpoints where the first planned visit falls later than 8 weeks after randomisation, the baseline will not be carried forward
- the secondary estimand based on FAS using the in-trial observation period

No sensitivity analyses are planned for these.

## Continuous efficacy endpoints

Change from baseline to week 26 in:

- FPG
- Body weight (%)
- BMI
- Waist circumference
- Fasting lipid profiles (total cholesterol, LDL cholesterol, VLDL cholesterol, HDL cholesterol, triglycerides, free fatty acids)

BMI will be calculated based on body weight and height based on the formulae: BMI kg/m<sup>2</sup> = body weight (kg)/(height (m) × height (m)) or (kg/m<sup>2</sup> = [lb/in<sup>2</sup> × 703])

Change from baseline to week 26 in the below derived endpoints from the 7-point SMPG profile:

- Mean of the 7-point profile, defined as the area under the profile, calculated using the trapezoidal method, divided by the measurement time
- Mean post prandial increment (over all meals)

The above continuous endpoints will be analysed separately using similar model approaches as for the primary endpoint with the associated baseline response as a covariate. Fasting lipid profile endpoints will be log-transformed prior to analysis with the associated log-transformed baseline value as a covariate.

Protocol v 3 consol | 92 of 145

Protocol Trial ID: NN9924-4309

Date: 28 January 2019 Novo Nordisk

UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38 Status:
Page:

3.0 Final 93 of 120

#### **Binary efficacy endpoints**

If a subject after week 26 achieves (yes/no):

- $HbA_{1c} < 7.0 \%$  (53 mmol/mol) (ADA target)
- $HbA_{1c} \le 6.5 \%$  (48 mmol/mol) (AACE target)
- Body weight loss  $\geq 5 \%$
- Body weight loss  $\geq 10 \%$
- ${\rm HbA_{1c}}$  < 7.0 % (53 mmol/mol) without hypoglycaemia ( severe or BG confirmed symptomatic hypoglycaemia) and no body weight gain
- HbA<sub>1c</sub> reduction  $\geq$  1 %-point (10.9 mmol/mol) and body weight loss  $\geq$  3 %

When addressing the treatment-policy estimand the 'without hypoglycaemia' component of the composite endpoint will also include non-treatment-emergent events of severe or BG-confirmed symptomatic hypoglycaemia as data collected regardless of discontinuation of trial product or initiation of rescue medication(s) is used.

Missing data for the above six binary endpoints will be accounted for using multiple imputation techniques. For the treatment-policy estimand the binary endpoints will be calculated as dichotomisations of the 1000 multiple imputations underlying the primary MI analysis. For the hypothetical estimand the model will be implemented using a sequential imputation approach as in the tipping-point sensitivity analysis. The binary endpoints will be derived as dichotomisations of the 1000 imputed complete data sets from the sequential imputation.

The imputed complete data sets will be analysed using a logistic regression model with treatment and region as categorical fixed effects and baseline response as covariate (i.e. baseline  $HbA_{1c}$  for binary  $HbA_{1c}$  endpoints, baseline weight for binary weight endpoints and both baseline  $HbA_{1c}$  and body weight for the binary endpoints that combines both parameters). Inference comparing treatments will be drawn using Rubin's rule<sup>51</sup>.

For the composite endpoints involving both HbA<sub>1c</sub> and body weight the imputed data sets will be combined by imputation number.

#### Time to event endpoint

- Time to additional anti-diabetic medication (to support the treatment policy estimand)
- Time to rescue medication (to support the hypothetical estimand)

**Definition of additional anti-diabetic medication:** New anti-diabetic medication and/or intensification of anti-diabetic medication initiated at or after randomisation and before (planned) end-of-treatment.

Protocol v 3 consol 93 of 145

Protocol
Trial ID: NN9924-4309
UTN: U1111-1188-1256
EudraCT no.: 2018-002589-38

Date: 28 January 2019 Novo Nordisk
Status: Final


**Definition of rescue medication:** New anti-diabetic medication and/or intensification of anti-diabetic medication initiated at or after randomisation and before last date on trial product. This is a subset of the additional anti-diabetic medication.

The following rules will be applied based on the concomitant medication data reported by the investigator, to determine whether or not the recorded anti-diabetic medication is 1. *New anti-diabetic medication* or 2. *Intensification of anti-diabetic medication* 

- 1. *New anti-diabetic medication:* Anti-diabetic medication (4th-level ATC code) that is initiated at or after randomisation and is new compared to the anti-diabetic background medication at randomisation (see above) and with a dosing duration of more than 21 days
- 2. *Intensification of anti-diabetic medication*: A more than 20% increase in the dose of anti-diabetic medication at or after randomisation as compared to the anti-diabetic medication dose at randomisation (5th-level ATC code not changed) and with a dosing duration of more than 21 days.

More than 21 days is chosen as a minimum duration for the medication to be considered as 'anti-diabetic medication'. This threshold is set to ensure that the short-term durations (i.e.  $\leq$  21 days) of anti-diabetic medication (e.g. in connection with concurrent illnesses) are not included because such intensifications are not likely to affect the effect endpoints.

#### Treatment policy estimand: Time to additional anti-diabetic medication

The treatment policy estimand is addressed for the FAS using the in-trial observation period and additional anti-diabetic medication will be considered an event regardless of whether or not subjects prematurely discontinued treatment. Time from randomisation to additional anti-diabetic medication will be analysed using a Cox proportional hazards model with treatment and stratification factor as categorical fixed effects and baseline HbA<sub>1c</sub> as a covariate. From this analysis the estimated Hazard ratios between each of the oral semaglutide dose levels and placebo together with associated two-sided 95% CIs and unadjusted two-sided p-values will be presented. The analysis aims to address the need of additional anti-diabetic medication regardless of this is due to lack of effect or tolerability. Switch to other anti-diabetic treatment is therefore also considered an event and withdrawn subjects or subject lost to follow-up will be considered as having an event on the day of withdrawal. Subjects will be censored on the day before planned end of treatment visit.

#### Hypothetical estimand: Time to rescue medication

The hypothetical estimand is addressed for the FAS using the on-treatment without rescue medication observation period. Time from first dose of trial product to initiation of rescue medication will be analysed using the same model as described above. The analysis aims to address lack of effect and only initiation of rescue medication as add-on to randomised treatment is

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


considered an event. Switch to other anti-diabetic treatment is not considered an event and as a consequence subjects will be censored on the day before date of last trial product. Potential events occurring between randomisation and first date on trial product will be included in the analysis as events at day 0, in order to count all events of rescue medication.

## 17.3.2.2 Safety endpoints

EudraCT no.: 2018-002589-38

The safety endpoints will be evaluated based on SAS using the on-treatment observation period and based on SAS using the in-trial observation period unless otherwise stated. The following endpoints are used to support the safety objectives:

#### **Adverse events**

Number of TEAEs during exposure to trial product, assessed up to approximately 31 weeks

All AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) coding.

A TEAE is defined as an AE with onset in the on-treatment observation period (see definition of observation periods in Section  $\underline{0}$ ).

TEAEs will be summarised in terms of the number of subjects with at least one event (N), the percentage of subjects with at least one event (%), the number of events (E) and the event rate per 100 patient-years of observation time (R) for the on-treatment observation period. Supportive summaries of AEs will be made for the in-trial observation period. The development over time in GI AEs will be evaluated by the use of graphical methods.

#### Other safety endpoints

Change from baseline to week 26 in:

- Amylase
- Lipase
- Pulse rate
- Systolic blood pressure
- Diastolic blood pressure

The above safety endpoints will be evaluated using the primary analysis for the primary estimand based on SAS using the on-treatment observation period and using the primary analysis for the secondary estimand based on SAS using the in-trial observation period. Endpoints will be analysed separately as described above for continuous efficacy endpoints. Results at week 26 will be presented. Amylase and lipase endpoints will be log-transformed prior to analysis with the associated log-transformed baseline value as a covariate.

Protocol v 3 consol 95 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

Page:


Change from baseline to week 26 in:

• ECG category

EudraCT no.: 2018-002589-38

- Physical examination category
- Eye examination category

•

#### Safety assessments

Change from baseline to week 26 in:

- Haematology
- Biochemistry (except for amylase and lipase)
- Calcitonin

The above safety endpoints and assessments will be summarised descriptively by treatment arm and visit. Categorical safety endpoints will be summarised as counts and relative frequencies. Calcitonin will also be presented by gender.

#### Hypoglycaemia

- Number of treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes during exposure to trial product, assessed up to approximately 31 weeks
- Treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes during exposure to trial product, assessed up to approximately 31 weeks (yes/no)

## Classification of Hypoglycaemia:

Hypoglycaemic episodes will be summarised for the SAS and the on-treatment observation period only.

<u>Treatment-emergent:</u> hypoglycaemic episodes will be defined as treatment-emergent if the onset of the episode occurs within the on-treatment observation period (see definition of observation periods in Section  $\underline{0}$ ).

Nocturnal hypoglycaemic episodes: episodes occurring between 00:01 and 05.59 both inclusive.

Hypoglycaemic episodes are classified according to the Novo Nordisk classification of hypoglycaemia and the ADA classification of hypoglycaemia (see <u>Figure 17–2</u>).

#### Novo Nordisk classification of hypoglycaemia

In normal physiology, symptoms of hypoglycaemia occur below a PG level of 3.1 mmol/L (56 mg/dL)55. Therefore, Novo Nordisk has included hypoglycaemia with PG levels below this cut-off point in the definition of BG confirmed hypoglycaemia.

Protocol v 3 consol 96 of 145

Protocol
Trial ID: NN9924-4309
UTN: U1111-1188-1256
EudraCT no.: 2018-002589-38

Date: 28 January 2019 Novo Nordisk
Status: Final


Novo Nordisk uses the following classification in addition to the ADA classification:

• Severe or BG confirmed symptomatic hypoglycaemia: An episode that is severe according to the ADA classification<sup>55</sup> or BG confirmed by a PG value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.

# ADA classification<sup>37</sup> of hypoglycaemia

- Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. PG concentrations may not be available during an event, but neurological recovery following the return of PG to normal is considered sufficient evidence that the event was induced by a low PG concentration.
- Asymptomatic hypoglycaemia: An episode not accompanied by typical symptoms of hypoglycaemia, but with a measured PG concentration ≤ 3.9 mmol/L (70 mg/dL).
- Documented symptomatic hypoglycaemia: An episode during which typical symptoms of hypoglycaemia are accompanied by a measured PG concentration ≤ 3.9 mmol/L (70 mg/dL).
- Pseudo-hypoglycaemia: An episode during which the person with diabetes reports any of the typical symptoms of hypoglycaemia with a measured PG concentration > 3.9 mmol/L (70 mg/dL) but approaching that level.
- Probable symptomatic hypoglycaemia: An episode during which symptoms of hypoglycaemia are not accompanied by a PG determination but that was presumably caused by a PG concentration ≤ 3.9 mmol/L (70 mg/dL).

Protocol v 3 consol 97 of 145



Note: Glucose measurements are performed with capillary blood calibrated to plasma equivalent glucose values PG: plasma glucose SMPG: Self-measured plasma glucose

Figure 17-2 ADA classification of hypoglycaemia

Data on treatment emergent hypoglycaemic episodes will be presented in terms of the number of subjects with at least one episode, the percentage of subjects with at least one episode (%), the total number of episodes and the episode rate per 100 patient years of observation time.

#### Analysis of severe or BG confirmed symptomatic hypoglycaemic endpoints

The number of treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes will be analysed using a negative binomial regression model with a log-link function and the logarithm of the duration of the subject's on-treatment observation period as offset. The model will include treatment and region as fixed factors and baseline HbA<sub>1c</sub> as covariate.

The binary endpoint showing whether a subject has at least one treatment emergent severe or BG confirmed symptomatic hypoglycaemic episode will be analysed using a logistic regression model with treatment and region as fixed factors and baseline HbA<sub>1c</sub> as covariate.

## 17.4 Interim analysis

No interim analyses or other analyses of unblinded data will be performed before the database is locked

Protocol v 3 consol 98 of 145

Protocol Date: 28 January 2019 Novo Nordisk

UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38 

 Date:
 28 January 2019

 Version:
 3.0

 Status:
 Final

 Page:

#### 17.5 Patient-reported outcomes

## **PRO** endpoints

Change from baseline to week 26 in:

• SF-36v2 (acute version) health survey: Scores from the 8 domains, the physical component summary score and mental component summary score

The PRO endpoints will be evaluated using the primary analysis for the primary estimand based on FAS using the on-treatment without rescue medication period and using the primary analysis for the secondary estimand based on FAS using the in-trial observation period. Scores will be analysed separately as the other continuous efficacy endpoints with the associated baseline response as a covariate.

## 17.5.1 SF-36v2® (acute version) health survey

The SF-36v2® Health Survey (SF-36v2) (acute version) instrument is a commonly used generic instrument measuring health-related quality of life (HRQoL)/general health status across disease areas including diabetes. The SF-36v2 (acute version) for adults with a 1-week recall period contains 36 items.

A total of 35 items measure eight domains of functional health and well-being as well as two component summary scores: physical functioning (10 items), role limitation due to physical health problems (4 items), bodily pain (2 items), general health perceptions (5 items), vitality (4 items), social functioning (2 items), role limitations due to emotional problems (3 items) and general mental health (5 items), mental component summary (MCS) score, physical component summary (PCS) score. There is an additional single item giving information on health change over the past week.

#### **Domain scores**

Norm-based scores (NBS) will be derived using the QualityMetric Health Outcomes<sup>™</sup> Scoring Software1 including the 2009 US general population norm. The most recent version of the QualityMetric Health Outcomes<sup>™</sup> Scoring Software available at time of licensing was used for the specific trial. Table 17–3 provides an overview of the domains. NBS standardises domain and component scores into T-scores using the means and standard deviations from the US general population. Higher scores on all domains and component summary measures (PCS and MCS) indicate better HRQoL/general health status. Item 2 (i.e. Question 2 in CRF) is not included in any score.

Protocol v 3 consol 99 of 145

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

Table 17–3 Overview of domains for SF-36v2 (acute version)

| Domain | Items numbers of items included in domain | Comment |
|---|---|---|
| Physical Functioning (PF) | Items 3a-j | |
| Role Limitations Due to Physical Health (Role-Physical; RP) | Items 4a-d | |
| Bodily Pain (BP) | Items 7, 8 | Both item scores reversed |
| General Health Perceptions (General Health; GH) | Items 1, 11a-d | Item scores 1, 11b and 11d reversed |
| Vitality (VT) | Items 9a, 9e, 9g, 9i | Item scores 9a and 9e reversed |
| Social Functioning (SF) | Items 6, 10 | Item score 6 reversed |
| Role Limitations Due To Emotional Problems (Role-<br>Emotional; RE) | Items 5a-c | |
| Mental Health (MH) | Items 9b, 9c, 9d, 9f, 9h | Item scores 9d and 9h reversed |
| Physical component summary (PCS) | NA | The PCS score is a weighted average of the 8 domain scores. |
| Mental component summary (MCS) | NA | The MCS score is also a weighted average of the 8 domain scores. Weights differ from PCS to MCS. |

Missing data at instrument level will be handled using the Maximum Data Recovery method: The method applies a value to a domain item rendered missing if at least one of the items in that domain has valid data. A domain score is considered missing if all item values in the domain are missing. PCS and MCS are calculated when at least seven of the eight domains have valid data, either actual or estimated. However, to calculate PCS, the PF domain must be one of the seven domains having valid data. Also, to calculate MCS, the MH domain must be one of the seven domains having valid data.

#### Responder threshold values

The responder threshold values, in terms of T-score points for change from baseline are defined in Table 17–4.

Table 17–4 Responder thresholds for SF-36v2 (acute version)

| Domain | Responder threshold |
|---|---|
| Physical Functioning (PF) | 4.3 |
| Role Limitations Due to Physical Health (Role-Physical; RP) | 4.0 |
| Bodily Pain (BP) | 5.5 |
| General Health Perceptions (General Health; GH) | 7.0 |
| Vitality (VT) | 6.7 |
| Social Functioning (SF) | 6.2 |
| Role Limitations Due To Emotional Problems (Role-Emotional; RE) | 4.6 |
| Mental Health (MH) | 6.7 |
| Physical component summary (PCS) | 3.8 |
| Mental component summary (MCS) | 4.6 |

Responder analyses will be based on the responder threshold values and are described in Section 17.5.2.

| Protocol | | Date: 28 January 2019 | Novo Nordisk | Version: 3.0 | UTN: U1111-1188-1256 | EudraCT no.: 2018-002589-38 | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | CONFIDENTIAL | | C

#### 17.5.2 Responder analyses

Responder analyses will be conducted for both estimands and separately for each score.

For descriptive statistics the following subject responder categorization is applied for all relevant time points and scores:

- Responder improvement: Individual change from baseline in score ≥ positive responder threshold
- Non-responder no change: Individual change from baseline in score > negative responder threshold value and < positive responder threshold value
- Non-responder worsening: Individual change from baseline in score ≤ negative responder threshold value

The following binary subject responder definition is applied for all relevant time points and scores:

- Responder: Individual change from baseline in score ≥ positive responder threshold
- Non-responder: Individual change from baseline in score < positive responder threshold

The binary responder endpoints will be analysed as the other supportive secondary binary efficacy endpoints. Estimated proportions and differences in proportions will be reported in addition to odds and odds ratios.

Protocol v 3 consol | 101 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

### 18 Ethics

#### 18.1 Benefit-risk assessment of the trial

#### 18.1.1 Risks and precautions

#### 18.1.1.1 Oral semaglutide

The non-clinical safety programme of oral semaglutide has not revealed any safety issues precluding use in humans.

The sections below describe the important identified and potential risks and precautions associated with oral semaglutide treatment. These are based on findings in non-clinical studies and clinical trials with oral semaglutide as well as other GLP-1 RAs. For each of these risks and precautions, mitigating actions have been implemented to minimise the risks for subjects enrolled in this trial.

#### **Identified risks**

#### Gastrointestinal adverse events

Consistent with findings with other GLP-1 RAs, the most frequently reported AEs in clinical trials with oral semaglutide have been GI disorders (nausea, vomiting, diarrhoea, dyspepsia and constipation). Clinical trials have indicated that a low starting dose and gradual dose escalation mitigates the risk of GI AEs. Consequently, a low starting dose and dose escalation with 4 week dose-escalation steps have been implemented in the trial.

#### **Potential risks**

#### Medullary thyroid cancer

The human relevance of the proliferative C-cell changes found in rodents treated with GLP-1 RAs is unknown, but data suggest that rodents are more sensitive to the mode of action of GLP-1 RAs for induction of C-cell tumours. However, as a precaution, subjects with a family or personal history of multiple endocrine neoplasia type 2 (MEN 2) or medullary thyroid carcinoma (MTC) will not be enrolled in the trial. During the trial, calcitonin will be measured on a regular basis, and guidance for investigators on further evaluation and action on elevated calcitonin concentrations is included in Appendix A.

#### **Acute pancreatitis**

Acute pancreatitis has been reported in subjects treated with GLP-1 RAs including oral semaglutide. As a precaution, subjects with a history of acute or chronic pancreatitis will not be enrolled in the trial. Also, subjects will be informed about the symptoms of acute pancreatitis and serum levels of lipase and amylase will be monitored throughout the trial.

Protocol v 3 consol | 102 of 145

Protocol Trial ID: NN9924-4309

Date: 28 January 2019 Novo Nordisk

#### Pancreatic cancer

Patients with T2D have an increased risk of certain types of cancer such as pancreatic cancer. There is currently no support from non-clinical studies or clinical trials or post-marketing data that GLP-1-based therapies increase the risk of pancreatic cancer. However, pancreatic cancer has been included as a separate potential risk due to the scientific debate surrounding a potential association to GLP-1-based therapies and the unknown long-term effects of stimulation of  $\beta$ -cells and suppression of  $\alpha$ -cells. Pancreatic cancer has been classified as a potential class risk of GLP-1 RAs by European Medicines Agency (EMA).

## Allergic reactions

As in the case with all protein-based pharmaceuticals, treatment with oral semaglutide may evoke allergic reactions. These may include urticaria, rash, pruritus as well as anaphylactic reactions. As a precaution, subjects with known or suspected hypersensitivity to trial product(s) or related products will not be enrolled in the trial. In addition, subjects will be instructed to contact the site staff as soon as possible for further guidance if suspicion of a hypersensitivity reaction to the trial product occurs.

## Hypoglycaemia

Based on current knowledge about the GLP-1 RA drug class, there is a risk of hypoglycaemic episodes. Hypoglycaemic episodes have mainly been observed when a GLP-1 RA is combined with sulphonylurea or insulin. The risk for development of hypoglycaemia with oral semaglutide in combination with sulphonylurea and insulin is currently unknown.

#### Acute renal impairment

In subjects treated with GLP-1 RAs, including oral semaglutide, GI AEs such as nausea, vomiting and diarrhoea may lead to significant dehydration and secondary acute renal impairment. Subjects with GI AEs are recommended to drink plenty of fluids to avoid volume depletion. Also, serum creatinine and other markers of kidney function will be monitored throughout the trial.

Impaired renal function may increase the risk of metformin-associated lactic acidosis when GLP-1 RAs are co-administered with metformin. As a precaution, serum creatinine will be measured regularly. In subjects treated with metformin who experience prolonged or severe nausea and vomiting, the investigator should monitor serum creatinine, and if clinically indicated, withhold metformin until resolution of renal dysfunction.

The use of the background medication should be used in accordance with standard of care or local label in the individual country.

Protocol v 3 consol | 103 of 145

28 January 2019 | Novo Nordisk Protocol Date: Trial ID: NN9924-4309 Version: 3.0

Final

UTN: U1111-1188-1256 Status: 104 of 120 EudraCT no.: 2018-002589-38 Page:

#### Other safety considerations

## **Diabetic retinopathy complications**

A transient worsening of diabetic retinopathy is a recognised complication in selected patients with diabetes after initiation of intensive antidiabetic treatment 56,57,58. Risk factors for these events include long-standing poor glycaemic control and presence of proliferative retinopathy, and initial large improvements in BG may be an additional aggravating factor. Several studies have, however, documented long-term beneficial effects of intensive glycaemic treatment in reducing retinopathy progression<sup>59,60</sup> even in intensively treated patients who experienced early worsening<sup>57</sup>. In a cardiovascular outcomes trial with s.c. semaglutide, results indicate an increased risk of events related to diabetic retinopathy in subjects treated with semaglutide compared to placebo<sup>61</sup>. As a precaution in this trial, all subjects are required to have a fundus photography or dilated fundoscopy performed before enrolment into the trial; moreover, subjects with proliferative retinopathy or maculopathy requiring acute treatment will be excluded. As part of good diabetes management the investigator is encouraged to ensure adequate monitoring and treatment of diabetic retinopathy in subjects enrolled into the trial<sup>62</sup>.

## **Teratogenicity (embryo-foetal development toxicity)**

Semaglutide caused embryo-foetal malformations in the rat through a GLP-1 receptor mediated effect on the inverted yolk sac placenta leading to impaired nutrient supply to the developing embryo. Primates do not have an inverted yolk sac placenta which makes this mechanism unlikely to be of relevance to humans. However, as a precaution, females who are pregnant, breast-feeding or intend to become pregnant or are of childbearing potential and not using an adequate contraceptive method will not be enrolled in the trial. In addition, pregnancy tests will be performed at all visits, including screening and follow-up and at any time during the trial if a menstrual period is missed, or as required by local law.

#### General precautions

All subjects will be included after a thorough evaluation with regards to in- and exclusion criteria defined in order to ensure that subjects are eligible for trial treatment. There are also strict glycaemic rescue criteria in place to ensure acceptable glycaemic control during the trial. If rescue medication is required, it should be in accordance with ADA/European Association for the Study of Diabetes<sup>23, 24</sup> (excluding GLP-1 RAs, DPP-4 inhibitors and amylin analogues) and the local label of sitagliptin

It is the responsibility of the investigator to ensure the best possible care according to the principles outlined in Diabetes Care 2017 Standards of Medical Care in Diabetes<sup>62</sup>. In addition to ensuring glycaemic control, appropriate risk factor modification also includes optimal treatment of hypertension, dyslipidaemia and other cardiovascular risk factors, as well as regular monitoring and treatment of diabetic kidney disease and diabetic retinopathy<sup>62</sup>.

Protocol v 3 consol 104 of 145

| Protocol | Date: | 28 January 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT no.: 2018-002589-38 | Page: | 105 of 120 | |

Further details with regards to safety of oral semaglutide are described in the current edition of the IB for oral semaglutide (NN9924)<sup>43</sup>, or any updates thereto.

#### 18.1.1.2 Sitagliptin

The most commonly reported side effects associated with sitagliptin are upper respiratory tract infection, nasopharyngitis and headache. Also acute pancreatitis, acute renal failure, hypersensitivity reactions and hypoglycaemia have been reported. Please consult the EU SmPC or locally approved label of Januvia<sup>®</sup> for information on warnings and precautions/risks<sup>48</sup>.

#### 18.1.2 Benefits

Randomised subjects will receive a trial product that is anticipated to be equally or more efficacious than the treatment they receive at trial entry. Based on the results of the phase 2 dose-finding trial, oral semaglutide is expected to provide clinically relevant improvements in glycaemic control and body weight in subjects with T2D.

Similarly, treatment with sitagliptin is expected to provide clinically significant improvements in glycaemic control<sup>48</sup>.

In addition, it is expected that all subjects, will benefit from participation through close contact with the trial site, with close follow-up of their T2D and a careful medical examination; all of which will most likely result in an intensified management of their T2D.

All subjects in this trial will receive trial products and auxiliary supplies free of charge.

#### 18.1.3 Risk and benefit conclusion

The safety profile for oral semaglutide generated from the clinical and non-clinical development programme has not revealed any safety issues that would prohibit administration of oral semaglutide in accordance with the planned clinical trial.

The phase 2 results indicate that oral semaglutide will provide clinically relevant improvements in glycaemic control and body weight. Sitagliptin is already a marketed drug approved for the use in subjects with T2D.

Safety and efficacy will be monitored regularly and acceptable glycaemic control will be reinforced at all times during the trial.

In conclusion, the potential risk to the subjects in this trial is considered low and acceptable in view of the anticipated benefits associated with oral semaglutide/sitagliptin in subjects with T2D.

Protocol v 3 consol | 105 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

#### 18.2 Informed consent

In seeking and documenting informed consent, the investigator must comply with applicable regulatory requirement(s) and adhere to ICH GCP<sup>44</sup> and the requirements in the Declaration of Helsinki<sup>2</sup>.

Before any trial-related activity, the investigator must give the subject verbal and written information about the trial and the procedures involved in a form that the subject can read and understand.

The subjects must be fully informed of their rights and responsibilities while participating in the trial as well as possible disadvantages of being treated with the trial products.

The investigator must ensure the subject ample time to come to a decision whether or not to participate in the trial.

A voluntary, signed and personally dated informed consent must be obtained from the subject before any trial-related activity.

The responsibility for seeking informed consent must remain with the investigator, but the investigator may delegate the task to a medically qualified person, in accordance with local requirements. The written informed consent must be signed and personally dated by the person who seeks the informed consent before any trial-related activity.

If information becomes available that may be relevant to the subject's willingness to continue participating in the trial, the investigator must inform the subject in a timely manner, and a revised written subject information must be provided and a new informed consent must be obtained.

In order to avoid missing data, the subjects will be informed about the importance of completing the trial also if the subjects discontinue trial product.

#### 18.3 Data handling

If the subject withdraws from the trial or is lost to follow up, then the subject's data will be handled as follows:

- Data already collected and any data collected at the end-of-trial visit including follow up visits will be retained by Novo Nordisk, entered into the database and used for the CTR.
- Safety events will be reported to Novo Nordisk and regulatory authorities according to local/national requirements.

If data is used, it will always be in accordance with local regulations and IRBs/IECs.
Protocol Date: 28 January 2019 Novo Nordisk

### 18.4 Information to subjects during trial

The subject may receive a "welcome to the trial letter" and a "thank you for your participation letter" after completion of the trial. Further the subject may receive letters during the trial.

All written information to subjects must be sent to IRB/IEC for approval/favourable opinion and to regulatory authorities for approval or notification according to local regulations.

#### 18.5 Premature termination of the trial and/or trial site

Novo Nordisk, the IRBs/IECs or a regulatory authority may decide to stop the trial, part of the trial or a trial site at any time, but agreement on procedures to be followed must be obtained.

If the trial is suspended or prematurely terminated, the investigator must inform the subjects promptly and ensure appropriate therapy and follow-up. The investigator and/or Novo Nordisk must also promptly inform the regulatory authorities and IRBs/IECs and provide a detailed written explanation.

If, after the termination of the trial, the benefit-risk analysis changes, the new evaluation must be provided to the IRBs/IECs in case it has an impact on the planned follow-up of subjects who have participated in the trial. If it has an impact, the actions needed to inform and protect the subjects should be described.

Protocol v 3 consol | 107 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

# 19 Protocol compliance

### 19.1 Protocol deviations

Deviations from the protocol should be avoided.

If deviations do occur, the investigator must inform the monitor and the implications of the deviation must be reviewed and discussed.

Deviations must be documented and explained in a protocol deviation by stating the reason, date, and the action(s) taken. Some deviations, for which corrections are not possible, can be acknowledged and confirmed via edit checks in the eCRF or via listings from the trial database.

Documentation on protocol deviations must be kept in the investigator trial master file and sponsor trial master file.

# 19.2 Prevention of missing data

The importance of subject retention will be addressed by Novo Nordisk in the training and communication with the trial sites.

The subjects will be carefully informed about the trial procedures before signing informed consent, so that they know the implications of participating in the trial.

Close surveillance of subject retention will be performed throughout the trial by Novo Nordisk with focus on reasons for premature discontinuation of trial product or withdrawal of consent to secure early mitigations in collaboration with the trial sites.

The investigator will make every effort to ensure that all assessments are performed and data is collected. If missing data does occur the reason will be collected via the protocol deviation process (see Section 19.1). Novo Nordisk will monitor protocol deviations on an on-going basis throughout the trial followed by appropriate actions (e.g. re-training of site staff).

Protocol v 3 consol | 108 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

# 20 Audits and inspections

Any aspect of the clinical trial may be subject to audits conducted by Novo Nordisk or inspections from domestic or foreign regulatory authorities or from IRBs/IECs. Audits and inspections may take place during or after the trial. The investigator and the site staff as well as Novo Nordisk staff have an obligation to cooperate and assist in audits and inspections. This includes giving auditors and inspectors direct access to all source documents and other documents at the trial site relevant to the clinical trial. This includes permission to examine, analyse, verify and reproduce any record(s) and report(s) that are relevant to the evaluation of the trial.

Protocol v 3 consol | 109 of 145

28 January 2019 | Novo Nordisk Protocol Date: Trial ID: NN9924-4309 Version: 3.0 Final

Status:

Page:


UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38

#### 21 Critical documents

Before a trial site is allowed to start screening subjects, written notification from Novo Nordisk must be received and the following documents must be available to Novo Nordisk:

- Regulatory approval and/or acknowledgement of notification as required
- Approval/favourable opinion from IRBs/IECs clearly identifying the documents reviewed as follows: protocol, any protocol amendments, subject information/informed consent form, any other written information to be provided to the subject and subject recruitment materials
- List of IRB/IEC members and/or constitution (or a general assurance number/statement of compliance)
- Curricula vitae of investigator and sub-investigator(s) (current, dated and signed must include documented GCP training or a certificate)
- Signed receipt of Investigator's Brochure for oral semaglutide
- Signed and dated Agreement on Protocol
- Signed and dated Agreement on Protocol Amendment, if applicable
- Contract, signed by the investigator and/or appropriate parties on behalf of the investigator's site and Novo Nordisk
- Source document agreement
- Central laboratory certification and normal ranges
- Insurance statement, if applicable
- Financial disclosure form from investigator and sub-investigator(s)

Novo Nordisk will analyse and report data from all sites together if more than one site is involved in the trial.

By signing the protocol agreement, each investigator agrees to comply fully with ICH GCP<sup>44</sup>, applicable regulatory requirements and the Declaration of Helsinki<sup>2</sup>.

By signing the protocol agreement, each investigator also agrees to allow Novo Nordisk to make investigator's name and information about site name and address publically available if this is required by national or international regulations.

Protocol v 3 consol | 110 of 145 Protocol Date: 28 January 2019 Novo Nordisk

# 22 Responsibilities

The investigator is accountable for the conduct of the trial at his/her site and must ensure adequate supervision of the conduct of the trial at the trial site. If any tasks are delegated, the investigator must maintain a log of appropriately qualified persons to whom he/she has delegated specified trial-related duties. The investigator must ensure that there is adequate and documented training for all staff participating in the conduct of the trial. It is the investigator's responsibility to supervise the conduct of the trial and to protect the rights, safety, and well-being of the subjects.

A qualified physician, who is an investigator or a sub-investigator for the trial, must be responsible for all trial-related medical decisions.

The investigator will follow instructions from Novo Nordisk when processing data.

The investigator is responsible for filing essential documents (i.e. those documents which individually and collectively permit evaluation of the conduct of a trial and the quality of the data produced) in the investigator trial master file. The documents including the subject identification code list must be kept in a secure locked facility, so no unauthorized persons can get access to the data.

The investigator will take all necessary technical and organisational safety measures to prevent accidental or wrongful destruction, loss or deterioration of data. The investigator will prevent any unauthorised access to data or any other processing of data against applicable law. The investigator must be able to provide the necessary information or otherwise demonstrate to Novo Nordisk that such technical and organisational safety measures have been taken.

During any period of unavailability, the investigator must delegate responsibility for medical care of subjects to a specific qualified physician who will be readily available to subjects during that time.

If the investigator is no longer able to fulfil the role as investigator (e.g. if he/she moves or retires), a new investigator will be appointed in consultation with Novo Nordisk.

The investigator and other site personnel must have sufficient English skills according to their assigned task(s).

Protocol v 3 consol | 111 of 145

Protocol Trial ID: NN9924-4309 Date: 28 January 2019 Version: 3.0

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

# 23 Reports and publications

The information obtained during the conduct of this trial is considered confidential, and may be used by or on behalf of Novo Nordisk for regulatory purposes as well as for the general development of the trial product. All information supplied by Novo Nordisk in connection with this trial shall remain the sole property of Novo Nordisk and is to be considered confidential information.

No confidential information shall be disclosed to others without prior written consent from Novo Nordisk. Such information shall not be used except in the performance of this trial. The information obtained during this trial may be made available to other physicians who are conducting other clinical trials with the trial product, if deemed necessary by Novo Nordisk. Provided that certain conditions are fulfilled, Novo Nordisk may grant access to information obtained during this trial to researchers who require access for research projects studying the same disease and/or trial product studied in this trial.

Novo Nordisk may publish on its clinical trials website a redacted CTR for this trial.

One or two investigators will be appointed by Novo Nordisk to review and sign the CTR (signatory investigator) on behalf of all participating investigators. The signatory investigator(s) will be appointed based upon the criteria defined by the ICMJE for research publications<sup>63</sup>.

### 23.1 Communication of results

Novo Nordisk commits to communicating, and otherwise making available for public disclosure, results of trials regardless of outcome. Public disclosure includes publication of a paper in a scientific journal, abstract submission with a poster or oral presentation at a scientific meeting, or disclosure by other means.

The results of this trial will be subject to public disclosure on external web sites according to international and national regulations, as reflected in the Novo Nordisk Code of Conduct for Clinical Trial Disclosure<sup>64</sup>.

Novo Nordisk reserves the right to defer the release of data until specified milestones are reached, for example when the CTR is available. This includes the right not to release the results of interim analyses, because the release of such information may influence the results of the entire trial.

At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

In all cases the trial results will be reported in an objective, accurate, balanced and complete manner, with a discussion of the strengths and limitations. All authors will be given the relevant

Protocol v 3 consol | 112 of 145

| Protocol | Date: | 28 January 2019 | Novo Nordisk |
|---|---|---|---|
| UTN: U1111-1188-1256 | Status: | Final | |
| EudraCT no.: 2018-002589-38 | Page: | 113 of 120 | |

statistical tables, figures, and reports needed to evaluate the planned publication. In the event of any disagreement on the content of any publication, both the investigators' and Novo Nordisk opinions will be fairly and sufficiently represented in the publication.

Where required by the journal, the investigator from each trial site will be named in an acknowledgement or in the supplementary material, as specified by the journal.

Novo Nordisk maintains the right to be informed of plans by any investigator to publish and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to Novo Nordisk before submission for comments. Comments will be given within four weeks from receipt of the planned communication.

# 23.1.1 Authorship

Authorship of publications should be in accordance with the Uniform Requirements of the International Committee of Medical Journal Editors<sup>63</sup> (sometimes referred to as the Vancouver Criteria). Novo Nordisk will appoint investigator(s) to prepare publications in collaboration with Novo Nordisk.

# 23.1.2 Site-specific publication(s) by investigator(s)

For a multicentre clinical trial, analyses based on single-site data usually have significant statistical limitations and frequently do not provide meaningful information for healthcare professionals or subjects, and therefore may not be supported by Novo Nordisk. It is a Novo Nordisk policy that such individual reports do not precede the primary manuscript and should always reference the primary manuscript of the trial.

Novo Nordisk reserves the right to prior review of such publications. Further to allow for the primary manuscript to be published as the first, Novo Nordisk asks for deferment of publication of individual site results until the primary manuscript is accepted for publication. As Novo Nordisk wants to live up to the industry publication policy, submission of a primary publication will take place no later than 18 months after trial completion.

#### 23.2 Investigator access to data and review of results

As owner of the trial database, Novo Nordisk has the discretion to determine who will have access to the database.

Individual investigators will have their own research subjects' data, and will be provided with the randomisation code after results are available.

Protocol v 3 consol | 113 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

# 24 Retention of clinical trial documentation and human biosamples

#### 24.1 Retention of clinical trial documentation

Subject's medical records must be kept for the maximum period permitted by the hospital, institution or private practice.

The investigator must agree to archive the documentation (this includes both electronic and paper-based records) pertaining to the trial in an archive after completion or discontinuation of the trial if not otherwise notified. The investigator should not destroy any documents without prior permission from Novo Nordisk. If the investigator cannot archive the documents at the trial site, Novo Nordisk can refer the investigator to an independent archive provider that has a system in place to allow only the investigator to access the files.

The investigator must be able to access his/her trial documents without involving Novo Nordisk in any way. Site-specific CRFs and other subject data (in an electronic readable format or as paper copies or prints) will be provided to the investigator before access is revoked to the systems and/or electronic devices supplied by Novo Nordisk. These data must be retained by the trial site. If the provided data (e.g. the CD-ROM) is not readable during the entire storage period, the investigator can request a new copy. A copy of all data will be stored by Novo Nordisk.

Novo Nordisk will maintain Novo Nordisk documentation pertaining to the trial for at least 20 years after discontinuation of the marketing authorisation, termination of the trial or cancellation of the research project whichever is longest.

The files from the trial site/institution must be retained for 15 years after end of trial as defined in Section 7, or longer if required by local regulations or Novo Nordisk. In any case trial files cannot be destroyed until the trial site/institution is notified by Novo Nordisk. The deletion process must ensure confidentiality of data and must be done in accordance with local regulatory requirements.

Protocol v 3 consol | 114 of 145

Protocol Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

# 25 Institutional Review Boards/Independent Ethics Committees and regulatory authorities

#### **IRB/IEC:**

Written approval or favourable opinion must be obtained from IRB/IEC prior to commencement of the trial.

During the trial, the investigator or Novo Nordisk, as applicable, must promptly report the following to the IRB/IEC, in accordance with local requirements: updates to IB, unexpected SAEs where a causal relationship cannot be ruled out, protocol amendments according to local requirements, deviations to the protocol implemented to eliminate immediate hazards to the subjects, new information that may affect adversely the safety of the subjects or the conduct of the trial (including new benefit-risk analysis in case it will have an impact on the planned follow-up of the subjects), annually written summaries of the trial status, and other documents as required by the local IRB/IEC.

The investigator must ensure submission of the CTR synopsis to the IRB/IEC.

Protocol amendments must not be implemented before approval or favourable opinion according to local regulations, unless necessary to eliminate immediate hazards to the subjects.

The investigator must maintain an accurate and complete record of all submissions made to the IRB/IEC. The records must be filed in the investigator trial master file and copies must be sent to Novo Nordisk.

#### **Regulatory Authorities:**

Regulatory authorities will receive the clinical trial application, protocol amendments, reports on SAEs, and the CTR according to national requirements.

Protocol v 3 consol 115 of 145

Protocol
Trial ID: NN9924-4309


Date: 28 January 2019 Version: 3.0

# 26 Indemnity statement

Novo Nordisk carries product liability for its products, and liability as assumed under the special laws, acts and/or guidelines for conducting clinical trials in any country, unless others have shown negligence.

Novo Nordisk assumes no liability in the event of negligence, or any other liability of the sites or investigators conducting the trial, or by persons for whom the said site or investigator are responsible.

Protocol v 3 consol | 116 of 145

# 27 References

- 1. International Conference on Harmonisation. ICH Harmonised Tripatite Guideline. Guideline for Good Clinical Practise E6(R2), Step 4. 09 Nov 2016.
- 2. World Medical Association. Declaration of Helsinki. Ethical Principles for Medical Research Involving Human Subjects. Last amended by the 64th WMA General Assembly, Fortaleza, Brazil. October 2013.
- 3. DeFronzo RA. Pathogenesis of type 2 diabetes mellitus. Med Clin North Am. 2004;88(4):787-835, ix.
- 4. Chuang LM, Tsai ST, Huang BY, Tai TY, Diabcare-Asia Study Group. The status of diabetes control in Asia--a cross-sectional survey of 24 317 patients with diabetes mellitus in 1998. Diabet Med. 2002;19(12):978-85.
- 5. Ford ES, Li C, Little RR, Mokdad AH. Trends in A1C concentrations among U.S. adults with diagnosed diabetes from 1999 to 2004. Diabetes Care. 2008;31(1):102-4.
- 6. Holst JJ, Vilsboll T, Deacon CF. The incretin system and its role in type 2 diabetes mellitus. Mol Cell Endocrinol. 2009;297(1-2):127-36.
- 7. Kieffer TJ, Habener JF. The glucagon-like peptides. Endocr Rev. 1999;20(6):876-913.
- 8. Bagger JI, Knop FK, Lund A, Vestergaard H, Holst JJ, Vilsboll T. Impaired regulation of the incretin effect in patients with type 2 diabetes. J Clin Endocrinol Metab. 2011;96(3):737-45.
- 9. Perley MJ, Kipnis DM. Plasma insulin responses to oral and intravenous glucose: studies in normal and diabetic sujbjects. J Clin Invest. 1967;46(12):1954-62.
- 10. Hojberg PV, Vilsboll T, Rabol R, Knop FK, Bache M, Krarup T, et al. Four weeks of near-normalisation of blood glucose improves the insulin response to glucagon-like peptide-1 and glucose-dependent insulinotropic polypeptide in patients with type 2 diabetes. Diabetologia. 2009;52(2):199-207.
- 11. Meier JJ. GLP-1 receptor agonists for individualized treatment of type 2 diabetes mellitus. Nat Rev Endocrinol. 2012;8(12):728-42.
- 12. Flint A, Raben A, Astrup A, Holst JJ. Glucagon-like peptide 1 promotes satiety and suppresses energy intake in humans. J Clin Invest. 1998;101(3):515-20.
- 13. Nauck MA, Niedereichholz U, Ettler R, Holst JJ, Orskov C, Ritzel R, et al. Glucagon-like peptide 1 inhibition of gastric emptying outweighs its insulinotropic effects in healthy humans. Am J Physiol. 1997;273(5 Pt 1):E981-8.
- 14. Nauck MA, Kleine N, Orskov C, Holst JJ, Willms B, Creutzfeldt W. Normalization of fasting hyperglycaemia by exogenous glucagon-like peptide 1 (7-36 amide) in type 2 (non-insulin-dependent) diabetic patients. Diabetologia. 1993;36(8):741-4.
- 15. Toft-Nielsen MB, Damholt MB, Madsbad S, Hilsted LM, Hughes TE, Michelsen BK, et al. Determinants of the impaired secretion of glucagon-like peptide-1 in type 2 diabetic patients. J Clin Endocrinol Metab. 2001;86(8):3717-23.
- 16. Nauck MA, Petrie JR, Sesti G, Mannucci E, Courreges JP, Atkin S, et al. The once-weekly human GLP-1 analogue semaglutide provides significant reductions in HbA1c and body weight in patients with type 2 diabetes. EASD abstract. 2012.
- 17. EMA. ICH guideline M3(R2) on non-clinical safety studies for the conduct of human clinical trials and marketing authorisation for pharmaceuticals (EMA/CPMP/ICH/286/1995). 2009 2009.

Protocol v 3 consol | 117 of 145

EudraCT no.: 2018-002589-38

 Protocol
 Date:
 28 January 2019
 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final


Waser B, Blank A, Karamitopoulou E, Perren A, Reubi JC. Glucagon-like-peptide-1 receptor expression in normal and diseased human thyroid and pancreas. Mod Pathol. 2015;28(3):391-402.

Novo Nordisk A/S. Investigator's Brochure, oral semaglutide, project NN9924 (edition 9 or any updates hereof). 13 Mar 2018.

Ahren B, Landin-Olsson M, Jansson PA, Svensson M, Holmes D, Schweizer A. Inhibition of dipeptidyl peptidase-4 reduces glycemia, sustains insulin levels, and reduces glucagon levels in type 2 diabetes. J Clin Endocrinol Metab. 2004;89(5):2078-84.

Limited MSDAP. JANUVIA - Labelling CFDA. 2011 2011.

Merck Sharp & Dohme Ltd. JANUVIA (sitagliptin), EU summary of product characteristics (SmPC). 24 Oct 2016.

Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, et al. Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012;35(6):1364-79.

Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, et al. Management of hyperglycaemia in type 2 diabetes, 2015: a patient-centred approach. Update to a position statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetologia. 2015;58(3):429-42.

Novo Nordisk Code of Conduct for Clinical Trial Disclosure. Avaliable from: <a href="http://novonordisk-trials.com/website/content/how-we-disclose-trial-information.aspx">http://novonordisk-trials.com/website/content/how-we-disclose-trial-information.aspx</a>. 11 Jan 2015.

- De Angelis C, Drazen JM, Frizelle FA, Haug C, Hoey J, Horton R, et al. Clinical trial registration: a statement from the International Committee of Medical Journal Editors. N Engl J Med. 2004;351(12):1250-1.
- 27. U.S. Department of Health and Human Services, Food and Drug Administration. Food and Drug Administration Amendments Act of 2007. 27 September 2007.
- 28. The European Parliament and the Council of the European Council. Directive 2001/20/EC of the European Parliament and of the Councill of 4 April 2001 on the approximation of the laws, regulations and administrative provisions of the Member States relating to the implementation of good clinical practice in the conduct of clinical trials on medicinal products for human use, article 11. Official Journal of the European Communities. 1 May 2001.
- 29. The European Parliament and the Council of the European Council. Regulation (EC) No 726/2004 of the European Parliament and of the Council of 31 March 2004 laying down Community procedures for the authorisation and supervision of medicinal products for human and veterinary use and establishing a European Medicines Agency, article 57. Official Journal of the European Communities. 2004.
- 30. Ware JE, Jr., Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992;30(6):473-83.
- 31. Ware JE, Kosinski M, Dewey JE. How to Score Version Two of the SF-36 Health Survey. 3<sup>rd</sup> ed: Lincoln RI: QualityMetric, Incorporated. 2000.
- 32. Turner-Bowker DM, Bartley PJ, Ware JE. SF-36® Health Survey and "SF" Bibliography. Lincoln, Rhode Island: QualityMetric Incorporated; 2002.
- 33. Hill AJ. The psychology of food craving. Proc Nutr Soc. 2007;66(2):277-85.

Protocol v 3 consol | 118 of 145

| Protocol | Date: | 28 January 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT no.: 2018-002589-38 | Page: | 119 of 120 | |

- 34. Hill AJ, Heaton-Brown L. The experience of food craving: a prospective investigation in healthy women. J Psychosom Res. 1994;38(8):801-14.
- 35. Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, et al. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016;26(1):1-133.
- 36. National Kidney F. KDOQI Clinical Practice Guideline for Diabetes and CKD: 2012 Update. Am J Kidney Dis. 2012;60(5):850-86.
- 37. Seaquist ER, Anderson J, Childs B, Cryer P, Dagogo-Jack S, Fish L, et al. Hypoglycemia and diabetes: a report of a workgroup of the American Diabetes Association and the Endocrine Society. Diabetes Care. 2013;36(5):1384-95.
- 38. McAulay V, Deary IJ, Frier BM. Symptoms of hypoglycaemia in people with diabetes. Diabet Med. 2001;18(9):690-705.
- 39. U.S. Department of Health and Human Services, Food and Drug Administration. Guidance for Industry. Patient-Reported Outcome Measures: Use in Medical Product Development to Support Labeling Claims. December 2009.
- 40. Stull DE, Leidy NK, Parasuraman B, Chassany O. Optimal recall periods for patient-reported outcomes: challenges and potential solutions. Curr Med Res Opin. 2009;25(4):929-42.
- 41. European Commission. The Rules Governing Medicinal Products in the European Union, Volume 4, Annex 13, Investigational Medicinal Products. Brussels, February 2010.
- 42. European Medicines Agency. Guideline on good pharmacovigilance practices (GVP) Module VIII Post-authorisation safety studies (EMA/813938/2011 Rev 3). 2017.
- 43. Investigators brochure for oral semaglutide (NN9924), edition 7 or any updates hereof. 2016 2016.
- 44. International Conference on Harmonisation. ICH Harmonised Tripartite Guideline. Guideline for Good Clinical Practice E6(R1), Step 4. 10 June 1996.
- 45. Hicks KA, Hung HMJ, Mahaffey KW, Mehran R, Nissen SE, Strockbridge NL, et al. Standardized Definitions for Cardiovascular and Stroke End Point Events in Clinical Trials (Draft). 20 Aug 2014.
- 46. Hicks KA, Mahaffey KW, Mehran R, Nissen SE, Wiviott SD, Dunn B, et al. 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials. Circulation. 2018;137(9):961-72.
- 47. KDIGO. KDIGO Clinical Practice Guideline for Acute Kidney Injury. Kidney international supplements. 2012;2(1):1-138.
- 48. Merck Sharp & Dohme Limited. JANUVIA European Summary of Product Characteristics Annex 1. 26 May 2015.
- 49. Bretz F, Posch M, Glimm E, Klinglmueller F, Maurer W, Rohmeyer K. Graphical approaches for multiple comparison procedures using weighted Bonferroni, Simes, or parametric tests. Biometrical Journal. 2011;53(6):894-913.
- 50. Rohmeyer K, Klinglmueller F. gMCP: Graph Based Multiple Test Procedures. R package version 0.8-8. 3 Oct 2014.
- 51. Little RJA, Rubin DB. Statistical analysis with missing data: New York: John Wiley & Sons. 1987.

Protocol v 3 consol | 119 of 145

28 January 2019 Novo Nordisk Protocol Date: Trial ID: NN9924-4309 Version: 3.0 UTN: U1111-1188-1256 Final Status: EudraCT no.: 2018-002589-38 120 of 120 Page:

- Koch GG. Comments on 'Current issues in non-inferiority trials' by Thomas R. Fleming, 52. Statistics in Medicine, DOI: 10.1002/sim.2855. Stat Med. 2008;27(3):333-42.
- European Medicines Agency, Committee for Medicinal Products for Human Use (CHMP). 53. Guideline on Missing Data in Confirmatory Clinical Trials (EMA/CPMP/EWP/1776/99 Rev. 1). 2 Jul 2010.
- 54. National Academy of Sciences (NAS). The Prevention and Treatment of Missing Data in Clinical Trials. Washington D.C.: The National Academies Press. 2010.
- Schwartz NS, Clutter WE, Shah SD, Cryer PE. Glycemic thresholds for activation of 55. glucose counterregulatory systems are higher than the threshold for symptoms. J Clin Invest. 1987;79(3):777-81.
- 56. Dahl-Jørgensen K, Brinchmann-Hansen O, Hanssen KF, Sandvik L, Aagenaes O. Rapid tightening of blood glucose control leads to transient deterioration of retinopathy in insulin dependent diabetes mellitus: the Oslo study. Br Med J (Clin Res Ed). 1985;290(6471):811-
- The Diabetes Control and Complications Trial Research Group. Early worsening of diabetic 57. retinopathy in the Diabetes Control and Complications Trial. Arch Ophthalmol. 1998;116(7):874-86.
- Varadhan L, Humphreys T, Walker AB, Varughese GI. The impact of improved glycaemic 58. control with GLP-1 receptor agonist therapy on diabetic retinopathy. Diabetes Res Clin Pract. 2014;103(3):e37-9.
- 59. Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998;352(9131):837-53, Erratum 1999; 354: 602.
- 60. The Action to Control Cardiovascular Risk in Diabetes Follow-On (ACCORDION) Eye Study Group and the Action to Control Cardiovascular Risk in Diabetes Follow-On (ACCORDION) Study Group. Persistent Effects of Intensive Glycemic Control on Retinopathy in Type 2 Diabetes in the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Follow-On Study. Diabetes Care. 2016;39(7):1089-100.
- 61. Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jódar E, Leiter LA, et al. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016;375:1834-44.
- 62. American Diabetes Association. Standards of medical care in diabetes. Diabetes Care. 2017;40 (Suppl. 1):S1-S135.
- International Committee of Medical Journal Editors. Recommendations for the Conduct, 63. Reporting, Editing and Publication of Scholarly Work in Medical Journals; current version available at www.icmje.org.
- 64. Novo Nordisk A/S. http://www.novonordisk-trials.com/website/content/how-we-disclosetrial-information.aspx.

Protocol v 3 consol 120 of 145 Protocol - Appendix A Trial ID: NN9924-4309 UTN: U1111-1188-1256

EudraCT no.: 2018-002589-38


Date: Version: Status: Page:

28 January 2019 | Novo Nordisk 3.0 Final 1 of 6

# Appendix A

# **Monitoring of Calcitonin**

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.

Protocol v 3 consol | 121 of 145 Protocol - Appendix A
Trial ID: NN9924-4309

Date: 28 January 2019 Novo Nordisk

# 1 Background

Treatment with glucagon-like peptide-1 receptor agonists has shown to be associated with thyroid C-cell changes in rodents but not in non-human primates. The human relevance of this finding is unknown. However, based on the findings in rodents, monitoring of serum calcitonin (a sensitive biomarker for C-cell activation) is currently being performed in clinical trials with semaglutide.

While there is general agreement on the clinical interpretation of substantially elevated calcitonin levels (greater than 100 ng/L) as likely indicative of C-cell neoplasia, the interpretation of values between upper normal range (5.0 and 8.4 ng/L for women and men, respectively) and 100 ng/L is less clear with regards to indication of disease.

There are several known confounding factors affecting calcitonin levels, e.g.:

- renal dysfunction
- smoking
- autoimmune thyroiditis
- several drug classes (e.g. proton pump inhibitors, beta-blockers, H<sub>2</sub>-blockers and glucocorticoids)

Physiology of C-cell activation in various clinical conditions and in different patient populations (i.e. with various co-morbidities) is poorly understood. There may be various clinical conditions not identified so far which mildly or moderately affect calcitonin secretion by C-cells.

Protocol v 3 consol | 122 of 145

| Protocol - Appendix A | Date: | 28 January 2019 | Novo Nordisk |
|---|---|---|---|
| UTN: U1111-1188-1256 | Status: | Final | |

Page:


# 2 Calcitonin monitoring

EudraCT no.: 2018-002589-38

A blood sample will be drawn at pre-specified trial visits for measurement of calcitonin.

In case a subject has a calcitonin value  $\geq 10$  ng/L the algorithm outlined in <u>Figure 1</u> and described below should be followed. The algorithm applies for all calcitonin values in the trial.



Figure 1 Flow of calcitonin monitoring

# 2.1 Calcitonin $\geq$ 100 ng/L

**Action:** The subject must immediately be referred to a thyroid specialist for further evaluation and the trial product must be discontinued (see protocol Section  $\underline{6.5}$  premature discontinuation of trial

Protocol v 3 consol | 123 of 145

product). The subject should remain in the trial, however, all medications suspected to relate to this condition must be discontinued until diagnosis has been established.

**Background:** These values were found in 9 (0.15%) of a population of 5817 patients with thyroid nodular disease<sup>1</sup>. All of these patients were diagnosed with medullary thyroid carcinoma resulting in a positive predictive value of 100 %.

Diagnostic evaluation should include:

- thyroid ultrasound examination
- fine needle aspiration of any nodules > 1 cm
- potentially surgery with neck dissection

In case a subject is diagnosed with medullary thyroid carcinoma, it is common clinical practice to explore the family history of medullary thyroid carcinoma or multiple endocrine neoplasia and perform a genetic test for RET proto-oncogene mutation.

# 2.2 Calcitonin $\geq$ 50 and < 100 ng/L

**Action:** The subject should be referred to a thyroid specialist for further evaluation. The subject should remain in the trial and continuation on trial product should be based on the evaluation done by the thyroid specialist.

**Background:** These values were found in 8 (0.14%) of the population of 5817 patients with thyroid nodular disease<sup>1</sup>. Two of these subjects were diagnosed with medullary thyroid carcinoma and two were diagnosed with C-cell hyperplasia, resulting in a positive predictive value of a C-cell anomaly of 50%.

Diagnostic evaluation should include:

- thyroid ultrasound examination
- if available and there are no contraindication, a pentagastrin stimulation test should be done. For subjects with positive pentagastrin stimulation test, surgery should be considered.
- if pentagastrin stimulation test is not available, thyroid ultrasound and fine needle aspiration biopsy may add important clinical information about the need for surgery.

# 2.3 Calcitonin $\geq$ 10 and $\leq$ 50 ng/L

**Action:** The subject can continue in the trial on trial product. Continue sampling of calcitonin according to the protocol.

If the value is from the last sample taken in the trial, the subject should be referred to a thyroid specialist for further evaluation.

Protocol v 3 consol | 124 of 145

**Background:** Calcitonin values from 20-50 ng/L were found in up to 1% of subjects of the population of 5817 patients with thyroid nodular disease<sup>1</sup>. The predictive value of a C-cell anomaly for this calcitonin level was 8.3%. However, the likelihood of having a medullary carcinoma >1 cm with calcitonin in this range is extremely low.

For calcitonin values between 10-20 ng/L Costante et al $^1$  identified 216 (3.7%) patients. One patient out of the 216 had a subsequent basal (unstimulated) calcitonin of 33 ng/L, and had C-cell hyperplasia at surgery. Two other studies used a cut-off of calcitonin > 10 ng/L to screen for C-cell disease, but they do not provide sufficient information on patients with basal calcitonin > 10 and < 20 ng/L to allow conclusions $^{2.3}$ .

Protocol v 3 consol | 125 of 145

# 3 References

- 1 Costante G, Meringolo D, Durante C, Bianchi D, Nocera M, Tumino S et al. Predictive value of serum calcitonin levels for preoperative diagnosis of medullary thyroid carcinoma in a cohort of 5817 consecutive patients with thyroid nodules. J Clin Endocrinol Metab 2007; 92(2):450-455.
- 2 Scheuba C, Kaserer K, moritz A, drosten R. Sporadic hypercalcitoninemia: clinica and therapeutic consequences. Endocrine Related Cancer 2009; 16(1):243-253.
- 3 Verga U, Ferrero S, Vicentini L, Brambilla T, Cirello V, Muzza M et al. Histopathological and molecular studies in patients with goiter and hypercalcitoninemia: reactive or neoplastic C-cell hyperplasia? Endocr Relat Cancer 2007; 14(2):393-403.

Protocol v 3 consol | 126 of 145

Protocol - Appendix B Trial ID: NN9924-4309 UTN: U1111-1188-1256

EudraCT no.: 2018-002589-38


Date: Version: Status: Page:

28 January 2019 | Novo Nordisk 3.0 Final 1 of 8

# Appendix B

# Adverse events requiring additional data collection

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.

Protocol v 3 consol | 127 of 145 Protocol - Appendix B
Trial ID: NN9924-4309

Date: 28 January 2019 | Novo Nordisk

UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38 Status: Final Page: 2 of 8

# 1 Adverse events requiring additional data collection

For the following adverse events (AEs) additional data collection is required and specific event forms must be completed in the electronic case report form (eCRF) in addition to the AE form:

- Acute coronary syndrome (myocardial infarction or unstable angina pectoris requiring hospitalisation)
- Acute gallstone disease
- Cerebrovascular event (stroke or transient ischaemic attack)
- Heart failure
- Hypersensitivity reaction
- Neoplasm (excluding thyroid neoplasm)
- Thyroid disease (including thyroid neoplasm)
- Pancreatitis
- Renal event
- Medication error (concerning trial products):
  - Administration of wrong drug. Note: Use of wrong dispensing unit number (DUN) is not considered a medication error.
  - Wrong route of administration.
  - Accidental administration of a higher dose than intended. A higher dose is a dose of at least one tablet more than the intended dose; however the administered dose must deviate from the intended dose to an extent where clinical consequences for the trial subject were likely to happen as judged by the investigator, although they did not necessarily occur.
- Abuse and misuse of trial product

Abuse is defined as:

Persistent or sporadic, intentional excessive use of a medicinal product, which is accompanied by harmful physical or psychological effects (e.g. overdose with the intention to cause harm). Misuse is defined as:

Situations where the medicinal product is intentionally and inappropriately used not in accordance with the protocol.

- Lactic acidosis
- Creatine kinase (CK) > 10 x upper limit of the normal (ULN)
- Hepatic event defined as:
  - alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 x ULN and total bilirubin  $\leq$  2 x ULN
  - ALT or AST >3 x ULN and total bilirubin > 2 x ULN\*
  - Hepatic event leading to trial product discontinuation
- Diabetic retinopathy and related complications
- \*Please note that in case of a hepatic event defined as ALT or AST > 3 x ULN and total bilirubin > 2 x ULN, where no alternative aetiology exists (Hy's law), this must be reported as an serious

adverse event (SAE) using the important medical event criterion if no other seriousness criteria are applicable.

In case any of these events fulfil the criteria for a SAE, please report accordingly, see protocol Section 12.1.2.

Some of these events will undergo event adjudication by the event adjudication committee (EAC), see protocol Section 12.7.2 and protocol Table 12-1 and Table 12-2.

### 1.1 Acute coronary syndrome

If an event of acute coronary syndrome (ranging from unstable angina pectoris requiring hospitalisation to myocardial infarction) is observed during the trial, the following additional information must be reported if available:

- Duration of symptoms
- Changes in electrocardiogram (ECG)
- Collection of cardiac biomarkers
- Cardiac imaging
- Cardiac stress testing
- Angiography
- Use of thrombolytic drugs
- Revascularisation procedures

### 1.2 Acute gallstone disease

If an event of acute gallstone disease or clinical suspicion of this is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms of acute gallstone disease
- Specific laboratory tests supporting a diagnosis of gallstone
- Imaging performed and consistency with gallstone disease
- Treatment given for the condition
- Relevant risk factors for acute gallstone disease
- Family history of gallstones

#### 1.3 Cerebrovascular event

If a cerebrovascular event (e.g. transient ischaemic attack, stroke) is observed during the trial, the following additional information must be reported if available:

- Type of event (e.g. transient ischaemic attack, stroke)
- Contributing condition
- Neurologic signs and symptoms
- History of neurologic disease

Protocol v 3 consol | 129 of 145

- Imaging supporting the condition
- Treatment given for the condition

#### 1.4 Heart failure

If an event of heart failure is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms of heart failure
- New York Heart Association (NYHA) Class
- Supportive imaging
- Supportive laboratory measurements
- Initiation or intensification of treatment for this condition

# 1.5 Hypersensitivity reaction

All events of hypersensitivity reactions must be reported and the following additional information must be reported if available:

- Signs and symptoms associated to the event
- Time of appearance after administration of trial drug
- Relevant immunological tests performed
- Treatment given for the reaction
- Previous history of similar reaction
- Risk or confounding factors identified

#### 1.5.1 Assessments in case of suspicion of hypersensitivity reaction

If suspicion of a hypersensitivity reaction occurs, the subjects should be instructed to contact the site staff as soon as possible.

In case of suspicion of a severe immediate systemic hypersensitivity reaction<sup>3</sup> to the trial product, the subject must be discontinued from trial product but should remain in the trial (see protocol Section 6.5 and 8.1.5).

In the event of a severe systemic hypersensitivity reaction to trial product it is recommended to test tryptase locally (total and/or mature tryptase) within 3 hours of reaction. Moreover, a baseline tryptase measurement is necessary 1-2 weeks after the immediate severe hypersensitivity reaction due to individual variation in tryptase baseline concentration. Tryptase concentrations, if available, should be included in the specific event form when reporting the AE.

Tryptase measurements are not required at the follow up visits.

Protocol v 3 consol | 130 of 145

In case of suspicion of immune complex disease<sup>3</sup>, the subject must be discontinued from trial product but should remain in the trial (see protocol Section 6.5 and 8.1.5). It is recommended to draw a blood sample for local assessment of complement levels (C3 and C4) to assist in the diagnostic evaluation. Complement level results should be included in the specific event form when reporting the AE.

### 1.6 Neoplasm

All events of neoplasms (excluding thyroid neoplasm, which will be reported under thyroid disease) must be reported during the trial and the following additional information must be reported if available:

- Type of neoplasm
- Symptoms leading to identification of event
- Diagnostic imaging
- Pathological examination results
- Treatment for the event
- Participation in screening programs
- Risk factors associated to the event

### 1.7 Thyroid disease

If an event of thyroid disease, including any thyroid neoplasms, is observed during the trial, the following additional information must be reported if available:

- History of thyroid disease
- Signs and symptoms leading to investigations of thyroid disease
- Specific laboratory tests describing thyroid function
- Diagnostic imaging performed and any prior imaging supporting the disease history
- Pathologic examinations
- Treatment given for the condition
- Risk factors identified
- Family history of thyroid disease

# 1.8 Pancreatitis

For all confirmed events of pancreatitis the following additional information must be reported if available:

- Signs and symptoms of pancreatitis
- Specific laboratory test supporting a diagnosis of pancreatitis
- Imaging performed and consistency with pancreatic disease
- Treatment for and complications of the event
- Relevant risk factors for pancreatic disease

Protocol v 3 consol | 131 of 145

Family history of pancreatic disease

#### 1.8.1 Assessments in case of suspicion of acute pancreatitis

Most patients with acute pancreatitis experience severe abdominal pain that is located generally in the epigastrium and radiates to the back. The onset of the pain may be swift reaching maximum intensity within 30 min, it is frequently unbearable and characteristically persists for more than 24 hours without relief. The pain is often associated with nausea and vomiting. Physical examination usually reveals severe upper abdominal tenderness at times associated with guarding.

In general, both amylase and lipase are elevated during the course of acute pancreatitis. The serum lipase may remain elevated slightly longer than amylase. The level of the serum amylase and/or lipase does not correlate with the severity of acute pancreatitis. In general, serum lipase is thought to be more sensitive and specific than serum amylase in the diagnosis of acute pancreatitis.

In case of suspicion of acute pancreatitis, trial product treatment should be promptly interrupted. Appropriate additional examinations must be performed, including measurement of amylase and lipase.

The diagnosis of acute pancreatitis requires two of the following three features $\frac{2}{3}$ :

- abdominal pain **consistent** with acute pancreatitis (acute onset of a persistent, severe, epigastric pain often radiating to the back)
- serum lipase activity (and/or amylase activity) at least three times greater than the upper limit of the normal
- **characteristic** findings of acute pancreatitis on imaging.

If acute pancreatitis is ruled out, trial product should be re-initiated.

If acute pancreatitis is confirmed, appropriate treatment and careful monitoring of the subject should be initiated. The subject must be discontinued from trial product (treatment discontinuation call), but should remain in the trial (see protocol Section 6.5 and 8.1.5).

#### 1.9 Renal event

If a renal event is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms of renal failure
- Specific laboratory tests supporting the diagnosis
- Imaging performed supporting the diagnosis
- Kidney biopsy results
- Risk or confounding factors identified including exposure to nephrotoxic agents

Protocol v 3 consol | 132 of 145

#### 1.10 Medication error

If a medication error is observed during the trial, the following information is required and a specific event form must be completed in the eCRF in addition to the AE form (see Section 8.4.1.1 and 12.1.5):

- Trial product(s) involved
- Classification of medication error
  - Wrong drug(s) administered
  - o Administration of an overdose
- Whether the subject experienced any hypoglycaemic episode and/or AE(s) as a result of the medication error
- Suspected primary reason for the medication error

For definition of medication error, see protocol Section 12.1.4.

#### 1.11 Lactic acidosis

If an event of lactic acidosis is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms of lactic acidosis
- Specific laboratory tests describing the event
- Possible cause(s) of the event

#### 1.12 Creatine kinase > 10 x ULN

If an event of  $CK > 10 \times ULN$  is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms associated to the event
- Recent physical activity
- Possible cause(s) of the event

### 1.12.1 Assessments in case of increased levels of creatine kinase

In case of CK > 10 x ULN, prompt repeat testing (at central laboratory) of CK should be done. Repeat testing (at central laboratory) should be done regularly until CK levels return to normal or baseline state. Additional clinical information should be gathered to seek the possible cause of the observed CK elevation.

#### 1.13 Hepatic event

- ALT or AST > 5 x ULN and total bilirubin  $\leq$  2 x ULN
- ALT or AST >3 x ULN and total bilirubin > 2 x ULN\*

Protocol v 3 consol | 133 of 145

Hepatic event leading to trial product discontinuation

\*Please note that risk of liver injury defined as ALT or AST > 3 x ULN and total bilirubin > 2 x ULN, where no alternative aetiology exits (Hy's law), should also be reported as a SAE (important medical event, according to protocol Section 12.1.2).

If one of the above events is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms associated to the event
- Risk factors
- Relevant laboratory test results
- Diagnostic imaging performed
- Possible cause(s) of the event

#### 1.13.1 Assessments in case of increased levels of aminotransferases

Both events should prompt repeat testing (at central laboratory) including ALT, AST, alkaline phosphatase (ALP) and total bilirubin and discontinuation of trial product should be considered. Thereafter, repeat testing (at central laboratory) of ALT, AST, ALP and total bilirubin should be done regularly until the abnormalities return to normal or baseline state. Additional clinical information such as related symptoms, risk factors and contributing conditions (e.g. viral hepatitis, autoimmune hepatitis, alcoholic hepatitis, hepatobiliary or pancreatic disorders) should be gathered to seek a possible cause of the observed laboratory test abnormalities.

### 1.14 Diabetic retinopathy and related complications

If an event of diabetic retinopathy or related complications is observed during the trial the following additional information must be reported, if available:

- Signs and symptoms associated with the event
- Results of the eye examination
- Treatment for and complications of the event
- Contributing conditions

# 2 References

- 1. Banks PA, Freeman ML, Practice Parameters Committee of the American College of G. Practice guidelines in acute pancreatitis. Am J Gastroenterol. 2006;101(10):2379-400.
- 2. Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, et al. Classification of acute pancreatitis-2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013;62(1):102-11.
- 3. U.S. Department of Health and Human Services, Food and Drug Administration. Guidance for Industry: Immunogenicity Assessment for Therapeutic Protein Products. August 2015.

Protocol v 3 consol | 134 of 145

Protocol - Appendix C Trial ID: NN9924-4309

UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38 CONFIDENTIAL

28 January 2019 | Novo Nordisk Date: Version: 3.0 Status: Final

Page:


# **Appendix C**

# Contraceptive guidance and collection of pregnancy information

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.

Protocol v 3 consol | 135 of 145 1 0 | NN9924 - 4309

Protocol - Appendix C Trial ID: NN9924-4309 UTN: U1111-1188-1256

EudraCT no.: 2018-002589-38

28 January 2019 | Novo Nordisk Date: Version: 3.0 Final Status: 

# Contraceptive guidance and collection of pregnancy information

It must be recorded in the eCRF whether female subjects are of childbearing potential

#### **Definitions**

### Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile.

# Women in the following categories are not considered WOCBP

- 1. Premenarcheal
- 2. Premenopausal female with one of the following:
- Documented hysterectomy
- Documented bilateral salpingectomy
- Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's review of subject's medical records, medical examination or medical history interview.

3. Postmenopausal female

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high Follicle Stimulating Hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or Hormonal Replacement Therapy (HRT). However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

Females on HRT and whose menopausal status is in doubt will be required to use one of the non-hormonal highly effective contraception methods if they wish to continue their HRT during the trial. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before trial enrolment.

### Contraception guidance

### Male subjects

No contraception measures are required for male subjects as the risk of teratogenicity/fetotoxicity caused by transfer of semaglutide in seminal fluid is unlikely.

### Female subjects

Female subjects of childbearing potential are eligible to participate if they agree to use methods of contraception consistently and correctly as described in table below:

Protocol v 3 consol 136 of 145 Protocol - Appendix C
Trial ID: NN9924-4309

CONICIDENTIAL

Date: 28 January 2019 Novo Nordisk


### Table 1 Highly effective contraceptive methods

# Highly effective contraceptive methods that are user dependent a and b

Failure rate of <1% per year when used consistently and correctly.

Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation

- oral
- intravaginal
- transdermal

Progestogen only hormonal contraception associated with inhibition of ovulation

- oral
- injectable

# Highly effective methods that are user independent b

#### Sexual abstinence

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial product. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the trial and the preferred and usual lifestyle of the subject.

Implantable progestogen only hormonal contraception associated with inhibition of ovulation

- Intrauterine Device (IUD)
- Intrauterine hormone-releasing System (IUS)
- Bilateral tubal occlusion

#### Vasectomised partner

A vasectomised partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

#### Notes:

<sup>a</sup> Failure rates may differ from < 1% per year, if not used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for subjects participating in clinical trials.

b Contraception should be utilised during the treatment period and for at least 35 days after the last dose of trial product.

#### **Pregnancy testing**

- WOCBP should only be included in the trial after a negative urine pregnancy test at visit 1 and at visit 2.
- Urine pregnancy tests should be performed throughout the trial in accordance with the protocol flowchart, section 2. WOCBP needs the last urine pregnancy test at the end of trial visit (visit 9).
- Pregnancy testing should be performed whenever a menstrual period is missed or when pregnancy is otherwise suspected.
- Additional urine pregnancy testing should be performed during the treatment period, if required locally.

Protocol v 3 consol | 137 of 145

Protocol - Appendix C
Trial ID: NN9924-4309

Date: 28 January 2019 Novo Nordisk

UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38 Date: 28 January 2019 Version: 3.0 Status: Final 

# **Collection of pregnancy information**

### Female subjects who become pregnant

- Investigator will collect pregnancy information on any female subject, who becomes pregnant while participating in this trial.
- Information will be recorded on the appropriate form and submitted to Novo Nordisk within 14 calendar days of learning of a subject's pregnancy.
- Subject will be followed to determine the outcome of the pregnancy. The investigator will collect follow-up information on subject and neonate, which will be forwarded to Novo Nordisk. Generally, follow-up will not be required for longer than 1 month beyond the delivery date.
- Any termination of pregnancy will be reported, regardless of foetal status (presence or absence of anomalies) or indication for procedure.
- While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy will be reported as an AE or SAE.
- A spontaneous abortion is always considered to be an SAE and will be reported as such.
- Any SAE occurring as a result of a post-trial pregnancy which is considered possibly/probably related to the trial products by the investigator will be reported to Novo Nordisk as described in section 12 of the protocol. While the investigator is not obligated to actively seek this information in former subjects, he or she may learn of an SAE through spontaneous reporting.

Any female subject who becomes pregnant while participating in the trial must discontinue trial product.

Protocol v 3 consol | 138 of 145

Protocol - Appendix A
Trial ID: NN9924-4309


Date: 28 January 2019 | Novo Nordisk

UTN: U1111-1188-1256 CONFIDENTIAL Status: Final EudraCT no.: 2018-002589-38 Page: 1 of 6

# Appendix A

# **Monitoring of Calcitonin**

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.

Protocol v 3 0 appx a | 1 of 6

Protocol - Appendix A
Trial ID: NN9924-4309


Date: 28 January 2019 | Novo Nordisk

UTN: U1111-1188-1256 CONFIDENTIAL Status: Final Page: 2 of 6

# 1 Background

Treatment with glucagon-like peptide-1 receptor agonists has shown to be associated with thyroid C-cell changes in rodents but not in non-human primates. The human relevance of this finding is unknown. However, based on the findings in rodents, monitoring of serum calcitonin (a sensitive biomarker for C-cell activation) is currently being performed in clinical trials with semaglutide.

While there is general agreement on the clinical interpretation of substantially elevated calcitonin levels (greater than 100 ng/L) as likely indicative of C-cell neoplasia, the interpretation of values between upper normal range (5.0 and 8.4 ng/L for women and men, respectively) and 100 ng/L is less clear with regards to indication of disease.

There are several known confounding factors affecting calcitonin levels, e.g.:

- renal dysfunction
- smoking
- autoimmune thyroiditis
- several drug classes (e.g. proton pump inhibitors, beta-blockers, H<sub>2</sub>-blockers and glucocorticoids)

Physiology of C-cell activation in various clinical conditions and in different patient populations (i.e. with various co-morbidities) is poorly understood. There may be various clinical conditions not identified so far which mildly or moderately affect calcitonin secretion by C-cells.

Protocol v 3 0 appx a 2 of 6

| Protocol - Appendix A | CONFIDENTIAL | Date: | 28 January 2019 | Novo Nordisk |
|---|---|---|---|---|
| UTN: U1111-1188-1256 | | Status: | Final | |
| EudraCT no.: 2018-002589-38 | | Page: | 3 of 6 | |

# 2 Calcitonin monitoring

A blood sample will be drawn at pre-specified trial visits for measurement of calcitonin.

In case a subject has a calcitonin value  $\geq 10$  ng/L the algorithm outlined in Figure 1 and described below should be followed. The algorithm applies for all calcitonin values in the trial.



Figure 1 Flow of calcitonin monitoring

### 2.1 Calcitonin $\geq$ 100 ng/L

**Action:** The subject must immediately be referred to a thyroid specialist for further evaluation and the trial product must be discontinued (see protocol Section  $\underline{6.5}$  premature discontinuation of trial

Protocol v 3 0 appx a 3 of 6

| Protocol - Appendix A | CONFIDENTIAL | Date: | 28 January 2019 | Novo Nordisk |
|---|---|---|---|---|
| UTN: U1111-1188-1256 | | Status: | Final | |
| EudraCT no.: 2018-002589-38 | | Page: | 4 of 6 | |

product). The subject should remain in the trial, however, all medications suspected to relate to this condition must be discontinued until diagnosis has been established.

**Background:** These values were found in 9 (0.15%) of a population of 5817 patients with thyroid nodular disease<sup> $\frac{1}{2}$ </sup>. All of these patients were diagnosed with medullary thyroid carcinoma resulting in a positive predictive value of 100 %.

Diagnostic evaluation should include:

- thyroid ultrasound examination
- fine needle aspiration of any nodules > 1 cm
- potentially surgery with neck dissection

In case a subject is diagnosed with medullary thyroid carcinoma, it is common clinical practice to explore the family history of medullary thyroid carcinoma or multiple endocrine neoplasia and perform a genetic test for RET proto-oncogene mutation.

### 2.2 Calcitonin $\geq$ 50 and < 100 ng/L

**Action:** The subject should be referred to a thyroid specialist for further evaluation. The subject should remain in the trial and continuation on trial product should be based on the evaluation done by the thyroid specialist.

**Background:** These values were found in 8 (0.14%) of the population of 5817 patients with thyroid nodular disease<sup>1</sup>. Two of these subjects were diagnosed with medullary thyroid carcinoma and two were diagnosed with C-cell hyperplasia, resulting in a positive predictive value of a C-cell anomaly of 50%.

Diagnostic evaluation should include:

- thyroid ultrasound examination
- if available and there are no contraindication, a pentagastrin stimulation test should be done. For subjects with positive pentagastrin stimulation test, surgery should be considered.
- if pentagastrin stimulation test is not available, thyroid ultrasound and fine needle aspiration biopsy may add important clinical information about the need for surgery.

# 2.3 Calcitonin $\geq$ 10 and $\leq$ 50 ng/L

**Action:** The subject can continue in the trial on trial product. Continue sampling of calcitonin according to the protocol.

If the value is from the last sample taken in the trial, the subject should be referred to a thyroid specialist for further evaluation.
**Background:** Calcitonin values from 20-50 ng/L were found in up to 1% of subjects of the population of 5817 patients with thyroid nodular disease <sup>1</sup>. The predictive value of a C-cell anomaly for this calcitonin level was 8.3%. However, the likelihood of having a medullary carcinoma >1 cm with calcitonin in this range is extremely low.

For calcitonin values between 10-20 ng/L Costante et al $^1$  identified 216 (3.7%) patients. One patient out of the 216 had a subsequent basal (unstimulated) calcitonin of 33 ng/L, and had C-cell hyperplasia at surgery. Two other studies used a cut-off of calcitonin > 10 ng/L to screen for C-cell disease, but they do not provide sufficient information on patients with basal calcitonin > 10 and < 20 ng/L to allow conclusions $^{2.3}$ .

Protocol v 3 0 appx a 5 of 6

## 3 References

- 1 Costante G, Meringolo D, Durante C, Bianchi D, Nocera M, Tumino S et al. Predictive value of serum calcitonin levels for preoperative diagnosis of medullary thyroid carcinoma in a cohort of 5817 consecutive patients with thyroid nodules. J Clin Endocrinol Metab 2007; 92(2):450-455.
- 2 Scheuba C, Kaserer K, moritz A, drosten R. Sporadic hypercalcitoninemia: clinica and therapeutic consequences. Endocrine Related Cancer 2009; 16(1):243-253.
- 3 Verga U, Ferrero S, Vicentini L, Brambilla T, Cirello V, Muzza M et al. Histopathological and molecular studies in patients with goiter and hypercalcitoninemia: reactive or neoplastic C-cell hyperplasia? Endocr Relat Cancer 2007; 14(2):393-403.

Protocol v 3 0 appx a

Protocol - Appendix B
Trial ID: NN9924-4309

Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

## Appendix B

# Adverse events requiring additional data collection

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.

Protocol v 3 0 appx b | 1 of 8

Protocol - Appendix B Trial ID: NN9924-4309 UTN: U1111-1188-1256

EudraCT no.: 2018-002589-38

ONFIDENTIAL

Date: 28 January 2019 | Novo Nordisk
Status: Final
Page: 2 of 8

## 1 Adverse events requiring additional data collection

For the following adverse events (AEs) additional data collection is required and specific event forms must be completed in the electronic case report form (eCRF) in addition to the AE form:

- Acute coronary syndrome (myocardial infarction or unstable angina pectoris requiring hospitalisation)
- Acute gallstone disease
- Cerebrovascular event (stroke or transient ischaemic attack)
- Heart failure
- Hypersensitivity reaction
- Neoplasm (excluding thyroid neoplasm)
- Thyroid disease (including thyroid neoplasm)
- Pancreatitis
- Renal event
- Medication error (concerning trial products):
  - Administration of wrong drug.

    Note: Use of wrong dispensing unit number (DUN) is not considered a medication error.
  - Wrong route of administration.
  - Accidental administration of a higher dose than intended. A higher dose is a dose of at least one tablet more than the intended dose; however the administered dose must deviate from the intended dose to an extent where clinical consequences for the trial subject were likely to happen as judged by the investigator, although they did not necessarily occur.
- Abuse and misuse of trial product

Abuse is defined as:

Persistent or sporadic, intentional excessive use of a medicinal product, which is accompanied by harmful physical or psychological effects (e.g. overdose with the intention to cause harm). Misuse is defined as:

Situations where the medicinal product is intentionally and inappropriately used not in accordance with the protocol.

- Lactic acidosis
- Creatine kinase (CK) > 10 x upper limit of the normal (ULN)
- Hepatic event defined as:
  - alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 x ULN and total bilirubin  $\leq$  2 x ULN
  - ALT or AST >3 x ULN and total bilirubin > 2 x ULN\*
  - Hepatic event leading to trial product discontinuation
- Diabetic retinopathy and related complications
- \*Please note that in case of a hepatic event defined as ALT or AST > 3 x ULN and total bilirubin > 2 x ULN, where no alternative aetiology exists (Hy's law), this must be reported as an serious

| Protocol - Appendix B<br>Trial ID: NN9924-4309 | CONFIDENTIAL | Date:<br>Version: | 28 January 2019<br>3.0 | Novo Nordisk |
|---|---|---|---|---|
| UTN: U1111-1188-1256<br>EudraCT no.: 2018-002589-38 | | Status:<br>Page: | Final<br>3 of 8 | |

adverse event (SAE) using the important medical event criterion if no other seriousness criteria are applicable.

In case any of these events fulfil the criteria for a SAE, please report accordingly, see protocol Section 12.1.2.

Some of these events will undergo event adjudication by the event adjudication committee (EAC), see protocol Section 12.7.2 and protocol Table 12-1 and Table 12-2.

### 1.1 Acute coronary syndrome

If an event of acute coronary syndrome (ranging from unstable angina pectoris requiring hospitalisation to myocardial infarction) is observed during the trial, the following additional information must be reported if available:

- Duration of symptoms
- Changes in electrocardiogram (ECG)
- Collection of cardiac biomarkers
- Cardiac imaging
- Cardiac stress testing
- Angiography
- Use of thrombolytic drugs
- Revascularisation procedures

### 1.2 Acute gallstone disease

If an event of acute gallstone disease or clinical suspicion of this is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms of acute gallstone disease
- Specific laboratory tests supporting a diagnosis of gallstone
- Imaging performed and consistency with gallstone disease
- Treatment given for the condition
- · Relevant risk factors for acute gallstone disease
- Family history of gallstones

### 1.3 Cerebrovascular event

If a cerebrovascular event (e.g. transient ischaemic attack, stroke) is observed during the trial, the following additional information must be reported if available:

- Type of event (e.g. transient ischaemic attack, stroke)
- Contributing condition
- Neurologic signs and symptoms
- History of neurologic disease

- Imaging supporting the condition
- Treatment given for the condition

### 1.4 Heart failure

If an event of heart failure is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms of heart failure
- New York Heart Association (NYHA) Class
- Supportive imaging
- Supportive laboratory measurements
- Initiation or intensification of treatment for this condition

## 1.5 Hypersensitivity reaction

All events of hypersensitivity reactions must be reported and the following additional information must be reported if available:

- Signs and symptoms associated to the event
- Time of appearance after administration of trial drug
- Relevant immunological tests performed
- Treatment given for the reaction
- Previous history of similar reaction
- Risk or confounding factors identified

### 1.5.1 Assessments in case of suspicion of hypersensitivity reaction

If suspicion of a hypersensitivity reaction occurs, the subjects should be instructed to contact the site staff as soon as possible.

In case of suspicion of a severe immediate systemic hypersensitivity reaction<sup>3</sup> to the trial product, the subject must be discontinued from trial product but should remain in the trial (see protocol Section 6.5 and 8.1.5).

In the event of a severe systemic hypersensitivity reaction to trial product it is recommended to test tryptase locally (total and/or mature tryptase) within 3 hours of reaction. Moreover, a baseline tryptase measurement is necessary 1-2 weeks after the immediate severe hypersensitivity reaction due to individual variation in tryptase baseline concentration. Tryptase concentrations, if available, should be included in the specific event form when reporting the AE.

Tryptase measurements are not required at the follow up visits.

Protocol v 3 0 appx b  $\hspace{1.5cm} |\hspace{.05cm} 4 \hspace{.05cm} of \hspace{.05cm} 8$ 

In case of suspicion of immune complex disease<sup>3</sup>, the subject must be discontinued from trial product but should remain in the trial (see protocol Section 6.5 and 8.1.5). It is recommended to draw a blood sample for local assessment of complement levels (C3 and C4) to assist in the diagnostic evaluation. Complement level results should be included in the specific event form when reporting the AE.

### 1.6 Neoplasm

All events of neoplasms (excluding thyroid neoplasm, which will be reported under thyroid disease) must be reported during the trial and the following additional information must be reported if available:

- Type of neoplasm
- Symptoms leading to identification of event
- Diagnostic imaging
- Pathological examination results
- Treatment for the event
- Participation in screening programs
- Risk factors associated to the event

### 1.7 Thyroid disease

If an event of thyroid disease, including any thyroid neoplasms, is observed during the trial, the following additional information must be reported if available:

- History of thyroid disease
- Signs and symptoms leading to investigations of thyroid disease
- Specific laboratory tests describing thyroid function
- Diagnostic imaging performed and any prior imaging supporting the disease history
- Pathologic examinations
- Treatment given for the condition
- Risk factors identified
- Family history of thyroid disease

## 1.8 Pancreatitis

For all confirmed events of pancreatitis the following additional information must be reported if available:

- Signs and symptoms of pancreatitis
- Specific laboratory test supporting a diagnosis of pancreatitis
- Imaging performed and consistency with pancreatic disease
- Treatment for and complications of the event
- Relevant risk factors for pancreatic disease

Family history of pancreatic disease

### 1.8.1 Assessments in case of suspicion of acute pancreatitis

Most patients with acute pancreatitis experience severe abdominal pain that is located generally in the epigastrium and radiates to the back. The onset of the pain may be swift reaching maximum intensity within 30 min, it is frequently unbearable and characteristically persists for more than 24 hours without relief. The pain is often associated with nausea and vomiting. Physical examination usually reveals severe upper abdominal tenderness at times associated with guarding.

In general, both amylase and lipase are elevated during the course of acute pancreatitis. The serum lipase may remain elevated slightly longer than amylase. The level of the serum amylase and/or lipase does not correlate with the severity of acute pancreatitis. In general, serum lipase is thought to be more sensitive and specific than serum amylase in the diagnosis of acute pancreatitis.

In case of suspicion of acute pancreatitis, trial product treatment should be promptly interrupted. Appropriate additional examinations must be performed, including measurement of amylase and lipase.

The diagnosis of acute pancreatitis requires two of the following three features $\frac{2}{3}$ :

- abdominal pain consistent with acute pancreatitis (acute onset of a persistent, severe, epigastric
  pain often radiating to the back)
- serum lipase activity (and/or amylase activity) at least three times greater than the upper limit of the normal
- **characteristic** findings of acute pancreatitis on imaging.

If acute pancreatitis is ruled out, trial product should be re-initiated.

If acute pancreatitis is confirmed, appropriate treatment and careful monitoring of the subject should be initiated. The subject must be discontinued from trial product (treatment discontinuation call), but should remain in the trial (see protocol Section 6.5 and 8.1.5).

## 1.9 Renal event

If a renal event is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms of renal failure
- Specific laboratory tests supporting the diagnosis
- Imaging performed supporting the diagnosis
- Kidney biopsy results
- Risk or confounding factors identified including exposure to nephrotoxic agents

Protocol v 3 0 appx b

#### 1.10 Medication error

If a medication error is observed during the trial, the following information is required and a specific event form must be completed in the eCRF in addition to the AE form (see Section 8.4.1.1 and 12.1.5):

- Trial product(s) involved
- Classification of medication error
  - Wrong drug(s) administered
  - Administration of an overdose
- Whether the subject experienced any hypoglycaemic episode and/or AE(s) as a result of the medication error
- Suspected primary reason for the medication error

For definition of medication error, see protocol Section 12.1.4.

### 1.11 Lactic acidosis

If an event of lactic acidosis is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms of lactic acidosis
- Specific laboratory tests describing the event
- Possible cause(s) of the event

### 1.12 Creatine kinase > 10 x ULN

If an event of  $CK > 10 \times ULN$  is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms associated to the event
- Recent physical activity
- Possible cause(s) of the event

### 1.12.1 Assessments in case of increased levels of creatine kinase

In case of CK > 10 x ULN, prompt repeat testing (at central laboratory) of CK should be done. Repeat testing (at central laboratory) should be done regularly until CK levels return to normal or baseline state. Additional clinical information should be gathered to seek the possible cause of the observed CK elevation.

### 1.13 Hepatic event

- ALT or AST > 5 x ULN and total bilirubin  $\le 2$  x ULN
- ALT or AST >3 x ULN and total bilirubin > 2 x ULN\*

| Protocol - Appendix B | CONFIDENTIAL | Date: | 28 January 2019 | Novo Nordisk |
|---|---|---|---|---|
| UTN: U1111-1188-1256 | | Status: | Final | |
| EudraCT no.: 2018-002589-38 | | Page: | 8 of 8 | |

Hepatic event leading to trial product discontinuation

\*Please note that risk of liver injury defined as ALT or AST > 3 x ULN and total bilirubin > 2 x ULN, where no alternative aetiology exits (Hy's law), should also be reported as a SAE (important medical event, according to protocol Section 12.1.2).

If one of the above events is observed during the trial, the following additional information must be reported if available:

- Signs and symptoms associated to the event
- Risk factors
- Relevant laboratory test results
- Diagnostic imaging performed
- Possible cause(s) of the event

### 1.13.1 Assessments in case of increased levels of aminotransferases

Both events should prompt repeat testing (at central laboratory) including ALT, AST, alkaline phosphatase (ALP) and total bilirubin and discontinuation of trial product should be considered. Thereafter, repeat testing (at central laboratory) of ALT, AST, ALP and total bilirubin should be done regularly until the abnormalities return to normal or baseline state. Additional clinical information such as related symptoms, risk factors and contributing conditions (e.g. viral hepatitis, autoimmune hepatitis, alcoholic hepatitis, hepatobiliary or pancreatic disorders) should be gathered to seek a possible cause of the observed laboratory test abnormalities.

### 1.14 Diabetic retinopathy and related complications

If an event of diabetic retinopathy or related complications is observed during the trial the following additional information must be reported, if available:

- Signs and symptoms associated with the event
- Results of the eye examination
- Treatment for and complications of the event
- Contributing conditions

## 2 References

- 1. Banks PA, Freeman ML, Practice Parameters Committee of the American College of G. Practice guidelines in acute pancreatitis. Am J Gastroenterol. 2006;101(10):2379-400.
- 2. Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, et al. Classification of acute pancreatitis-2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013;62(1):102-11.
- 3. U.S. Department of Health and Human Services, Food and Drug Administration. Guidance for Industry: Immunogenicity Assessment for Therapeutic Protein Products. August 2015.

Protocol - Appendix C Trial ID: NN9924-4309

UTN: U1111-1188-1256 EudraCT no.: 2018-002589-38

Date: Version: Status: Page:

28 January 2019 | Novo Nordisk 3.0 Final


## **Appendix C**

# Contraceptive guidance and collection of pregnancy information

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.

Protocol v 3 0 appx c | 1 of 4 Protocol - Appendix C
Trial ID: NN9924-4309


Date: 28 January 2019 | Novo Nordisk

UTN: U1111-1188-1256 CONFIDENTIAL Version: 3.0 Status: Final EudraCT no.: 2018-002589-38 

## Contraceptive guidance and collection of pregnancy information

It must be recorded in the eCRF whether female subjects are of childbearing potential

#### **Definitions**

## Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile.

## Women in the following categories are not considered WOCBP

- 1. Premenarcheal
- 2. Premenopausal female with one of the following:
- Documented hysterectomy
- Documented bilateral salpingectomy
- Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's review of subject's medical records, medical examination or medical history interview.

3. Postmenopausal female

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high Follicle Stimulating Hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or Hormonal Replacement Therapy (HRT). However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

Females on HRT and whose menopausal status is in doubt will be required to use one of the non-hormonal highly effective contraception methods if they wish to continue their HRT during the trial. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before trial enrolment.

### **Contraception guidance**

## Male subjects

No contraception measures are required for male subjects as the risk of teratogenicity/fetotoxicity caused by transfer of semaglutide in seminal fluid is unlikely.

## Female subjects

Female subjects of childbearing potential are eligible to participate if they agree to use methods of contraception consistently and correctly as described in table below:

Protocol v 3 0 appx c 2 of 4

Protocol - Appendix C
Trial ID: NN9924-4309

Date: 28 January 2019 Novo Nordisk

 Trial ID: NN9924-4309
 Version:
 3.0

 UTN: U1111-1188-1256
 Status:
 Final

 EudraCT no.: 2018-002589-38
 Page:

### Table 1 Highly effective contraceptive methods

## Highly effective contraceptive methods that are user dependent <sup>a and b</sup>

Failure rate of <1% per year when used consistently and correctly.

Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation

- oral
- intravaginal
- transdermal

Progestogen only hormonal contraception associated with inhibition of ovulation

- oral
- injectable

### Highly effective methods that are user independent <sup>b</sup>

#### Sexual abstinence

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial product. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the trial and the preferred and usual lifestyle of the subject.

Implantable progestogen only hormonal contraception associated with inhibition of ovulation

- Intrauterine Device (IUD)
- Intrauterine hormone-releasing System (IUS)
- Bilateral tubal occlusion

#### Vasectomised partner

A vasectomised partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

### Notes:

<sup>a</sup> Failure rates may differ from < 1% per year, if not used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for subjects participating in clinical trials.

Contraception should be utilised during the treatment period and for at least 35 days after the last dose of trial product.

#### Pregnancy testing

- WOCBP should only be included in the trial after a negative urine pregnancy test at visit 1 and at visit 2.
- Urine pregnancy tests should be performed throughout the trial in accordance with the protocol flowchart, section 2. WOCBP needs the last urine pregnancy test at the end of trial visit (visit 9).
- Pregnancy testing should be performed whenever a menstrual period is missed or when pregnancy is otherwise suspected.
- Additional urine pregnancy testing should be performed during the treatment period, if required locally.

Protocol v 3 0 appx c | 3 of 4

Protocol - Appendix C
Trial ID: NN9924-4309
UTN: U1111-1188-1256

Date: 28 January 2019 | Novo Nordisk
Status: Final

Page:


## Collection of pregnancy information

EudraCT no.: 2018-002589-38

### Female subjects who become pregnant

- Investigator will collect pregnancy information on any female subject, who becomes pregnant while participating in this trial.
- Information will be recorded on the appropriate form and submitted to Novo Nordisk within 14 calendar days of learning of a subject's pregnancy.
- Subject will be followed to determine the outcome of the pregnancy. The investigator will collect follow-up information on subject and neonate, which will be forwarded to Novo Nordisk. Generally, follow-up will not be required for longer than 1 month beyond the delivery date.
- Any termination of pregnancy will be reported, regardless of foetal status (presence or absence of anomalies) or indication for procedure.
- While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy will be reported as an AE or SAE.
- A spontaneous abortion is always considered to be an SAE and will be reported as such.
- Any SAE occurring as a result of a post-trial pregnancy which is considered possibly/probably related to the trial products by the investigator will be reported to Novo Nordisk as described in section 12 of the protocol. While the investigator is not obligated to actively seek this information in former subjects, he or she may learn of an SAE through spontaneous reporting.

Any female subject who becomes pregnant while participating in the trial must discontinue trial product.

Protocol v 3 0 appx c 4 of 4

Oral semaglutide Trial ID: NN9924 4309 (PIONEER 12) Clinical Trial Report Appendix 16.1.1


Date: Version: Status: 11 February 2022 | **Novo Nordisk** 1.0

Final

## **16.1.01** Protocol Attachment

Protocol Attachment I is located in the Trial Master File.

If applicable, Protocol Attachment II is also located in the Trial Master File.

Content: Global key staff and Country key staff.